## **Reporting and Analysis Plan**

**Study ID: 213500** 

Official Title of Study: Reporting and Analysis Plan Amendment 1 for 213500: A Phase IIIb, Randomized, Multicenter, Active-controlled, Parallel group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Longacting Cabotegravir Plus Long-acting Rilpivirine Administered Every Two Months from a Bictegravir/emtricitabine/tenofovir alafenamide Single Tablet Regimen in HIV-1 Infected Adults who are Virologically Suppressed.

**IND No.:** 109,678

**EudraCT No.:** 2020-002623-11

**Date of Document:** 10-May-2023

#### The GSK group of companies

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan Amendment 1 for 213500: A Phase IIIb, Randomized, Multicenter, Active-controlled, Parallel group, Non-inferiority, Open-label Study Evaluating the Efficacy, Safety, and Tolerability of Switching to Long-acting Cabotegravir Plus Long-acting Rilpivirine Administered Every Two Months from a Bictegravir/emtricitabine/tenofovir alafenamide Single Tablet Regimen in HIV-1 Infected Adults who are Virologically Suppressed |
|---|---|---|
| Compound Number | : | GSK1265744 |
| Clinical Study<br>Identifier | : | 213500 |
| Effective Date | : | Refer to Document date |

## Description:

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 213500.
- This RAP describes the statistical analyses required for the interim analysis when all participants have completed their Month 6 (OLI and BIK)/Month 5 (D2I) visit.
- The RAP also provides the content of the Primary Month 12 (OLI and BIK)/Month 11 (D2I) Statistical Analysis Complete (SAC) deliverable.
- The second amendment provides the content of the End of Study (EoS) reporting.

## RAP Author(s):

| Author | Date |
|---------------------------------------------------|-------------------|
| Lead | |
| PPD | Refer to Document |
| Principal Statistician (HIV, Clinical Statistics) | Date |

Copyright 2023 the GSK group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# Clinical Statistics & Clinical Programming Line Approvals (Method: Pharma TMF eSignature)

| Approver | |
|----------|----------------------------|
| PPD | |
| PPD | (HIV, Clinical Statistics) |

## **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTR | ODUCTION | 7 |
| 2. | CLIM | MARY OF KEY PROTOCOL INFORMATION | 0 |
| ۷. | 2.1. | | |
| | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan Study Objective(s) and Estimand(s) / Endpoint(s) | |
| | 2.2. | Study Objective(s) and Estimand(s) / Endpoint(s) | |
| | 2.4. | Statistical Hypotheses / Statistical Analyses | |
| | 2.4. | Statistical Hypotheses / Statistical Arialyses | 13 |
| 3. | PLAN | INED ANALYSES | 14 |
| | 3.1. | Interim Analyses | 14 |
| | 3.2. | Final Analyses | |
| | 3.3. | End of Study (EOS) Analyses | 14 |
| 4. | ANAI | YSIS POPULATIONS | 15 |
| | 4.1. | Protocol Deviations | |
| 5. | CON | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| | | VENTIONS | 1/ |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | |
| | 5.2. | Baseline Definitions | |
| | 5.3.<br>5.4. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | 18 |
| | 5.5. | 5.4.2. Examination of Subgroups and Covariates | |
| | 5.5. | 5.5.1. Primary Analysis | |
| | | 5.5.2. Other Comparisons of Interest | |
| | | 5.5.3. Secondary Comparisons | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | 0.0. | Conventions | 23 |
| 6. | | DY POPULATION ANALYSES | |
| | 6.1. | Overview of Planned Study Population Analyses | 23 |
| 7. | EFFI | CACY ANALYSES | 25 |
| | 7.1. | Primary Efficacy Analyses | |
| | | 7.1.1. Endpoint / Variables | |
| | | 7.1.2. Summary Measure | |
| | | 7.1.3. Population of Interest | 25 |
| | | 7.1.4. Strategy for Intercurrent (Post-Randomization) Events | 26 |
| | | 7.1.5. Statistical Analyses / Methods | 26 |
| | 7.2. | Secondary Efficacy Analyses | |
| | | 7.2.1. Endpoint / Variables | |
| | | 7.2.2. Summary Measure | |
| | | 7.2.3. Population of Interest | |
| | | 7.2.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | CCI | 7.2.5. Statistical Analyses / Methods | 30 |

| 8. | | TY ANALYSES | |
|---|---|---|---|
| | 8.1. | Adverse Events Analyses | |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | | 8.2.1. Analyses for Injection Site Reaction Adverse Events | |
| | 8.3. | Clinical Laboratory | |
| | 8.4. | Biomarker Analyses | |
| | | 8.4.1. Bone Biomarkers | |
| | | 8.4.2. Renal Biomarkers | 43 |
| | 8.5. | Other Safety Analyses | 44 |
| | | 8.5.1. ECG | |
| | | 8.5.2. Metabolic Syndrome | |
| | | 8.5.3. Anthropometric profile | |
| | | 8.5.4. HOMA-Insulin Resistance | |
| 9. | POPU | ILATION PHARMACOKINETIC (POPPK) ANALYSES | 48 |
| 10. | PHAR | MACOKINETIC ANALYSES | 48 |
| 11. | PHAR | MACODYNAMIC (AND / OR BIOMARKER) ANALYSES | 48 |
| 12. | PHAR | MACOKINETIC / PHARMACODYNAMIC ANALYSES | 48 |
| 13. | HEAL | TH OUTCOMES ANALYSIS | 48 |
| | 13.1. | | |
| | 13.2. | | |
| | 13.3. | | |
| | 13.4. | Strategy for Intercurrent (Post-Randomization) Events | 49 |
| | 13.5. | Statistical Analyses / Methods | |
| | | 13.5.1. Statistical Methodology Specification | 51 |
| 14. | VIRO | LOGY | 54 |
| 15. | REFE | RENCES | 56 |
| 10 | | | |
| 10. | 16.1. | NDICESAppendix 1: Protocol Deviation Management and Definitions for Per | 58 |
| | 10.1. | Protocol Population | 58 |
| | | 16.1.1. Exclusions from Per Protocol Population | |
| | 16.2. | Appendix 2: Schedule of Activities | |
| | 16.3. | Appendix 3: Assessment Windows | |
| | | 16.3.1. Definitions of Assessment Windows for Analyses | |
| | | 16.3.2. Definitions of Assessment Windows for Data Other than | |
| | | Health Outcomes | |
| | | 16.3.3. Assessment Window for Study Conclusion | |
| | | 16.3.4. Assessment Window for Health Outcome Data | |
| | | 16.3.5. Multiple assessments within an Analysis Window | |
| | 16.4. | Appendix 4: Study Phases and Treatment State | |
| | | 16.4.1. Study Phases | |
| | | 16.4.2. Study Periods | |
| | | 16.4.3. Treatment State | |
| | 16 E | 16.4.4. Combining Treatment Phases and States | |
| | 16.5. | Appendix 5: Data Display Standards & Handling Conventions | 98 |

| | 40.54 | |
|---|---|---|
| | 16.5.1. Reporting Process | |
| 40.0 | 16.5.2. Reporting Standards | |
| 16.6. | Appendix 6: Derived and Transformed Data | |
| | 16.6.1. General | |
| | 16.6.2. Study Population | |
| | 16.6.3. Efficacy | |
| | 16.6.4. Safety | |
| | 16.6.5. Pharmacokinetic | 114 |
| | | 440 |
| 16.7. | 16.6.7. Viral Genotype and Phenotype | |
| 10.7. | Appendix 7: Reporting Standards for Missing Data | |
| | 16.7.1. Premature Withdrawals | |
| 16.0 | 16.7.2. Handling of Missing Data | |
| 16.8.<br>16.9. | Appendix 8: Values of Potential Clinical Importance | |
| | Appendix 9: Snapshot Algorithm Details | 127 |
| 16.10. | Appendix 10: Variables Defined for Time to Event Analysis | 134 |
| 10.11. | (AESI) | 126 |
| | · · | |
| | 16.11.1. Hepatic Safety Profile | |
| | 16.11.3. Rash | |
| | 16.11.4. Prolongation of the Corrected QT Interval of the ECG in | 140 |
| | Supratherapeutic Doses | 1.11 |
| | 16.11.5. Suicidal Ideation/Behaviour | |
| | 16.11.6. Depression | |
| | 16.11.7. Bipolar Disorder | |
| | 16.11.8. Psychosis | |
| | 16.11.9. Mood Disorders | |
| | 16.11.10. Anxiety | |
| | 16.11.11.Sleep Disorders | |
| | 16.11.12.Injection Site Reactions (ISR) | |
| | 16.11.13. Seizures and Seizure-like Events | |
| | 16.11.14. Weight Gain | |
| | 16.11.15.Rhabdomyolysis | |
| | 16 11 16 Pancreatitis | |
| | 16.11.17.Impact on Creatinine | |
| | 16.11.18. Safety in Pregnancy | |
| 16 12 | Appendix 12: Identification of COVID-19 Adverse Events | |
| | Appendix 13: Data Handling for Pregnant Subjects | |
| | Appendix 14: Abbreviations & Trade Marks | |
| 10.14. | 16.14.1. Abbreviations | |
| | 16.14.2. Trademarks | |
| 16 15 | Appendix 15: List of Data Displays | |
| 10.10. | 16.15.1. Data Display Numbering | |
| | 16.15.2. Mock Example Shell Referencing | |
| | 16.15.3. Deliverables | |
| | 16.15.4. Study Population Tables | |
| | 16.15.5. Efficacy Tables | |
| | 16.15.6. Efficacy Figures | |
| | 16.15.7. Safety Tables | |
| | 16.15.8. Safety Figures | |
| | 16.15.9. Health Outcome Tables | |

| | 213500 |
|-----------------------------------------------------------|--------|
| 16.15.10. Virology Tables | 199 |
| 16.15.11.ICH Listings | 201 |
| 16.15.12.Non-ICH Listings | 204 |
| 16.16. Appendix 16: Example Mock Shells for Data Displays | 210 |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | | |
|---|---|---|
| 2019N425725_00 | 27-MAY-2020 | Original |
| 2019N425725_01 | 30-JUN-2020 | The primary reason for protocol amendment 01 is to add minor clarifications to address study completion, PK collection, and endpoint timings. Country-specific details were added to Appendix 10 to address UK MHRA requirements. The protocol short title was updated. Corrections to typographical errors in protocol text and title were made throughout. |
| TMF-12473407 | 08-SEP-2021 | The primary reason for protocol amendment 02 is to address and clarify comments raised during the course of the study and to implement country specific changes following regulatory review. |
| TMF-14364917 | 10-FEB-2022 | The primary reason for protocol amendment 03 is to address and clarify comments raised during the course of the study. |

This first amendment includes amendments to the originally approved RAP effective 27Dec2021. The following changes were made prior to the M12 primary analysis:

Major (applicable to M12 only):

- Updated primary analysis population to mITT-E excluding subjects from site PPD
- Added modified CVF (mCVF) population excluding subjects from site PPD
- Updated that Per Protocol (PP) will be based on mITT-E
- Updated in Appendix 15 analysis population for the M12 analysis tables

Minor (typo corrections, clarifications, additional displays and format changes):

- Updated in Section 2.2 in consistency with updates in protocol amendment 3
- Updated in Appendix 2
- Updated in Section 8.4 that "Interactions between treatment and each of the covariates will not be assessed" For MMRM models.
- Updated the title for the listing "Listing of HIV-1 Associated Conditions" to "Listing of Stage 3 HIV-1 Associated Conditions".
- Updated the title for Safety Figure 3.2 "Plot of Incidence of Maintenance Phase Drug-Related Injection Site Reaction Adverse Events by Visit (Overall and Common)" by adding "Drug-Related" to the title for accuracy
- Updated the title for Safety Figure 3.3 "Plot of Incidence of Grade 3-5 Maintenance Phase Drug-Related Injection Site Reaction Adverse Events by Visit (Overall and Common)" by adding "Drug-Related" to the title for accuracy
- Updated the title for Safety Figure 3.9 "Plot of Incidence of Maintenance Phase Drug-Related Injection Site Reaction Adverse Events by Strata and Visit (Overall and Common) - CAB and/or RPV" by adding "Drug-Related" to the title for accuracy

- Clarified Safety Table 3.64 "Summary of Percent of Subjects with Metabolic Syndrome and Risk Factors" is for "Maintenance Phase"
- Removed the output "Proportion of Subjects with Plasma HIV-1 RNA <2 c/mL Observed Case Analysis (Maintenance Phase)"
- Moved the listing of net assessment data into separate listings for CVF and non-CVF subjects due to space limit in the output files (2 extra listings added)
- Divided the figure "Patient Profile Plot of Clinical Diagnosis Factors for Patients with Metabolic Syndrome at Any Time Point" to separate figures for OLI, D2I and BIK due to space limit in the output files (2 extra figures added)
- Corrected a typo in Section 16.15.9 that the analysis population for Health Outcomes table 6.13
   "Proportion of Subjects Scoring Each Option in the Communication Questionnaire at Month 13" is "Extension Switch" instead of ITT-E.
- Added in Section 16.15.9 "Statistical Analysis of HIVTSQs Change from Maintenance Baseline (Day 1) in Total Treatment Satisfaction Score and individual items 5 (convenient), 6 (flexible) and 10 (continue) (Maintenance Phase) by Baseline Score Group" and "Summary of Shift in Column
- Updated description in the cell questionnaire in Section 16.6.6 to align with eCRF wording.
- Corrected that the analysis population for listing "Listing of Plasma PK Concentrations at Withdrawal" will be ITT-E.
- Added in Section 16.15.12 "Listing of All Plasma PK Concentrations for CVF Subjects".
- Added clarification in Section 16.15.12 that the following two displays will not be produced if no subject becomes pregnant on Q2M: "Listing of Selected Laboratory Data for Subjects Who Became Pregnant During the Study", "Listing of Plasma PK Concentrations for Subjects Who Became Pregnant During the Study".
- Added clarification on data handling strategy for Q2M subjects who become pregnant on study in Section 16.13.

The second amendment includes amendments to the RAP amendment #1 effective 15-Jun-2022, the following changes were made:

Section 16.5 was updated to provide additional details of the planned analyses and data displays for 213500 EOS Final reporting.

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Due to critical audit findings at site PPD related to critical inclusion/exclusion criteria violations and major GCP non-compliance (reporting letter to FDA submitted), efficacy data from this site is deemed unreliable and as such the M12 primary analysis population will exclude all 11 randomized site participants (mITT-E). Efficacy analysis in the "mITT-E" population will be considered primary. Additional (sensitivity) efficacy analyses will be performed for the ITT-E population and this analysis will be considered secondary/supportive. Safety analyses will remain as planned and will include all randomized subjects who received at least one dose of study treatment (Safety). For virology tables (if applicable) and one efficacy table, the mCVF population will be summarized excluding any subject from the site. All listings and subject-level figures will be produced as planned, without exclusion of the site, where applicable. See Appendix 15. Note this update is made after the Month 6 but prior to the M12 analysis therefore such changes are only applicable to the M12 analysis.

## 2.2. Study Objective(s) and Estimand(s) / Endpoint(s)

| Objectives | Estimands/Endpoints |
|---|---|
| Primary | |
| To demonstrate the non-inferior antiviral activity of CAB LA + RPV LA every two months compared to a BIK single tablet regimen administered once daily over 12 months in suppressed HIV-1 infected antiretroviral therapy (ART)-experienced participants | Proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Month 12 (OLI and BIK)/Month 11 (D2I) (Intent-to-Treat Exposed [ITT-E] population) |
| Secondary | |
| To demonstrate the antiviral and immunologic response with the use of CAB LA + RPV LA every 2 months compared to a BIK single tablet regimen administered once daily | Proportion of participants with plasma HIV-1 RNA<br><50 c/mL (c/mL) at Month 6 and Month 12 (OLI<br>and BIK)/Month 5 and Month 11 (D2I) using the<br>FDA Snapshot algorithm (Intent-to-Treat Exposed<br>[ITT-E] population) |
| | Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| | Proportion of participants with HIV-RNA greater than or equal to 50 c/mL as per FDA Snapshot algorithm at Month 6, and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I) |
| | Absolute values and changes from Baseline in viral load and CD4+ cell count over time including Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I) |
| To assess viral resistance in participants experiencing protocol-defined confirmed virologic failure | Incidence of treatment emergent genotypic and phenotypic resistance to CAB, RPV, BIC, FTC, and TAF through Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| To evaluate renal (in urine and blood) and bone (in blood) biomarkers in participants treated with CAB LA + RPV LA compared to BIK | Change from Baseline (Day 1) in renal and bone biomarkers at Months 6 and 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| To evaluate Metabolic Syndrome for participants treated with CAB + RPV and BIK | Change from Baseline in proportions of participants with Metabolic syndrome at Months 6 and 12 (OLI and BIK)/Month 5 and Month 11 (D2I) |

| Objectives | Estimands/Endpoints |
|---|---|
| To evaluate insulin resistance in participants treated with CAB LA + RPV LA compared to BIK | Change from Baseline (Day 1) in homeostasis model of assessment-insulin resistance (HOMA-IR) at Months 6 and 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| To assess preference for CAB LA + RPV LA administered every 2 months compared to a BIK single tablet regimen administered once daily | Preference for CAB LA + RPV LA every 2 months compared to a BIK single tablet regimen will be assessed using a preference questionnaire at Month 12 (OLI )/Month 11 (D2I) (or Withdrawal). |
| To assess patient reported treatment satisfaction, and injection tolerability. | Change from baseline (Day 1) in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I), (or Withdrawal) |
| | Change in treatment satisfaction over time using the HIV Treatment Satisfaction Change Questionnaire HIVTSQc total score and individual item scores at Month 12 (OLI and BIK)/Month 11 (D2I) (or Withdrawal). |
| | Change from Month 2 in Dimension scores ("Acceptance of ISRs", "Bother of ISRs", "Leg movement", "Sleep") and individual item scores (assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time) will be assessed using the Perception of injection questionnaire (PIN) at Months 2, 6, and 12 (OLI)/Months 1, 5, 11 (D2I) (or Withdrawal) |
| Safety | |
| To evaluate the safety and tolerability of CAB LA + RPV LA every 2 months compared to a BIK single tablet regimen administered once daily | Incidence and severity of AEs and laboratory abnormalities over time including Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| | Proportion of participants who discontinue treatment due to AEs over time including Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |
| | Change from Baseline in laboratory parameters over time including Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I). |

| Objectives | Estimands/Endpoints |
|------------|---------------------|
| CCI | |



## 2.3. Study Design



| Overview of St | udy Design and Key Features |
|---|---|
| Overview of St | and/or RPV LA and discontinues the CAB LA + RPV LA regimen for any reason will enter the Long-term Follow-up Phase on suppressive HAART for at least 52 weeks after the last dose of CAB LA and/or RPV LA. |
| Dosing | <ul> <li>Maintenance Phase: <ul> <li>CAB LA (600 mg) + RPV LA (900 mg) IM every 2 months</li> <li>Oral BIK once daily</li> </ul> </li> <li>Extension Phase: <ul> <li>CAB LA (600 mg) + RPV LA (900 mg) IM every 2 months</li> </ul> </li> </ul> |
| Time & Events | [Refer to Appendix 2] |
| Treatment<br>Assignment | <ul> <li>Maintenance Phase: Approximately 654 subjects randomized 2:1 to CAB LA + RPV LA vs. Oral BIK. Subjects randomized to receive CAB LA + RPV LA may choose to begin oral therapy with CAB 30 mg + RPV 25 mg once daily (OLI) prior to administration of CAB LA + RPV LA, or transition directly to injections (D2I).</li> <li>Extension Phase: if meeting eligibility requirements, subjects randomized to CAB LA + RPV LA will continue to have access to their randomized regimen; subjects randomized to BIK will have the option to either continue study participation by switching to CAB LA + RPV LA, or complete the study at Month 12.</li> <li>GSK RandAll NG will be used to generate randomization schedules.</li> <li>Stratified Randomization by participants' Baseline BMI (&lt; 30 kg/m², ≥ 30 kg/m²) and Gender at Birth (female, male).</li> </ul> |
| Interim<br>Analysis | <ul> <li>An interim analysis will be conducted when all participants have completed their Month 6 (OLI and BIK)/Month 5 (D2I) visit.</li> <li>The main analysis will be conducted to evaluate the primary objective of the protocol at Month 12(OLI and BIK)/Month 11(D2I).</li> <li>Further data cuts and analyses may be conducted as necessary in order to support regulatory submissions and publications.</li> </ul> |

## 2.4. Statistical Hypotheses / Statistical Analyses

The study is to demonstrate the non-inferior antiviral activity of CAB LA + RPV LA (Q2M) every 2 months compared to a BIK single tablet regimen administered once daily over 12 months in suppressed HIV-1 infected antiretroviral therapy (ART)-experienced participants.

Non-inferiority will be concluded if the upper limit of a two-sided 95% confidence interval for the difference in proportion of participants with HIV-1 RNA  $\geq$  50 c/mL at Month 12 (OLI and BIK)/Month 11 (D2I) between the two treatment arms (Q2M - BIK) is less than 4%. Note that efficacy data for the primary endpoint from the OLI subjects at Month 12 and from the D2I subjects at Month 11 will be combined for the Q2M arm when assessing non-inferiority.

Let pc, pb be the proportion of participants with HIV-1 RNA  $\geq$  50 c/mL in the CAB LA+RPV LA (Q2M) and BIK arms respectively, then the primary statistical hypothesis can be written as follows:

H<sub>0</sub>: pc - pb 
$$\geq$$
 4% vs. H<sub>a</sub>: pc - pb  $\leq$  4%

## 3. PLANNED ANALYSES

## 3.1. Interim Analyses

An interim analysis will be conducted when all participants have completed their Month 6 (OLI and BIK)/Month 5 (D2I) visit, focusing on the interim efficacy and key secondary efficacy endpoints, as well as key safety endpoints.

To minimise bias, the Month 6 interim results will not be shared with any participant and with most investigators. However, when a lead author(s) for a potential abstract presentation of the Month 6 interim results is (are) identified, that investigator(s) and the other co-authors on the abstract will have access to the interim results prior to its presentation. No other investigators will have knowledge of this data prior to the last participant completing their last visit for the primary Month 12 analysis. A Month 6 interim analysis abstract may be submitted to a conference for consideration only if the conference convenes after the Month 12 data collection has been completed.

Further data cuts and analyses may be conducted as necessary to support regulatory submissions, publications or for other purposes. Additionally, information collected on pregnant participants as collected in the eCRF may be reported descriptively or listed. The Month 12 analysis will be primary. No adjustment for multiplicity caused by repeated evaluation of the primary endpoint will be made as the Month 6 interim analyses will be secondary.

## 3.2. Final Analyses

The primary Month 12 analysis will be conducted to evaluate the primary objective of the protocol when all participants have completed their Month 12 (OLI and BIK)/Month 11 (D2I) visit. These analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed their Month 12 (OLI and BIK)/Month 11 (D2I) visit as defined in the protocol and had a re-test if necessary
- 2. All required database cleaning activities have been completed and final database release (DBR), source data lock (SDL) and database freeze (DBF) have been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG procedures.

## 3.3. End of Study (EOS) Analyses

A final End-of-Study analysis will be conducted when all subjects have completed the study.

Details of which outputs will be produced at End of Study can be found in Section 16.5.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | <ul> <li>All participants who were screened for eligibility.</li> <li>Subjects may be re-screened once and will be assigned a new subject number.</li> <li>For disposition displays, except for the listing of subjects who were rescreened, only the latest rescreening data will be included.</li> </ul> | Study Population |
| Enrolled | <ul> <li>All participants who passed screening and entered the study.</li> <li>Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study are excluded from the Enrolled population as they did not enter the study.</li> </ul> | Study Population |
| Randomized | <ul> <li>All participants who were randomly assigned to treatment in the study.</li> <li>This population will be based on the treatment the participant was randomized to.</li> </ul> | Study Population |
| Safety | <ul> <li>All randomized participants who received at least one dose of study treatment.</li> <li>This population will be based on the actual treatment the participant received.</li> <li>Note: participants who were not randomized but received at least one dose of study treatment will be listed separately.</li> </ul> | <ul> <li>Safety</li> <li>Virology (if applicable)</li> </ul> |
| Intent-to-Treat<br>Exposed (ITT-E) | <ul> <li>All randomized participants who receive at least<br/>one dose of IP during the Maintenance Phase of<br/>the study (on or after Day 1).</li> <li>Participants will be analyzed according to the<br/>randomized treatment regardless of the actual<br/>treatment received.</li> </ul> | <ul><li>Study Population</li><li>Efficacy</li></ul> |
| Modified Intent-<br>to-Treat (mITT-<br>E) | All ITT-E subjects excluding those from sitePPD | <ul><li>Study Population</li><li>Efficacy</li><li>Health<br/>Outcomes</li></ul> |
| Per-Protocol<br>(PP) | <ul> <li>All participants in the mITT-E population except major protocol violators.</li> <li>Protocol deviations that exclude subjects from the Per-Protocol population are defined in Section 4.1 (Protocol Deviations) and Appendix 1 (Protocol Deviation Management and Definition for Per-Protocol Population).</li> </ul> | Efficacy (Sensitivity Analysis) |
| Extension Switch<br>(ES) | <ul> <li>All randomized subjects from BIK arm who receive at least one dose of CAB and/or RPV during the Extension Phase of the study.</li> <li>Participants will be assessed according to actual treatment received during the Extension Phase.</li> </ul> | Safety and efficacy for BIK subjects switching to Extension Q2M if applicable |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Pharmacokinetic (PK) | <ul> <li>All participants who receive CAB and / or RPV and<br/>undergo PK sampling during the study and provide<br/>evaluable CAB and / or RPV plasma concentration<br/>data with at least 1 non-missing PK assessment<br/>(Non-quantifiable [NQ] values will be considered as<br/>non-missing values).</li> </ul> | PK (Pregnant<br>subjects on Q2M<br>arm only for this<br>RAP) |
| | <ul> <li>Note: PK samples that may be affected by protocol<br/>deviations will be reviewed by the study team to<br/>determine whether or not the sample will be<br/>excluded.</li> </ul> | |
| Confirmed | All participants in the ITT-E population who met | <ul> <li>Virology</li> </ul> |
| Virologic Failure<br>(CVF) | Confirmed Virologic Failure (CVF) • CVF during the Maintenance and/or Extension Phases is defined as: Rebound as indicated by two consecutive plasma HIV-1 RNA levels ≥200 c/mL (Day 1 values not applicable) after prior suppression to <200 c/mL | Efficacy |
| Modified | All participants in the mITT-E population who met | <ul> <li>Virology</li> </ul> |
| Confirmed Virologic Failure (mCVF) | <ul> <li>Confirmed Virologic Failure (CVF)</li> <li>Note this population is only applicable to summary tables</li> </ul> | Efficacy |
| Long-term<br>Follow-up<br>(LTFU) | <ul> <li>Discontinued subjects who have received at least one dose of CAB LA and/or RPV LA and have met any of the following criteria:</li> <li>have at least one Long-term Follow-up phase clinic visit,</li> <li>have filled out the LTFU phase conclusion form,</li> <li>or have indicated the continuation to LTFU phase in the subject continuation form.</li> </ul> | Safety |

Refer to Appendix 15: List of Data Displays which details the population used for each display.

#### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Important deviations which result in exclusion from the analysis population will also be summarised and listed. (Please refer to Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population)].

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.

- Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations which may lead to exclusion from the analysis population(s) are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

## 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| Ran | RandAll NG Randomization System Data Displays for Reporting | | |
| Code | Description | Description Order in TL | |
| Α | CAB LA + RPV LA Q2M | Q2M | 1 |
| В | BIK QD | BIK | 2 |

Note: Treatment comparisons will be displayed as follows using the descriptors as specified: Q2M vs. BIK (Q2M – BIK)

The following sub-display may be used as appropriate under the Q2M treatment group as noted in Appendix 15: List of Data Displays.

| | Data Display for Reporting | Order for sub-display |
|---|---|---|
| For subjects randomized to Q2M during the | OLI | 1 |
| Maintenance Phase | D2I | 2 |

In data displays of Extension Phase data for the Extension Switch population who switched from BIK, "Switch Q2M" will be used. In displays where sub study treatment will be displayed, descriptors are as shown below.

| | Data Display for Reporting | Order for sub-display |
|---|---|---|
| Extension Phase data for the Extension Switch | Switch OLI | 1 |
| population (Switch Q2M) | Switch D2I | 2 |

#### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled

visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and used as baseline.

Electrocardiograms (ECGs) are to be performed in triplicate prior to first dose on Day 1. The baseline value for an ECG parameter will be the mean of the last pre-treatment set of assessments from the same date.

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

#### 5.3. Multicentre Studies

Data will be summarized for all centres combined. Country may be treated analyses of the primary efficacy endpoint (HIV-1 RNA ≥50 c/mL) as described in Section 7.1.5.1. and secondary efficacy endpoint (HIV-1 RNA <50 c/mL) as described in Section 7.2.5.1. □□

## 5.4. Examination of Covariates, Other Strata and Subgroups

#### 5.4.1. Covariates and Other Strata

The list of covariates and other strata may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses. Additional covariates of clinical interest may also be considered for additional analyses on Health Outcomes and Biomarker analyses.

| Category | Details |
|---|---|
| Strata | <ul> <li>For the proportion of participants with plasma HIV-RNA greater than or equal to 50 c/mL per FDA Snapshot algorithm at Month 12 (OLI and BIK)/Month 11 (D2I) (primary endpoint), a stratified analysis with Cochran-Mantel Haenszel (CMH) weights will be used to adjust the primary treatment comparison with the randomization strata corresponding to Gender at Birth (female, male) and Baseline BMI (&lt;30 kg/m², ≥30 kg/m²).</li> <li>A similar approach will be used to adjust the analysis of the proportion of participants with HIV-1 RNA &lt;50 c/mL (per the FDA's Snapshot algorithm) at Month 12(OLI and BIK)/Month 11 (D2I)</li> <li>The analyses as described above will also be applied in the interim analysis for key efficacy endpoints at Month 6 (OLI and BIK)/Month 5 (D2I).</li> </ul> |
| Covariates | See details in Section 5.4.2 |

### 5.4.2. Examination of Subgroups and Covariates

The following is a list of subgroups that may be used in descriptive summaries and statistical analyses. Additional subgroups of clinical interest may also be considered.

- If the percentage of participants is small within a particular subgroup, then the subgroup categories may be combined prior to unblinding the trial.
- If the category cannot be refined further, then descriptive rather than statistical comparisons may be performed for the particular subgroup.
- For subgroup analysis, per European Medicines Agency Guideline on the investigation of subgroups in confirmatory clinical trials (EMA, 2019), factors defining a subgroup population may be put in three categories:
  - 1. Factors with strong reason to expect an inconsistent response to treatment across the different levels of the factor to an extent that would make an overall assessment uninterpretable. In this case separate trials should usually be planned.
  - 2. Factors with reason to consider it prognostic for outcome, or at least some biological plausibility or external evidence such that an inconsistent response might be observed. In this study, stratified randomization strata, key demographic and baseline characteristic factors, will fall into this category. For these factors, subgroup analyses will be performed but likely underpowered so that a formal proof of efficacy will not be available individually in all subgroups. If consistent findings across multiple comparisons were observed, then these analyses would still be suggestive of a generalizable finding from the overall population.
  - 3. Factors with good argumentation why consistency of response to treatment is plausible or for which there is absence of pharmacological rationale and absence of clinical evidence from which to determine the plausibility of consistent drug effects. The impact of factor(s) falling into this category will be explored.

| Subgroup Category | Subgroup and Subgroup Levels |
|---|---|
| EMA Subgroup Category 2: | |
| Randomization Strata | <ul> <li>Baseline BMI: &lt;30 kg/m², ≥30 kg/m²</li> <li>Gender at Birth: female, male</li> </ul> |
| | For analysis purposes, randomization strata will be derived using eCRF data (which may differ from the strata captured in RAMOS NG). |
| | All statistical analyses will adjust for the above randomization strata, unless stated otherwise. Treatment-by-Strata interactions will be assessed as specified in the analysis sections. |
| Demographic and Baseline<br>Characteristic Subgroups | <ul> <li>Age</li> <li>Descriptive summaries: &lt; 35, 35 - &lt; 50, ≥ 50</li> <li>Statistical analyses: &lt; 50, ≥ 50</li> <li>FDAAA: ≤18, 19 - 64, ≥ 65</li> <li>EMA: 18 - 64, 65 - 84, ≥ 85</li> </ul> |
| | Race |

| Subgroup Category | Subgroup and Subgroup Levels |
|---|---|
| EMA Subgroup Category 2: | • |
| | <ul> <li>White; Non-White</li> <li>Black/ African American; Non- Black/ African American</li> <li>White, Black/African American, Other</li> <li>For statistical modelling of biomarkers, use White, Black/African American vs. Other.</li> <li>For other statistical modelling, use White vs Non-White.</li> </ul> |
| | <ul> <li>Country (not used for statistical modelling)</li> <li>Canada</li> <li>United Kingdom</li> <li>Ireland</li> <li>France</li> <li>Germany</li> <li>Spain</li> <li>Italy</li> <li>Switzerland</li> <li>Austria</li> <li>Netherlands</li> <li>Belgium</li> <li>Japan</li> <li>Australia</li> <li>United States</li> </ul> |
| | <ul> <li>Region North America, Europe, Rest of World</li> <li>Baseline CD4+ cell count (cells/mm³) &lt;350, 350 to &lt;500, ≥ 500 cells/mm³</li> </ul> |
| | <ul> <li>Derived Maintenance Baseline (Day 1) Centres for<br/>Disease Control and Prevention (CDC) category:</li> <li>Stage I, Stage II, Stage III</li> </ul> |
| | <ul> <li>Baseline HIV-1 Subtype (if available at the time of the analysis)</li> <li>A, A1, AE, AG, B, C, Other</li> </ul> |
| | <ul> <li>INI Regimen prior to BIK</li> <li>Raltegravir, Elvitegravir, Dolutegravir, none.</li> </ul> |
| | Duration of Prior ART (including BIK) use before study entry (<1 year, 1 - <2, 2 - <3 ,3-<4, >=4 years) |

| Subgroup Category | Subgroup and Subgroup Levels |
|---|---|
| EMA Subgroup Category 2: | |
| EMA Subgroup Category 3: | |
| ISR-related: Needle length | <ul> <li>For the maximum toxicity grade of each preferred term of the common ISR (pain, induration, nodules and any other ISR with &gt;=5% subjects in the Q2M treatment arm) during the maintenance phase:</li> <li>Needle Length for Last CAB Injection prior to and including the onset date of the earliest corresponding CAB ISR with maximum toxicity grade during the Maintenance Phase: (&lt;1.5, 1.5 to &lt;2, ≥2 inch);</li> <li>Needle Length for Last RPV Injection prior to and including the onset date of the earliest corresponding RPV ISR with maximum toxicity grade during the Maintenance Phase: (&lt;1.5, 1.5 to &lt;2, ≥2 inch);</li> <li>Note: If there is no ISR of interest reported during maintenance phase for a subject, the needle length of last injection during maintenance phase will be used in the summary.</li> </ul> |

## 5.5. Multiple Comparisons and Multiplicity

There are no planned adjustments for multiple comparisons or multiplicity.

## 5.5.1. Primary Analysis

The primary comparison of interest is the comparison between CAB LA + RPV LA (Q2M) and BIK for the primary endpoint in the mITT-E population at Month 12 (OLI and BIK)/Month 11 (D2I). The primary comparison will be made at a one-sided 2.5% level of significance. Treatment with CAB LA + RPV LA (Q2M) will be declared non-inferior to BIK if the upper bound of a two-sided 95% confidence interval for the difference (Q2M – BIK) in proportion of participants with HIV-1 RNA  $\geq$  50 c/mL is below 4%.

If the primary analysis demonstrates non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring CAB LA + RPV LA (Q2M) will be declared if the upper limit of the confidence interval is below 0% for the mITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

No multiple comparison adjustment is necessary for testing non-inferiority followed by superiority (conditional on achieving significance in the non-inferiority test) since testing follows a pre-specified sequence of hypothesis such that if the first hypothesis tested is not significant, all subsequent tests will not be performed. This fixed sequence procedure controls the type I error rate at the nominal level.

Subjects who became pregnant during the study will be allowed to continue CAB LA + RPV LA (Q2M) treatment, while those who became pregnant on BIK will be withdrawn. To minimize bias, a "while on-treatment" strategy will be implemented. Viral load data collected after confirmed pregnancy will not be evaluated for summary tables and statistical analysis in the primary analysis (see Appendix 13: Data Handling for Pregnant Subjects).

## 5.5.2. Other Comparisons of Interest

The following sensitivity analysis will also be performed for consistency with the results from the primary analysis:

- Same analysis as described above with the PP population
- Same analysis as described above with the ITT-E population
- Same analysis as described above with all data as observed (not applicable if no subject on the Q2M arm becomes pregnant)

## 5.5.3. Secondary Comparisons

If the primary comparison of interest (Section 5.5.1) using the mITT-E population demonstrates non-inferiority of CAB LA + RPV LA (Q2M) compared to BIK at the primary analysis timepoint, then the following key secondary comparisons using the mITT-E population will be tested:

- Treatment comparisons between the two arms (Q2M BIK) with respect to the proportion of participants with HIV-1 RNA < 50 copies/mL at Months 12 (OLI and BIK)/Month 11 (D2I) (defined by the US FDA snapshot algorithm), including the two-sided 95% confidence interval. If the lower limit of the confidence interval for the difference in response rates (Q2M-BIK) lies **above -12%** then non-inferiority can be concluded.
- Sensitivity analysis as described in Section 5.5.2 in the PP population and with all data observed will also be performed, for secondary comparisons. Additional comparisons of clinical interest between two treatment arms may also be performed as supportive analyses.
- In addition to the primary and the key secondary comparisons, the comparisons between two treatment arms for HIVTSQs (Treatment Satisfaction Status Score), HIVTSQc (Treatment Satisfaction Change score), the statistical test on change in PIN acceptance score within the Q2M arm over time using a two-sided 5% level of significance will also be performed as supportive analyses.

## 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---|---|
| 16.3 | Appendix 3: Assessment Windows |
| 16.4 | Appendix 4: Study Phases and Treatment State |
| 16.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 16.5 | 16.5 Appendix 6: Derived and Transformed Data |
| 16.7 | Appendix 7: Reporting Standards for Missing Data |
| 16.8 | Appendix 8: Values of Potential Clinical Importance |
| 16.9 | Appendix 9: Snapshot Algorithm Details |
| 16.10 | Appendix 10: Variables Defined for Time to Event Analysis |
| 16.11 | Appendix 11: Identification of Adverse Events of Special Interest (AESI) |
| 16.12 | Appendix 12: Identification of COVID-19 Adverse Events |
| 16.13 | Appendix 13: Data Handling for Pregnant Subjects |

## 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified. Note in the Month 12 analysis, mITT-E will be used in summary tables.

Study population analyses including analyses of participant's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards.

Table 1 provides an overview of the planned study population analyses, with full details of data displays presented in Appendix 15: List of Data Displays

Table 1 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | |
|---|---|---|
| | Table | Listing |
| Randomization | | |
| Randomization [1] | | <b>Y</b> [2] |
| Subject Disposition | | |
| Study Populations [3] | Y | |
| Study Recruitment [3] | Y | |
| Reasons for Screening Failures [3] | Y | Υ |
| Age categories | Y | |
| Subject Disposition | <b>Y</b> [4][5] | |
| Reasons for Withdrawal | <b>Y</b> [4][5] | Υ |
| IP discontinuation | Υ | Υ |
| Important Protocol Deviations | Υ | Υ |
| Deviations leading to exclusion from PP | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | Y | Υ |
| Demography and Baseline | | |
| Demographics Characteristics [6] | Y | Υ |
| Race & Racial Combinations [7] | Y | Υ |
| Hepatitis Status at Entry | Y | |
| CDC Classification of HIV infection (2014) at Maintenance<br>Baseline (Day 1) | Y | |
| Distribution of CD4+ Cell Counts at Screening and Maintenance Baseline (Day 1) | Y | |
| HIV Risk Factors | Υ | |
| Medical Conditions, Concomitant Medications & Antiretroviral | Therapy | |
| Medical Conditions (Current/Past) [8] | Υ | |
| Medical Conditions: Sub-conditions (Current/Past) [9] | Υ | |
| Concomitant Medications (non-ART) | <b>Y</b> [10] | |
| Prior Antiretroviral Therapy | Υ | Υ |
| Concomitant Antiretroviral Therapy during Maintenance Phase | | Y |
| ART Medications Received during LTFU Phase | | Y |
| Lipid Modifying Agents (Maintenance Baseline (Day 1) and During Maintenance Phase) | Y | |
| Substance use at Screening | Υ | |
| Medical History of Seizure | | Υ |
| Other | | |
| Study Treatment Accountability [11] | | Υ |

#### NOTES:

- T = Tables, L = Listings, Y = Display Generated,
- 1. Based on Randomized population
- 2. One listing of participants randomized but not treated, and one listing of planned and actual treatment strata.
- 3. All Subjects screened population.
- 4. Participants who have not been recorded as either completing or withdrawing from the study will be categorized as "Ongoing at time of the analysis" for summary purposes.
- 5. Analysis of subject disposition may be performed for each study Phase separately if applicable, as well as for overall study conclusion.
- 6. Age and ethnicity collected at Screening; weight, height and BMI collected at Day 1,
- 7. The five high level FDA race categories and designated Asian subcategories will be summarised along with all combinations of high-level categories which exist in the data. The nine race categories collected will be summarised along with categories for mixed race. A by-subject listing of race will also be produced.
- 8. Medical conditions will be coded using the Medical Dictionary for Regulatory Activities (MedDRA).
- 9. Sub conditions include Cardiac, Gastrointestinal, Metabolism and Nutrition, Psychiatric, Renal and Urinary, and Nervous system Conditions.
- 10. Summarised by Ingredient combinations.
- 11. Dispensation information (dates and number of tablets dispensed and returned).

#### 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

## 7.1.1. Endpoint / Variables

The primary objective of the study is to demonstrate the non-inferior antiviral activity of CAB LA + RPV LA every two months (Q2M) compared to a BIK single tablet regimen administered once daily over 12 months in suppressed HIV-1 infected antiretroviral therapy (ART)-experienced participants. The primary endpoint is proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL as per Food and Drug Administration (FDA) Snapshot algorithm at Month 12 (OLI and BIK)/Month 11 (D2I).

## 7.1.2. Summary Measure

Difference between the two treatment groups (Q2M – BIK) in the proportion of participants with HIV-RNA ≥50 c/mL at Month 12 (OLI and BIK)/Month 11(D2I) (as defined by the US FDA snapshot algorithm) and its two-sided 95% confidence interval will be produced. Note for the Q2M arm, primary endpoint data from the Q2M OLI subjects at Month 12 and data from the Q2M D2I subject at Month 11 will be combined for demonstration of non-inferiority.

#### 7.1.3. Population of Interest

The primary efficacy analyses will be based on the modified Intent-To-Treat Exposed (mITT-E) population, unless otherwise specified.

## 7.1.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the Snapshot algorithm, HIV-RNA  $\geq$  50 copies/mL is determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest.

Participants without evaluable HIV-RNA data for the visit of interest and who discontinue treatment for reasons not related to adverse event while having HIV-1 RNA  $\geq$  50 copies/mL at time of discontinuation, or who change study treatment not permitted per protocol prior to the analysis window are classified as having HIV-RNA  $\geq$  50 copies/mL.

A "while on-treatment" strategy will be implemented when a Q2M subject becomes pregnant on study but is allowed to continue. Viral load data collected after confirmed pregnancy will not be evaluated for summary tables and statistical analysis in the primary analysis. Additional sensitivity analysis including all observed data may be performed to assess consistency. See Appendix 13: Data Handling for Pregnant Subjects for details.

## 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 7.1.5.1. Statistical Methodology Specification

#### **Primary Statistical Analysis**

#### **Endpoint / Variables**

• Proportion of participants with plasma HIV-RNA greater than or equal to 50 copies/mL at Month 12 (OLI and BIK)/Month 11 (D2I) per Snapshot algorithm for the mITT-E population.

#### **Snapshot Dataset**

- Virologic outcome ("HIV-RNA <50" or "≥50 c/mL") per Snapshot algorithm is determined by the
  last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest
  (refer to analysis window defined in Section 16.3). In addition, participants who discontinue for
  reasons not related to adverse event with on-treatment HIV-1 RNA result at the time of
  discontinuation ≥50 c/mL or who change study treatment not permitted per protocol during
  Maintenance Phase before the analysis visit are classified as 'HIV-RNA ≥50 c/mL'.</li>
- Full details of the Snapshot algorithm are provided in Appendix 9: Snapshot Algorithm Details

#### **Model Specification**

• The primary efficacy endpoint will be analysed using a stratified analysis with Cochran-Mantel-Haenszel (CMH) weights, adjusting for the randomization strata BMI (<30, ≥30 kg/m²) and Gender at Birth (female, male)

- The CMH estimate of the adjusted treatment difference will be calculated as a weighted average of strata-specific estimates of the treatment difference calculated within each stratum as follows:
  - o Baseline BMI < 30 kg/m<sup>2</sup> and Male Gender at Birth
  - o Baseline BMI < 30 kg/m<sup>2</sup> and Female Gender at Birth
  - o Baseline BMI ≥ 30 kg/m² and Male Gender at Birth
  - o Baseline BMI ≥ 30 kg/m² and Female Gender at Birth
- If  $n_k$  is the number of CAB LA + RPV LA (Q2M) treated participants,  $m_k$  is the number of BIK arm treated participants, and  $N_k = n_k + m_k$  is the total number of participants in the  $k^{th}$  stratum, then the CMH estimate is given by

$$\hat{d}_{cmh} = \frac{\sum W_k \hat{d}_k}{\sum W_k}$$

where

$$W_k = \frac{n_k m_k}{N_k}$$

are CMH weights and treatment arms, p<sub>Q2M</sub>-

 $\hat{d}_k$  are estimates of the differences in proportions between the two p<sub>BIK</sub>, for the  $k^{\text{th}}$  stratum.

The corresponding two-sided 95% CI will be calculated as

$$\hat{d}_{cmh} \pm 1.96 \times \sqrt{\hat{\text{var}}(\hat{d}_{cmh})}$$

where the variance estimator [Sato, 1989] consistent in both sparse data and large strata is given below

$$\operatorname{var}(\hat{d}_{cmh}) = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum n_k m_k / N_k\right)^2} = \frac{\hat{d}_{cmh}(\sum P_k) + \sum Q_k}{\left(\sum W_k\right)^2}$$

where

$$P_k = \frac{n_k^2 y_k - m_k^2 x_k + n_k m_k (m_k - n_k)/2}{N_k^2}$$

$$Q_k = \frac{x_k (m_k - y_k) / N_k + y_k (n_k - x_k) / N_k}{2}$$

with  $x_k$  and  $y_k$  corresponding to the number of participants with Plasma HIV-1  $\geq$  50 c/mL at Month 12 (OLI and BIK)/Month 11 (D2I) per FDA Snapshot for the Q2M and BIK arm, respectively, for the *kth* stratum.

#### Model Results Presentation

- Adjusted CMH estimate of the difference in the proportion of participants with "HIV-1 RNA ≥50" between each treatment group (Q2M – BIK) and corresponding 95% confidence interval.
- Non-inferiority will be concluded if the upper bound of the two-sided 95% confidence interval (CI) for the CMH adjusted difference in proportion of participants with 'HIV-1 RNA≥50' in the CAB LA + RPV LA (Q2M) group minus proportion of participants with 'HIV-1 RNA≥50' in the BIK group is less than 4%.
- If the analysis shows non-inferiority, then a superiority hypothesis will be tested at the two-sided 5% level of significance. Superiority favoring CAB LA + RPV LA (Q2M) will be declared if the upper limit of the confidence interval is below 0% for the mITT-E population analysis. If superiority is declared, the p-value for superiority will also be calculated.

### Subgroup Analyses

- Treatment Heterogeneity across randomization strata:
  - The weighted least squares chi-squared statistic [Fleiss, 1981] will be used to test for one-way homogeneity across the levels of each categorical variable, with each categorical variable considered separately.
  - Following Lui and Kelly [Lui, 2000] ½ will be added to each cell in any strata for which
    the stratum-specific rate estimates of either p<sub>Q2M</sub> or p<sub>BIK</sub> are zero or one, and tests will
    be one-sided.
  - Any heterogeneity found to be statistically significant will be explored and if necessary, results will be reported for each level of the categorical variable. Investigation of heterogeneity will be confined to the primary endpoint. Tests of homogeneity will be assessed at the one-sided 10% level of significance.



## Per-Protocol population analysis:

To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-Protocol population and compared for consistency with the results from the primary mITT-E population analysis.

- All Data as Observed:
  - This analysis will include all observed data including those collected after confirmed pregnancy, in the mITT-E population.
- Efficacy Sensitivity:
   This analysis will be based on the ITT-E population at Month 12.

## 7.2. Secondary Efficacy Analyses

## 7.2.1. Endpoint / Variables

The key secondary efficacy endpoint is proportion of participants with plasma HIV-1 RNA <50 c/mL (c/mL) at Month 12 (OLI and BIK)/Month 11(D2I) using the FDA Snapshot algorithm.

Other secondary efficacy endpoints are listed below:

- Proportion of participants with plasma HIV-1 RNA <50 c/mL (c/mL) at Month 6 (OLI and BIK)/Month 5 (D2I).
- Proportion of participants with plasma HIV-1 RNA ≥50 c/mL (c/mL) at Month 6 (OLI and BIK)/Month 5(D2I)
- Proportion of participants with protocol-defined confirmed virologic failure (CVF) through Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I).
- Changes from Baseline in viral load and CD4+ cell count over time including Month 6 and Month 12 (OLI and BIK)/Month 5 and Month 11 (D2I)

## 7.2.2. Summary Measure

Binary endpoints: difference in the proportion of participants with HIV-RNA  $\geq$  50 c/mL (or < 50 c/mL) as defined by the US FDA snapshot algorithm at specified time point between treatment groups (Q2M – BIK) will be produced.

Continuous endpoints (e.g. CD4+ cell count): descriptive summary statistics per GSK data standards will be produced.

## 7.2.3. Population of Interest

The secondary efficacy analyses will be based on the Intent-to-Treat Exposed (ITT-E) population, unless otherwise specified. Note in the Month 12 analysis, mITT-E will be used in summary tables.

## 7.2.4. Strategy for Intercurrent (Post-Randomization) Events

As defined by the snapshot algorithm, only participants with last available HIV-1 RNA measurement less than 50 c/mL while the participant is on treatment within the analysis visit window of interest are classified as HIV-1 RNA < 50 c/mL.

A "while on-treatment" strategy will be implemented as described in Section 7.1.4. Same approach will be applied to efficacy tables for protocol-defined confirmed virologic failure (CVF) and CD4+ cell count. Data after confirmed pregnancy will not be evaluated for the summary tables unless otherwise noted, but will be included in the listings if applicable.

## 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

## 7.2.5.1. Statistical Methodology Specification

## **Key Secondary Statistical Analysis**

#### **Endpoint / Variables**

- Proportion of participants with plasma HIV-RNA < 50 copies/mL at Month 12(OLI and BIK)/Month11(D2I) per Snapshot algorithm for the mITT-E population.
- Proportion of participants with plasma HIV-RNA < 50 copies/mL at Month 6(OLI and BIK)/Month 5(D2I) per Snapshot algorithm for the ITT-E population.</li>
- Proportion of participants with plasma HIV-RNA ≥50 copies/mL at Month 6(OLI and BIK)/Month 5(D2I) per Snapshot algorithm for the ITT-E population.

#### **Snapshot Dataset**

- Virologic outcome ("HIV-RNA <50" or "≥50 c/mL") per Snapshot algorithm is determined by the last available on-treatment HIV-1 RNA measurement within the analysis visit window of interest (please refer to analysis window defined in Section 16.3). In addition, participants who discontinue for reasons not related to adverse event with on-treatment HIV-1 RNA result at the time of discontinuation ≥50 c/mL or who change study treatment not permitted per protocol during Maintenance Phase before the analysis visit are classified as 'HIV-RNA ≥50 c/mL'.</p>
- Full details of the Snapshot algorithm are provided in Appendix 9: Snapshot Algorithm Details

#### **Model Specification**

As specified in Section 7.1.5.1, with outcome being "HIV-1 RNA <50 c/mL" or "HIV-1 RNA ≥50 c/mL"</li>

#### **Model Results Presentation**

- Adjusted CMH estimate of the difference in the proportion of participants with 'HIV-1 RNA <50' or with 'HIV-1 RNA ≥50' between two treatment groups (Q2M BIK) and corresponding 95% confidence interval.</li>
- Non-inferiority will be concluded if the lower bound of the two-sided 95% confidence interval (CI) for the CMH adjusted difference (Q2M BIK) in proportion of participants with 'HIV-1 RNA <50' is greater than -12% at Month 12 (OLI and BIK)/Month 11 (D2I).</li>

#### **Subgroup Analyses**

Treatment Heterogeneity across randomization strata at Month 12 (OLI and BIK)/Month 11 (D2I)
 As specified in Section 7.1.5.1, with outcome being "HIV-1 RNA <50 c/mL" or "HIV-1 ≥50 c/mL"</li>

## Sensitivity and Supportive Analyses

Per-Protocol population analysis:

To assess the impact of important protocol deviations, statistical analysis will be repeated using the Per-Protocol population and compared for consistency with the results from the primary ITT-E population analysis. Note for Month 12, PP population is based on the mITT-E population.

- All Data as Observed:
  - This analysis will include all observed data including those collected after confirmed pregnancy, in the ITT-E population. Note for Month 12, this analysis will be based on the mITT-E population.
- Efficacy Sensitivity:
   This analysis will be based on the ITT-E population at Month 12.







## 8. SAFETY ANALYSES

The safety analyses will be based on the Safety population, unless otherwise specified. A "while on-treatment" strategy which considers data collected after confirmed pregnancy non-evaluable in the Q2M arm will be implemented for selected analysis including clinical laboratory, biomarker, and metabolic analysis. See Appendix 13: Data Handling for Pregnant Subjects for details. Note for safety-related reporting including adverse events and ECG, all observed data will be included.

## 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. Table 3 below provides an overview of the planned analyse with further details of data displays provided in Appendix 15: List of Data Displays.

Table 3 Overview of Adverse Events Analyses

| Endpoint | | Al | osolu | te | Change from Maintenance<br>Baseline | | | | | | Max Post<br>Maintenance Baseline | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Stats<br>Analysis | Summary | | Individual | | Summary | | Individual | |
| | Т | F | F | L | Т | Τ | F | F | L | Т | F | F | L |
| Exposure | | | | | | | | | | | | | |
| Extent of Exposure[1] | Υ | | | <b>Y</b> [2] | | | | | | | | | |
| Adherence to Dosing Schedule [1] | Y | | | | | | | | | | | | |
| Dosing Errors and IP<br>Device Malfunctions | | | | Υ | | | | | | | | | |
| Injection Needle | | | | | | | | | | | | | |
| Length and Gauge | Υ | | | | | | | | | | | | |
| Adverse Events[3] | | | | | | | | | | | | | |
| All AEs by SOC and PT | Υ | | | | | | | | | | | | |
| All AEs by SOC, PT and Toxicity | Υ | | | | | | | | | | | | |
| All Drug-Related AEs by SOC and PT | Y | | | | | | | | | | | | |
| All Drug-Related AEs<br>by SOC, PT and<br>Toxicity | Υ | | | | | | | | | | | | |
| Common AEs by frequency [5] | Υ | <b>Y</b> [6] | | | | | | | | | | | |
| Common Grade 2-5<br>AEs [5] by frequency | Υ | | | | | | | | | | | | |

| Endpoint | Absolute | | | | Change | Max Post<br>Maintenance Baseline | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Stats<br>Analysis | Summary | | Individual | | Summary | | Individual | |
| | Т | F | F | L | T | Τ | F | F | L | T | F | F | L |
| Drug-related Grade 2-5 AEs | Υ | | | | | | | | | | | | |
| All AEs | | | | <b>Y</b> [4] | | | | | | | | | |
| Serious and other significant adverse events | | | | | | | | | | | | | |
| All SAEs by SOC and PT | Y | | | | | | | | | | | | |
| Reason for<br>Considering as a<br>Serious Adverse<br>Event (FDA) | | | | Y | | | | | | | | | |
| All Drug-Related SAEs by SOC and PT | Y | | | | | | | | | | | | |
| Fatal SAEs | | | | Υ | | | | | | | | | |
| Non-Fatal SAEs | Υ | | | Υ | | | | | | | | | |
| Drug-related non-fatal SAEs | Y | | | | | | | | | | | | |
| AEs Leading to<br>Withdrawal/Permanent<br>Discontinuation of IP | Y | | | Y | | | | | | | | | |
| Common Non-serious<br>AEs by SOC and PT | Υ | | | | | | | | | | | | |
| Subjects and Number<br>of occurrences of<br>SAEs, Fatal SAEs,<br>and Drug-related<br>SAEs | Y | | | | | | | | | | | | |
| AESI | | | | | | | | | | | | | |
| Depression, Suicidal<br>and Self-Injury AEs by<br>Prior History | Y | | | | | | | | | | | | |
| AESI by SOC and PT | Υ | | | | | | | | | | | | |
| Characteristics of AESI | Υ | | | | | | | | | | | | |
| Syncope and Presyncope AE | Υ | | | | | | | | | | | | |
| Suicidality assessment | | | | | | | | | | | | | |
| PSRAE | | | | <b>Y</b> [7] | | | | | | | | | |
| Endpoint | | Al | bsolu | te | Change | | Main<br>eline | itena | ince | Main | Max<br>tenan | Post<br>ce Bas | seline |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | /idual | Stats<br>Analysis | Sum | mary | Indi | vidual | Sum | mary | Indiv | vidual |
| | T | F | F | L | T | T | F | F | L | T | F | F | L |
| Columbia suicidality (eC-SSRS) | Y | | | | | | | | | | | | |
| Injection Site Reaction | n Adve | erse E | ve <b>nts</b> | [12] | | | | | | | | | |
| ISR AEs (Event-Level) [17] | Y | | | | | | | | | | | | |
| ISR AEs (Subject-<br>Level) [18] | Υ | | | | | | | | | | | | |
| ISR AEs (Subject-<br>Level) by Visit and<br>Severity | Y | Υ[19] | | | | | | | | | | | |
| Maximum ISR AE<br>Grade by Needle<br>Length [21] | Y | | | | | | | | | | | | |
| Laboratory: Chemistry | / and | Hemat | ology | 1 | | | | | | | | | |
| Clinical Chemistry | | | | | | Υ | | | | Υ | | | |
| Lipids | | | | | | Υ | | | | | | | |
| NCEP shifts in lipids | | | | | | | | | | Y[8] | | | |
| Hematology | | | | | | Υ | | | | Υ | | | |
| CCI | | | | | | | | | | | | | |
| Laboratory: Urinalysis | (rega | rdles | of fa | sting | status) | | | | | | | | |
| Urine Dipstick | Υ | | | | | | | | | | | | |
| Urine Concentration | | | | | | Υ | | | | | | | |
| Proteinuria | | | | | | | | | | Y[8] | | | |
| Laboratory: Hepatobil | iary | | | | | | | | | | | | |
| Liver Assessment | | | | Y[14] | | | | | | | | | |
| Hepatobiliary<br>Abnormality criteria | Υ | | | Υ | | | | | | | | | |
| Liver Chemistries | | | | Y[11] | | | | | | | Y[9] | | |
| Laboratory: Biomarke | rs | • | | • | | | | | | | • | | |
| Bone markers | | | | | Υ | Υ[10] | | | | | | | |
| Renal markers<br>CCI | | | | | Y | Υ[10] | | | | | | | |
| HOMA-IR, insulin and<br>HbA1c | | | | | Y[16] | Υ | | | | | | | |
| ECG | | | | | | | | | | | | | |
| ECG findings | Υ | | | Υ | | | | | | | | | |

| Endpoint | Absolute | | | | Change | | Main<br>eline | Max Post<br>Maintenance Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | vidual | Stats<br>Analysis | Sum | mary | Indi | vidual | Summary | | Indiv | idual |
| | T F F L | | T | T | F | F | L | T | F | F | L | | |
| ECG values | | | | Y[22] | | Υ | | | | | | | |
| QTC values by<br>Category | Υ | | | | | Υ | | | | | | | |
| Other | | | | | | | | | | | | | |
| Vital Signs (BP, HR, temp) | | | | Υ | | Υ | | | | | | | |
| Weight, Height and<br>BMI | Υ | | | Υ | | Υ | | | | | | | |
| Waist Circumference<br>and Hip<br>Circumference | Y | | | Y | | Y | | | | | | | |
| CCI | | | | | | | | | | | | | |
| Tanita Scale Assessments (Body Fat Percentage, Bone Mineral Mass, Muscle Mass, Total Body Water Percentage) | Y | | | Y | | Y | | | | | | | |
| Abacavir HSR | | | | Y[13] | | | | | | | | | |
| Participants who became Pregnant | | | | Υ | | | | | | | | | |
| Patient Profiles | | | | Y <sup>[20]</sup> | | | | | | | | | |
| Metabolic Syndrome | Υ | | Υ | Υ | | Υ | | | | | | | |

### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Stats Analysis = Displays related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- Refer to Section 16.6.2 and Section 16.6.4 for defining extent of exposure and adherence to dosing intervals.
- Includes reason for any dose change/interruption.
- For AEs reported more than once by a participant, the most severe intensity will be included. Separate summary tables including and excluding injection site adverse reactions.
- 4. Listing of all AEs including verbatim text and preferred term, and listing of subject numbers for individual AEs.
- Common AEs are those with ≥5% incidence in Q2M or BIK summarised by frequency.
- Plots of incidence rates and relative risk with 95% CI for Q2M vs.BIK.
- Four PSRAE listings: Event and Description (Section 1 and Section 2), Possible Cause (Section 3), Section 4 and Section 5 - Section 8.

- Shift table summarising Maintenance Baseline (Day 1) vs. maximum Maintenance Phase result.
- Scatter plot of baseline vs. maximum post-baseline for ALT and BILT. Scatter plot of maximum ALT vs. maximum Bilirubin.
- Bone markers: Bone-specific alkaline phosphatase, procollagen type 1 N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin, 25 hydroxy-Vitamin D. Renal markers: Cystatin C; Beta-2-Microglobulin; Retinol Binding Protein (RBP).
- 11. For subjects meeting hepatobiliary lab abnormality criteria.
- Repeat for CAB/RPV, CAB, RPV respectively.
- 13. Separate listings for exposure to abacavir, history of drug allergies, family conditions, skin rash, symptoms, vital signs, individual symptoms and diagnostic category assignment. If no hypersensitivity to abacavir is observed, then only one blank listing will be provided for the exposure to abacavir.
- Separate listings for event reporting, RUCAM score, biopsy, imaging, substance use and medical conditions.
- Statistical analysis will be performed for HOMA-IR.
- Event-level summary: Percentages based on total number of ISR events including distribution of grade, duration, and event characteristics.
- Subject-Level summary: Characteristics of ISR AE (Overall and by Common ISRs); Percentage based on number of participants; Includes distribution of grade and max grade, event characteristics, number of events per subject, rate of number of events per injection visit.
- A corresponding plot for all grades and a separate plot for grade 3-5 events will be produced.
- 20. Patient profiles are not planned but can be produced post hoc, as necessary.
- Please refer to Section 5.4 for derivation of needle length used in this summary.
- 22. For subjects with any value of potential clinical importance.

# 8.2. Adverse Events of Special Interest Analyses

Adverse events of special interest (AESI) are determined for CAB and/or RPV based on pre-clinical and clinical experience, along with information for the Integrase Inhibitor class of HIV medications and RPV safety profile. Table 4 shows the currently identified AESI, drug(s) of Interest and the reasons for inclusion. Changes to the MedDRA dictionary may occur between the start of the study and the time of reporting and/or emerging data from ongoing studies may highlight additional adverse events of special interest, therefore the list of terms to be used for each event of interest and the specific events of interest will be based on the safety review team (SRT) agreements in place at the time of reporting.

A summary by system organ class and preferred term will be provided for each of AESI. The characteristics of event occurrences during the maintenance phase will be summarized for AESIs. For Depression, anxiety and suicidal ideation/behaviour AESI, a summary by system organ class, maximum DAIDS toxicity grade and prior history of suicidal ideation will be provided.

The details of the current planned grouping, including Standardized MedDRA Query (SMQ) values (as applicable), and planned displays are provided in Appendix 11: Identification of Adverse Events of Special Interest (AESI) and Appendix 15: List of Data Displays.

Table 4 Adverse Events of Special Interest

| Adverse Events of Special Interest | Drug(s) of<br>Interest | Reason for Inclusion |
|---|---|---|
| Hepatic Safety Profile: Assessment of Risk of hepatoxicity | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Hyperglycemia | CAB | Class, Regulatory Interest |
| Hypersensitivity Reactions (HSR) | CAB | Class, Regulatory Interest,<br>Occurs in HIV population |
| Rash | RPV | Class, Regulatory Interest,<br>Occurs in HIV population |
| Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses | RPV | Non-clinical, Clinical,<br>Regulatory Interest |
| Suicidal Ideation/Behaviour | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Depression | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Bipolar Disorder | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Psychosis | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Mood Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Anxiety | CAB+RPV | Clinical, Class, Regulatory<br>Interest |
| Sleep Disorders | CAB+RPV | Clinical, Class, Regulatory<br>Interest, More prevalent in<br>HIV population |
| Injection Site Reactions (ISR) from Study Drug Injections [1] | CAB+RPV | Clinical |
| Seizures and Seizure-like Events | CAB | Clinical, Regulatory Interest |
| Weight Gain | CAB | Clinical, Class |
| Rhabdomyolysis | CAB | Clinical, Class |
| Pancreatitis | CAB | Clinical, Therapeutic Area,<br>More prevalent in HIV<br>population |

| Adverse Events of Special Interest | Drug(s) of Interest Reason for Inclus | |
|---|---|---|
| Impact on Creatinine | CAB+RPV | Regulatory Interest,<br>Therapeutic Area, More<br>prevalent in HIV population |
| Safety in Pregnancy | CAB | Regulatory Interest, Class |
| NOTE: [1] A separate analysis will be performed for ISRs from s | study drug injections as d | lescribed in Section 8.2.1 |

# 8.2.1. Analyses for Injection Site Reaction Adverse Events

Injection Site Reaction (ISR) adverse events of interest are those from study drug injections. For the summary of ISR adverse events by visit and maximum severity (overall and by common ISRs): ISRs will be assigned based on onset date to the most recent planned IM injection visit prior or equal to the AE onset date.

Maximum grade at each visit will be derived as the maximum grade among ISRs assigned to the particular visit, with consideration for whether the summary applies to a particular preferred term (vs. across preferred terms), associated to CAB and/or RPV, or stratification by subgroup (such as needle length, refer to Section 5.4.2).

ISRs (based on investigator discretion) from study drug injections will be attributed to the causal agent (CAB vs. RPV) when this can be determined specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If the causal agent cannot be determined in cases where both drugs are given on one side or the ISR is reported non-specifically, then the attribution to a specific causal agent will remain unknown.

Common ISR adverse events during the Maintenance Phase are defined by MedDRA preferred terms including injection site pain, injection site induration, injection site nodules and preferred terms of any other ISR with ≥5% participants in the Q2M arm. The same set of common terms will be applied to 'overall' (CAB and/or RPV), CAB alone, RPV alone.

ISRs will be attributed to the needle length specifically based on the side of injection administration and the side of the reported ISR (as collected in the eCRF). If the needle length cannot be determined due to both drugs given on the same side with different needle lengths, then the attribution to a needle length will remain unknown.

# 8.3. Clinical Laboratory

Laboratory evaluations including the analyses of chemistry laboratory tests, hematology laboratory tests, urinalysis, and liver function tests will be based on GSK Core Data Standards.

For women who became pregnant on study, a data listing for selected parameters including the following will be provided. Additional parameters of interest may also be listed if applicable.

Clinical Chemistry: Creatinine, GFR, Glucose, HCG

Hematology: HbA1C, Hemoglobin, Hematocrit, Mean Corpuscular Volume, Platelets, Erythrocytes, Lymphocytes, Neutrophils, Basophils, Monocytes, Eosinophils

Immunology: CD4+ cell count, CD8+ cell count, CD4/CD8 cell count ratio, CD4/Lymphocytes, CD8/Lymphocytes

Urinalysis: Albumin/Creatinine, Glucose, Ketones, Occult Blood, Protein, Protein/Creatinine, Erythrocytes

# 8.4. Biomarker Analyses

Biomarker analysis (renal, bone, inflammation) will not be performed at the Month 6 interim analysis, and will only be performed when all expected data through Month 12 (OLI and BIK)/Month 11 (D2I) has been received from the laboratory. Statistical estimates for each planned visit will be provided in the Month 12 primary analysis using the MMRM model as describe in the below sections unless otherwise noted. The details of the planned displays are in Appendix 15: List of Data Displays.

### 8.4.1. Bone Biomarkers

### **Statistical Analyses**

## **Endpoints**

- Change from Maintenance Baseline (Day 1) in the following bone markers at Month 6 (OLI and BIK)/Month 5 (D2I) and at Month 12 (OLI and BIK)/Month 11 (D2I):
  - Bone-specific alkaline phosphatase
  - Procollagen type 1 N-propeptide
  - Type 1 collagen cross-linked C-telopeptide
  - Osteocalcin
  - ° 25 hydroxy-Vitamin D

### **Covariates**

- Baseline Value (continuous, log-transformed)
- Gender at Birth (male, female)
- Baseline BMI(<30 kg/m², >=30 kg/m²)
- Age (Continuous)
- Race (White, Black/African American, Other)
- Smoking Status (Never, Former, Current)
- Vitamin D use (Yes vs no)

### **Data Handling**

OC (Observed Case) dataset will be used.

### **Model Specification**

- Analysis values will be log-transformed (including the baseline value).
- The change in the log-transformed data from Maintenance baseline (i.e. log(value/ baseline value) or log(value) – log(baseline value)) for each bone marker will be analysed for the comparison between the two treatment arms.
- MMRM (Mix Model Repeated Measures) model with the observed margins (OM) option within PROC MIXED in SAS will be used including treatment group plus the above covariates, with visit as the repeated factor.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- No assumptions about the correlations between a subject's values will be made (the correlation
  matrix for within-subject errors will be unstructured). This will be estimated by treatment group by
  specifying "type=UN" and "group=treatment" options in the SAS MMRM models.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS. Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure if needed.
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model). Estimates and 95% confidence intervals will be produced for each visit.

### **Model Checking & Diagnostics**

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- Distributional assumptions underlying the model used for analysis may be examined by obtaining a
  normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e.
  checking the normality assumption and constant variance assumption of the model respectively) to
  gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriately transformed data.

# **Model Results Presentation**

- For each treatment: Adjusted geometric means (for ratio to Maintenance BL) and 95% CI. Exponential transformation on the estimates from the MMRM model (based on the log-transformed data) will reflect the mean ratio of values post-baseline vs. Maintenance BL for each treatment arm. This ratio can then be translated into percent change from maintenance baseline (Day 1) (e.g. the ratio bb<sub>M12</sub>/bbb<sub>bl</sub> = 1.3 can be translated into 30% increase from baseline).
- For treatment comparison: Adjusted geometric mean ratio between the two treatment groups (Q2M/BIK), 95% CI and *p*-value. This ratio can then be translated into percent comparisons in the ratio (value/baseline value) between Q2M vs. BIK (e.g. Q2M/BIK = 1.2 can be translated into 20% higher in the Q2M change from baseline ratio compared with BIK).

 Interactions between treatment and each of the covariates will not be assessed but may be explored post hoc.

### **Sensitivity Analyses**

Not applicable

# Subgroup Analyses

Not applicable

## 8.4.2. Renal Biomarkers

## **Statistical Analyses**

### **Endpoints**

- Change from Maintenance Baseline (Day 1) in the following renal markers at Month 6 (OLI and BIK)/Month 5 (D2I) and at Month 12 (OLI and BIK)/Month 11 (D2I):
  - Cystatin C
  - Retinol Binding Protein (RBP)
  - ° Beta-2-Microglobulin (B2M)

### **Covariates**

- Baseline Value (continuous)
- Gender at Birth (male, female)
- Baseline BMI(<30 kg/m2, >=30 kg/m2)
- Age (continuous)
- Race (White, Black/African American, Other)
- Hypertension (Yes vs no)
- Diabetes (Yes vs no)

### Note:

Hypertension is defined as having a medical history of hypertension or use of medication treating hypertension (current and past).

Diabetes is defined as having a medical history of Diabetes or use of medication treating Diabetes (current and past) or fasting glucose at  $\geq 126$  mg/dL with HbA1c > 6.5% at Day 1.

### **Data Handling**

• OC (Observed Case) dataset will be used.

## **Model Specification**

Same as in Section 8.4.1

### **Model Checking & Diagnostics**

• Same as in Section 8.4.1

### **Model Results Presentation**

Same as in Section 8.4.1

# **Sensitivity Analyses**

Not applicable

### **Subgroup Analyses**

Not applicable



# 8.5. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 15: List of Data Displays.

# 8.5.1. ECG

ECG Values of Potential Clinical Interest are defined as a QTc of > 500 msec or increase from baseline in QTc  $\geq$  60 msec.

## 8.5.2. Metabolic Syndrome

Diagnosis of Metabolic Syndrome is defined as follows per joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Three abnormal findings out of the five risk factors would qualify a person for the metabolic syndrome(waist circumference, triglycerides, HDL, BP and fasting glucose) at each planned time point. See Section 16.6.4 for cutoff details. Percent of subjects diagnosed with metabolic syndrome will be produced. Patient profile as well as listing of clinical diagnosis factors over time may also be provided for those who are diagnosed with metabolic syndrome.

### **Statistical Analyses**

### **Endpoints**

 Proportion of subjects with metabolic syndrome at Month 6 (OLI and BIK)/Month 5 (D2I) and at Month 12 (OLI and BIK)/Month 11 (D2I)

### Covariates

- Baseline CD4+ cell count (continuous)
- Gender at Birth (male, female)
- Baseline BMI(<30 kg/m<sup>2</sup>, >=30 kg/m<sup>2</sup>)
- Age (35-<50, >=50, <35 years)
- Race (White, Black/African American, Other)
- Smoking Status (Never, Current, Former)
- Hypertension (Yes vs no)
- Baseline Triglyceride (High vs. Normal)
- Baseline HDL (Low, High vs Normal)
- Baseline HOMA-IR (2 to <3, 3 to <4, >=4 vs <2)

Note: Hypertension is defined as having a medical history of hypertension or use of medication treating hypertension (current and past)

### **Data Handling**

OC (Observed Case) dataset will be used.

### **Model Specification**

 A logistic regression model will be performed on the proportion of subjects with metabolic syndrome at Month 6(OLI and BIK)/5(D2I) and at Month 12(OLI and BIK)/11(D2I) adjusting for the covariates as above.

### **Model Checking & Diagnostics**

- Upon delivery of data, an assessment regarding the amount of missing data will be made. If the
  amount of missing outcome data considered as a result of other impacts such as COVID-19 is
  substantial, the logistic regression analysis may not be performed.
- If the percent of subjects are below 5% of the total number of subjects (observed data), or if
  complete or quasi-complete separation is observed in the data, then the analysis may not be
  performed.

| Statistical Analyses |
|---|
| Model Results Presentation |
| <ul> <li>Odds ratios, confidence intervals and p-values will be presented for all covariates specified in the<br/>model.</li> </ul> |
| Sensitivity Analyses |
| Not applicable |
| Subgroup Analyses |
| Not applicable |

# 8.5.3. Anthropometric profile

Descriptive summaries will be provided for the following parameters to evaluate the metabolic profile of subjects:

- Weight, Height and BMI
- Waist circumference
- Hip circumference
- CC
- CCI
- Tanita scale parameters (total body fat percent, total body water percent, muscle mass, and bone mineral mass)

Subjects with cosmetic procedures of the torso/thighs (exclude face/neck) including but not limited to liposuction/liposculpture/implants will be excluded from the above summary statistics at Month 12 (OLI and BIK)/Month 11 (D2I).

Data collected after initiation of lipid-modifying agents on treatment will be considered non-evaluable for anthropometric profile summaries (while on-treatment strategy).

### 8.5.4. HOMA-Insulin Resistance

HOMA-Insulin Resistance analysis will only be performed when all expected data through Month 12 (OLI and BIK)/Month 11 (D2I) has been received from the laboratory. Statistical estimates for each planned visit will be provided in the Month 12 primary analysis using the MMRM model as describe in the below sections unless otherwise noted. The details of the planned displays are in Appendix 15: List of Data Displays.

# Statistical Analyses

### **Endpoints**

 Change from baseline in HOMA-IR at Month 6 (OLI and BIK)/Month 5 (D2I) and at Month 12 (OLI and BIK)/Month 11 (D2I)

Note: the following subjects will be excluded from the statistical analysis:

- diabetic or have taken an anti-diabetic medication up to screening
- fasting glucose >126mg/dl and HbA1C >6.5% at Day 1
- have had a cosmetic procedure including liposuction/liposculpture of the thighs, buttocks, hips and/or

#### abdomen

#### Covariates

## Statistical Analyses

- Baseline Value (continuous)
- Gender at Birth (male, female)
- Baseline BMI(<30 kg/m<sup>2</sup>, >=30 kg/m<sup>2</sup>)
- Age (Continuous)
- Race (White, Black/African American, Other)
- Smoking Status (Never, Current, Former)
- Hypertension (Yes vs no)

Note: Hypertension is defined as having a medical history of hypertension or use of medication treating hypertension (current and past)

### Data Handling

• OC (Observed Case) dataset will be used.

# **Model Specification**

Same as in Section 8.4.1

## **Model Checking & Diagnostics**

Same as in Section 8.4.1

### **Model Results Presentation**

Same as in Section 8.4.1

# **Sensitivity Analyses**

- Logistic regression models will be performed on the proportion of subjects with HOMA-IR >=2, >=3
  or >=4 at Month 12(OLI and BIK)/11(D2I) adjusting for the same covariates as specified in the
  MMRM analysis (without visit or interaction terms and without log transformation for the baseline
  value). Odds ratios, confidence intervals and p-values will be presented for all covariates specified in
  the model.
- Upon delivery of data, an assessment regarding the amount of missing data will be made. If the
  amount of missing HOMA-IR outcome data considered as a result of other impacts such as COVID19 is substantial, the logistic regression analysis may not be performed.
- If the percent of subjects above any of the cutoffs are below 5% of the total number of subjects (observed data), or if complete or quasi-complete separation is observed in the data, then the analysis may not be performed.

## Subgroup Analyses

Not applicable

# 9. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Not applicable.

## 10. PHARMACOKINETIC ANALYSES

PK data collected for pregnant participants and at withdrawal visits for all subjects will be listed given data availability. Other PK samples are put to storage and there is no planned PK analysis at the time of the interim or the primary analysis. Future amendment will be made if pharmacokinetic data are to be explored further in the future.

# 11. PHARMACODYNAMIC (AND / OR BIOMARKER) ANALYSES

Not applicable.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

There is no plan for PK/PD analysis for the interim or the Month 12 primary analysis. Analysis details will be provided in future amendments if necessary.

# 13. HEALTH OUTCOMES ANALYSIS

# 13.1. Endpoint/Variables

- Absolute values and Change from baseline in total "treatment satisfaction" score, and individual item scores of the HIV Treatment Satisfaction Status Questionnaire (HIVTSQs) at Month 12 (OLI and BIK)/Month 11 (D2I), and at Month 6(OLI and BIK)/Month 5(D2I).
- Change in treatment satisfaction using the HIV Treatment Satisfaction Change (HIVTSQc) questionnaire at Month 12 (OLI and BIK)/Month 11 (D2I)(or withdrawal).
- Preference for CAB LA + RPV LA every 2 months compared to an oral BIK single tablet regimen as well as reasons for preference at Month 12 (OLI)/Month 11 (D2I).
- Change from Month 2(OLI)/Month 1(D2I) in Dimension scores (e.g., "Bother of ISRs", "Leg movement", "Sleep", and "Acceptance of ISRs") and in individual item

scores assessing pain during injection, anxiety before and after injection, willingness to be injected in the future and overall satisfaction with mode of administration over time using the Perception of injection questionnaire (PIN) at Month 12 (OLI and BIK)/Month 11 (D2I), and at Month 6(OLI and BIK)/Month 5(D2I).



# 13.2. Summary Measure

Mean treatment difference (Q2M – BIK) in change from day 1 (baseline) at visits of interest for HIVTSQs and HIVTSQc.

Mean change at visits of interest for Change from Month 2(OLI)/Month 1 (D2I) in PIN Dimension and individual item scores.

# 13.3. Population of Interest

The primary health outcomes analyses will be based on the Intent-to-Treat Exposed population, unless otherwise specified. CCI

Note in the Month 12 analysis, mITT-E will be used in summary tables.

# 13.4. Strategy for Intercurrent (Post-Randomization) Events

If a participant discontinues treatment prior to the timepoint of interest such that there is no evaluable on-treatment assessment for the timepoint of interest, the data will not be computed or imputed. Assessment window slotting may be implemented for unscheduled and withdrawal visits per Section 16.3.4.

# 13.5. Statistical Analyses / Methods

| Endpoints | | | 1 | Absolu | ıte | | | Cha | nge f | rom I | <b>//aint</b> e | nance | nce Baseline | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | s Ana | lysis | Sum | mary | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | L | T | F | F | ш | Τ | F | L | T | F | F | L |
| Treatment Satisfaction (OLI and BIK)/Month 1 | | _ | VTSC | (s) at l | Day 1, | Mont | h 6(Ol | LI and | I BIK) | /Mon | th 5(D | 21), Mc | onth 1 | 2 |
| Individual Item<br>Scores by visit | | | | Υ | | | | <b>Y</b> [3] | | | Y | | | |
| Total Treatment<br>Satisfaction Score | | | | Υ | | | | Y | | | Y | | | |
| Treatment Satisfaction Score Change (HIVTSQc) at Day 1, Month 12 (OLI and BIK)/Month 11(D2I) | | | | | | | | | | | | | | |
| Individual Item<br>Scores | | | | Υ | | | | | | | | | | |
| Treatment<br>Satisfaction Score<br>Change | Y | | | Υ | | | | | | | | | | |
| | Treatment Preference for CAB LA + RPV LA every 2 months compared to an oral BIK single tablet regimen as well as reasons for preference | | | | | | | | | | | | | |
| Treatment: Every 2<br>Months vs Daily Oral<br>BIK | | | | Υ | | | | | | | | | | |
| Reasons for<br>Preference | | | | Υ | | | | | | | | | | |
| Perception of Injection<br>5(D2I), Month 12 (OLI | | | | | | | | 1(D2I) | , Mon | th 6(0 | OLI an | d BIK | /Mont | h |
| Individual Item<br>Scores (Anxiety<br>Before, Pain,<br>Satisfaction, Anxiety<br>After, Willingness) | | | | Υ | | | | | | | <b>Y</b> [2] | | | |
| Dimension scores<br>(e.g., "Bother of<br>ISRs", "Leg<br>movement", "Sleep",<br>and "Acceptance of<br>ISRs") | <b>Y</b> [1] | | | Y | | | | | | | <b>Y</b> [2] | | | |
| Individual<br>Questionnaire<br>Scores (21 items) | | | | Υ | | | | | | | | | | |

| Endpoints | | | - | Absolu | ıte | | | Cha | nge f | rom I | //ainte | nance | Base | line |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | | mary | Indivi | dual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | T | F | L | T | F | F | ш | T | F | _ | Τ | F | F | L |
| CCI | | | | | | | | | | | | | | |

#### NOTES:

- Table 1 T = Table, F = Figure, L = Listings, Y = Display generated.
- Table 2 Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Table 3 Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Table 4 Individual = Represents FL related to any displays of individual participant observed raw data.
- Statistical analysis (i.e. p-value) produced only for the acceptance score comparing to Month 2(OLI)/Month 1(D2I).
- 2. Change versus Month 2(OLI)/Month 1(D2I) for PIN.
- 3. Individual items 5 (convenient), 6 (flexible) and 10 (continue).

# 13.5.1. Statistical Methodology Specification

Details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 13.1 will be summarised using descriptive statistics and graphically presented (where appropriate). Observed data will be used for summaries and statistical analysis unless otherwise noted.

### 13.5.1.1. HIVTSQs

| Statistical Analyses |
|---|
| HIVTSQS |
| Endpoints |
| Change from Maintenance Baseline (Day 1) at Month 6(OLI and BIK)/Month 5(D2I) and at Month 12 (OLI and BIK)/Month 11 (D2I) in: |
| HIVTSQs total treatment satisfaction score |
| <ul> <li>Individual HIVTSQs items 5 (convenience), 6 (flexible), 10 (continue)</li> </ul> |
| Covariates |
| Baseline score(continuous) |
| Gender at Birth (male, female) |

# **Statistical Analyses**

Baseline BMI(<30 kg/m<sup>2</sup>, >=30 kg/m<sup>2</sup>)

Age (<50, >=50 Years)

Race (white, non-white)

# **Model Specification**

- Month 6(OLI and BIK)/Month 5(D2I) Analysis: ANCOVA (analysis of covariance) model will be used for Maintenance Phase data including treatment group plus above covariates.
- Month 12 (OLI and BIK)/Month 11 (D2I) Analysis: MMRM (Mixed Model Repeated Measures) will be used including treatment group plus above covariates. No assumptions will be made about the correlations between subject readings (i.e. the correlation matrix for within-subject errors is unstructured):
- MMRM (Mix Model Repeated Measures) model with the observed margins (OM) option within PROC MIXED in SAS will be used including treatment group plus the above covariates, with visit as the repeated factor.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- No assumptions about the correlations between a subject's value will be made (the
  correlation matrix for within-subject errors will be unstructured). This will be estimated by
  treatment group by specifying "type=UN" and "group=treatment" options in the SAS MMRM
  models.
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS. Akaike's Information Criteria (AIC) will be used to assist with the selection of covariance structure if needed.
- The repeated measures analysis will assume that the treatment difference can vary between visits (i.e. a treatment\*visit interaction will be included in the model). Estimates and 95% confidence intervals will be produced for each visit.

## **Dataset**

 OC (Observed Case) dataset (with data slotting for the withdrawal/unscheduled visits) will be used. see Section 16.3.4 for details. No additional imputations will be used.

# **Model Results Presentation**

- Adjusted means for each treatment group with 95% CI
- Adjusted treatment difference (Q2M-BIK), 95% CI and the associated p-value for difference
- Interaction between treatment and the baseline score

#### 13.5.1.2. HIVTSQc

## Statistical Analyses

### HIVTSQc

# **Endpoint**

Treatment Satisfaction Score (Change) at Month 12 (OLI and BIK)/Month 11 (D2I)

### Covariates

Gender at Birth (male, female)

Baseline BMI( $<30 \text{ kg/m}^2$ ,  $>=30 \text{ kg/m}^2$ )

Age (<50, >=50 Years)

Race (white, non-white)

# **Model Specification**

- An analysis of variance (ANOVA) model will be used with above covariates
- Adjusted point estimates will be derived as LSMEANS using the observed margins (OM)
  option within PROC MIXED in SAS.
- Interactions between treatment and each of the covariates will not be assessed unless the primary endpoint highlights significant interactions. In this situation, the interaction(s) of interest may be assessed and, if necessary, results will be reported in the clinical study report. If interactions are found to be significant (p<0.10), results may be presented separately by subgroup.</p>

### Dataset

 OC (Observed Case) dataset (with data slotting for the withdrawal/unscheduled visits) will be used, see Section 16.3.4 for details. No additional imputations will be used.

### Model Results Presentation

- Adjusted means for each treatment group with 95% CI
- Adjusted treatment difference (Q2M-BIK), 95% CI and the associated p-value for difference

### 13.5.1.3. PIN

### Statistical Analyses

### PIN (Q2M arm only)

### Endpoints

Change from Month 2(OLI)/Month 1(D2I) in the PIN acceptance score at:

- Month 12(OLI)/Month 11(D2I)
- Month 6(OLI)/Month 5(D2I)

### Statistical Test

 The Wilcoxon Signed-Rank Test will be used to evaluable whether the change from Month 2/Month 1 to Month 6(OLI)/Month 5(D2I), and to Month 12(OLI)/Month 11(D2I), respectively, is statistically different from zero based on a two-sided significance level of 0.05. Separate tests will be performed for the change at each time point.

# **Statistical Analyses**

### Dataset

 OC (Observed Case) dataset (with data slotting for the withdrawal/unscheduled visits) will be used. see Section 16.3.4 for details. No additional imputations will be used.

### **Results Presentation**

• Summary statistics at each analysis timepoint and p-value for each comparison.

# 14. VIROLOGY

Given data availability, the virology analyses will mainly use genotype and phenotype data based on plasma sample for CVF population, unless otherwise specified. Summary tables (if applicable) will be based on the mCVF population. Listings will include all CVFs in this study. Additional analyses for HIV-1 resistance may be carried out on peripheral blood mononuclear (PBMC) samples and/or on stored blood samples from relevant time points.

If pre-treatment genotypic/phenotypic results are available from both the central laboratory and Monogram Biosciences, then Monogram assays will take precedence.

Table 5 provides an overview of the planed analyses. Further details of the planned displays are provided in Appendix 15: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Table 5 Overview of Planned Virology Analysis

| Endpoint | | Abs | solute | |
|---|---|---|---|---|
| | Sum | nmary | Indivi | dual |
| | T | F | F | L |
| Genotypic resistance at time of CVF <sup>[1]</sup> | _ | | | |
| Prevalence of Resistance Mutations | <b>Y</b> [2] | | | Y |
| Prevalence of Genotypic Susceptibility | Υ | | | |
| Phenotypic resistance at time of CVF[1] | | | | |
| Prevalence of Phenotype | Y [3] | | | Y |
| Fold Change to CAB, RPV and BIC | Υ | | | <b>Y</b> [4] |
| IN, PR/RT Replication Capacity [5] | | | | Υ |
| Other | | | | |
| Viral load, Genotypic and Phenotypic data for Participants with genotype and/or phenotype data for CVF and non-CVF participants | | | | Υ[4] |
| Net Assessment | Y | | | |

### NOTES:

• T = Table, F = Figure, L = Listing, Y = Yes display generated.

- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual participant observed raw data.
- If less than 5 CVFs are observed during the maintenance phase in the mITT-E population, summary tables
  may not be produced. All data will be provided in listings in this case.
- 1. CVF defined by two consecutive plasma HIV-1 RNA levels ≥200 c/mL after prior suppression to <200 c/mL. The first of these two consecutive visits is defined as 'suspected', and the 2nd is defined as "confirmed". Sample used for resistance testing is taken at the suspected visit, and only tested once virologic failure at a subsequent visit is confirmed. If the test fails with the sample at the suspected visit, it will be reported as 'no data'. □CI</p>
- Number and percentage of participants with INI resistance mutations or major resistance mutations in the classes of NNRTI, NRTI, PI, respectively, as defined in Section 16.6.7.
- Separate outputs by phenotypic susceptibility and by number of drugs to which participants are phenotypic resistant, partially sensitive or sensitive.
- Fold change to CAB,RPV and BIC will be included in the listing for viral load, genotypic and phenotypic data for
  participants with genotype and/or phenotype data for CVF and non-CVF participants.
- 5. IN: integrase; PR: Protease; RT: reverse transcriptase

# 15. REFERENCES

Alberti KGMM et al. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009;120:1640 –1645.

Chan, I. S. F. and Zhang, Z. (1999), "Test-Based Exact Confidence Intervals for the Difference of Two Binomial Proportions," Biometrics, 55, 1202–1209.

Chevat C, Viala-Danten M, Dias-Barbosa C, Nguyen VH. Development and psychometric validation of a self-administered questionnaire assessing the acceptance of influenza vaccination: the Vaccinees' Perception of Injection questionnaire. Health Qual Life Outcomes. 2008 mar 4; 7:21

D'Agostino RB, Vasan RS, Pencina MJ, et al. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

EMA/CHMP/539146/2013, Guideline on the investigation of subgroups in 4 confirmatory clinical trials, 31 January 2019

FDA Guidance for Industry: Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment, Nov 2015

Fleiss J.L. Statistical Methods for Rates and Proportions. 2nd ed. New York: John Wiley; 1981.

Grundy S.M., et al. Executive summary of the third report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). JAMA. 2001;285 (19):2486-2497.

HIVTSQ user guidelines, Health Psychology Research Unit, Royal Holloway, University of London, 2016

Holmes WC, HIV/AIDS-Targeted Quality of Life Instrument 1999.

Kalbfleisch J.D., Prentice R.L. *The Statistical Analysis of Failure Time Data*. 1st ed. New York: John Wiley & Sons; 1980.

Levey AI, Christopher HS, Hocine T, John HE, Harold IF, Tom G, et al. Estimating Glomerular Filtration Rate from Serum Creatinine and Cystatin C. N Engl J Med 2012, 367: 20-29.

Lui K.J., Kelly C. A Revisit on Tests for Homogeneity of the Risk Difference, Biometrics, 2000;56:309-315.

Mary E. Nilsson, Shailaja Suryawanshi, Cristiana Gassmann-Mayer, Sarah, Dubrava, Paul McSorley, and Kaihong Jiang. Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013

Nilsson ME, Suryawanshi S, Gassmann-Mayer C et al, Columbia–Suicide Severity Rating Scale, Scoring and Data Analysis Guide, 2013.

Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. *Am J Psychiatry*. 2007;164:1035–1043.

Ralph B. D'Agostino, Ramachandran S. Vasan, Michael J. Pencina, Philip A. Wolf, Mark Cobain, Joseph M. Massaro, William B. Kannel. 2008. General Cardiovascular Risk Profile for Use in Primary Care (The Framingham Heart Study). Circulation 2008; 117: 743-753.

Sato T. On the variance estimator for the Mantel-Haenszel risk difference. *Biometrics*. 1989;42:311-323.

Wensing AM et al, 2019 Update of the Drug Resistance Mutations in HIV-1, Volume 27 Issue 3 July/August 2019.

# 16. APPENDICES

# 16.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

# 16.1.1. Exclusions from Per Protocol Population

Important protocol deviations leading to exclusion from the Per Protocol population are those deviations which may

- directly impact the efficacy endpoint of HIV-1 RNA; or
- lead to permanent discontinuation of IP/withdrawal and hence indirectly impact the efficacy endpoint by causing data to be missing.

The following criteria define the protocol deviations which, if they occur prior to an analysis timepoint of interest (e.g. Month 12 or Month 6), will lead to exclusion of a participant from the Per-Protocol population for that analysis. Potential protocol deviations leading to exclusion from PP population will be reviewed by the study team to confirm that they meet these criteria. A final review will occur before the clinical database has been frozen for analysis.

A participant meeting any of the following criteria will be excluded from the Per Protocol population **based on case-by-case clinical determination**. Note exclusion category # 2 below will only be applied in the Month 12 analysis. Other categories will be applied in both Month 6 and Month 12 analysis.

| Number | Exclusion Description |
|---|---|
| 01 | Participant deviates from inclusion or exclusion criteria that may significantly affect exposure, response to therapy or participant safety or that are fundamentally inconsistent with the intended study population, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| 02* | For Month 12 analysis only: Participant has non-compliance with IP (including IM dosing errors) or took/received incorrect IP (i.e., other than the one to which they were randomized) up to an analysis timepoint of interest, meeting the following conditions during the Maintenance Phase: 1. Two or more injection intervals affected by over dosage deviations, for example • Extra injection or excessive volume administered • Length of time between injections less than 21 days between the first and second injections (between M1 and M2 for OLI; between Day 1 and M1 for D2I), or less than 52 days for all subsequent dosing intervals, excluding split doses up to the analysis visit of interest (M12 for OLI /M11 for D2I) * 21 = 28 - 7; 52 = 28 + 31 - 7 (smallest possible dosing interval allowed - 7 days) |
| | 2. At least 10% of total time on-treatment with under dosing deviations in the Maintenance Phase up to the analysis visit of interest (i.e. Month 12 for OLI and BIK/Month11for D2I), where the % of non-compliance is calculated as: (total number of non-compliant dosing days / total number of intended exposure days) * 100% |

| Number | Exclusion Description |
|---|---|
| | Where : |
| | <ul> <li>Total number of intended exposure days = date of the last analysis timepoint snapshot viral load (up to Injection Study Day 372 for OLI subjects, up to Study Day 372 for D2I subjects and up to Study Day 378 for BIK subjects) – Start Date of Study Treatment + 1</li> </ul> |
| | <ul> <li>Total number of non-compliant dosing days up to the analysis timepoint visit<br/>(or date of IP discontinuation/ withdrawal, whichever is earlier), is derived as<br/>follows:</li> <li>BIK Arm:</li> </ul> |
| | <ul> <li>Duration of interruptions in BIK arm for reasons other than treatment-<br/>related adverse events/laboratory abnormalities (based on Exposure<br/>eCRF forms)</li> </ul> |
| | Q2M Arm: |
| | <ul> <li>Length of time (in days) in excess until next injection from date of dosage/administration deviation potentially resulting in under dosage.</li> <li>Examples include: <ul> <li>less than 3 ml administered</li> </ul> </li> </ul> |
| | - early stop of oral bridging prior to the next planned injection |
| | <ul> <li>Length of time (in days) in excess beyond 31 days between the first and<br/>second injections and beyond 69 days for all subsequent dosing intervals.</li> </ul> |
| | * 69 = 31+ 31 + 7 (largest possible dosing interval allowed + 7 days) - For those with oral bridging (OB), length of time (in days) is calculated between the start of oral bridging and the <i>preceding</i> injection |
| | Interrupted days in oral study treatment (oral lead-in or oral bridging) if<br>the oral dose has been interrupted for 3 or more consecutive days and<br>the primary interruption reason is not adverse event or laboratory<br>abnormality (based on the eCRF Exposure forms). 3 days will be<br>assumed if such interrupted days are not available in the database. |
| 03 | Prohibited medications: receiving ART medication other than that prescribed/allowed by the study (excluding permanent changes in ART regimen; such cases will be retained as 'HIV1-RNA ≥ 50 c/mL' in the per protocol snapshot analysis) or receiving prohibited concomitant medication that would impact exposure or response to therapy with duration and route of administration taken into consideration, as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination) |
| 04 | Permanent discontinuation of IP/withdrawal due to a reason of "Protocol Deviation" (as recorded in the eCRF Conclusion form). |
| 05 | Other important protocol deviations that exclude participant from Per Protocol population as recorded in the Protocol Deviation form in the eCRF based on study team review (where indicated in the PDMP as case-by-case determination). |
| * Note: Cat | egory 02 is only applicable to the Month 12 analysis. |

# 16.2. Appendix 2: Schedule of Activities

Time and Events Table for CAB LA + RPV LA Oral Lead In (OLI) Participants:

| | isit a | Maintenance Phase Extension Phase | | | | | | | | | al<br>ıts <sup>y</sup> | E Z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ing V | p | | | | | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z | | | | |
| | Screening Visit <sup>a</sup> | Day 1b | 1° | 2 | 4 | 6 | 8 | 10 | 12 | Q2M after<br>Month 12 | With | Lor |
| Written Informed Consent | Χ | | | | | | | | | | | |
| Eligibility Verification (Inclusion/<br>Exclusion Criteria) | X | Χď | | | | | | | | | | |
| Randomization | | Χ | | | | | | | | | | |
| Demography | Χ | | | | | | | | | | | |
| Medical History <sup>e</sup> | X | | | | | | | | | | | |
| Cardiovascular risk assessmente | X | Χ | | | | | | | X | | X | |
| Medication History/ Prior ART history | X | | | | | | | | | | | |
| Syphilis serology + reflex Rapid Plasma<br>Reagin (RPR) | X | X | | | | | | | | | | |
| Symptom Directed Physical Exam and<br>Medical Assessment <sup>f</sup> | Х | X | Х | X | Х | Х | Х | Х | Х | X | Х | Х |
| Weight, Height and BMl9 | | Χ | | Х | Χ | Χ | | | Χ | | X | |
| Waist Circumference | | Χ | | X | Χ | Χ | | | Х | | Х | |
| Hip Circumference | | X | | X | Х | Χ | | | Х | | Х | |
| Vital Signs (BP, HR, Temperature) <sup>h</sup> | Х | Χ | | Χ | X | Χ | | | Χ | | Χ | |
| CCI | | | | | | | | | | | | |
| 12-lead ECG <sup>i</sup><br>(triplicate at Day 1 pre-dose) | X | X | Х | | | | | | X | | X | |
| CDC HIV-1 stage# | Χ | Χ | | | | | | | | | | |
| HIV Associated Conditions | | Χ | Х | Х | Х | Х | X | Х | Х | X | Х | Х |
| AEs, SAEs, Concomitant Medications | Χj | X | X | X | X | Χ | X | X | Χ | X | X | X |
| ISR Assessment for IM injection | | | Х | X | X | X | X | X | X | X | X | X |

| | ısit <sup>a</sup> | | Maintenance Phase Extension Phase | | | | | | | | ral<br>ntsy | E Z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | V guin | q | | | | | Month | | | | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| | Screening Visit <sup>a</sup> | Day 1b | 1° | 2 | 4 | 6 | 8 | 10 | 12 | Q2M after<br>Month 12 | With | 집 |
| Columbia Suicide Severity Rating Scale<br>(eC-SSRS) k | X | Х | | X | | X | | | X | | Х | |
| Clinical chemistry and Hematology | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Testing | S | ٥ | U | U | U | U | U | U | U | U | S | U |
| HIV-1 RNA and sample for storage (S) <sup>m</sup> | Χ | Χ | X | X | X | X | X | X | X | X | X | X |
| HIV-1 RNA low copy sample | | Χ | | | | | | | X | | | |
| CD4+ cell count | Χ | Χ | X | X | X | Χ | X | X | X | X | X | X |
| CD8+ cell count | | Χ | | | | Χ | | | X | | X | |
| Urinalysis <sup>n</sup> | | Χ | X | | | X | | | X | | X | |
| Fasting Labs Glucose, Cholesterol (Total, HDL and LDL) and Triglycerideso | | X | | | | X | | | X | | Хp | |
| Hepatitis B (HBsAg), Anti-HBc, and Anti-<br>HBsAG, Hepatitis C<br>(anti-HCV Ab) | X | | | | | | | | | | | |
| PT/PTT/INR | X | Χ | | | | | | | | | | |
| Whole Blood (Virology) | | Χ | | | | X | | | X | | X | |
| | | V | | | | V | | | V | | V | |
| PBMCs q<br>Insulin, HbA1c and renal, and bone | | X | | | | X | | | X | | X | |
| biomarker analytes (blood urine) <sup>r</sup> | | Α | | | | X | | | X | | X | |
| Genetics sample t | | X | | | | | | | | | | |
| PK sampling <sup>u</sup><br>(S)=Storage only | | | S | s | S | S | S | S | S | | Х | s |
| Oral CAB and Oral RPV Dispensation v | | Χ | | | | | | | | | | |

| | Visit <sup>a</sup> | | Maintenance Phase | | | | | | | | al<br>nts/ | E Z |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | V gui | 16 | Month | | | | | | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z | | |
| | Screening | Day 1 | 1° | 2 | 4 | 6 | 8 | 10 | 12 | Q2M after<br>Month 12 | With | Lo<br>NS |
| IP accountability (Pill Counts) | | | X | | | | | | | | | |
| IM treatment administration w | | | X | X | X | X | X | X | Χ | X | | |
| HIV TSQs <sup>cc</sup> | | Χ | | | | X | | | X | | Xqq | |
| HIV TSQc <sup>∞</sup> | | | | | | | | | Х | | Xqq | |
| CCI | | | | | | | | | | | | |
| Preference <sup>cc</sup> | | | | | | | | | X | | Xqq | |
| PIN∞ | | | | X | | Х | | | Х | | Xqq | |
| CCI | | | | | | | | | | | | |
| History of Cosmetic procedures <sup>99</sup> | | | | | | | | | X | | X | |

# Time and Events Table for CAB LA + RPV LA Direct to Injection (D2I) Participants:

| | sit a | | Maintenance Phase Extension Phase | | | | | | | - ks | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ng Vie | , | | | | Mont | th | | | Withdrawal | Long-Term<br>Follow-up z |
| | Screening Visit <sup>a</sup> | Day 1₺ | 1° | 3 | 5 | 7 | 9 | 11 | Q2M after<br>Month 11 | Withdrawal<br>Assessments <sup>y</sup> | Lon<br>Folk |
| Written Informed Consent | Х | | | | | | | | | | |
| Eligibility Verification (Inclusion/<br>Exclusion Criteria) | X | Χα | | | | | | | | | |
| Randomization | | Χ | | | | | | | | | |
| Demography | X | | | | | | | | | | |
| Medical Historye | X | | | | | | | | | | |
| Cardiovascular risk assessmente | Х | Χ | | | | | | Х | | | |
| Medication History/ Prior ART history | X | | | | | | | | | | |
| Syphilis serology + reflex Rapid Plasma<br>Reagin (RPR) | X | X | | | | | | | | | |
| Symptom Directed Physical Exam and<br>Medical Assessment <sup>f</sup> | X | X | Х | Х | Х | Х | х | х | Х | Х | X |
| Weight, Height and BMI <sup>g</sup> | | Χ | Χ | Χ | Χ | | | X | | Χ | |
| Waist Circumference | | Χ | Χ | X | X | | | X | | Χ | |
| Hip Circumference | | Χ | X | X | X | | | X | | X | |
| Vital Signs (BP, HR, Temperature) <sup>h</sup> | X | X | X | X | X | | | X | | X | |
| 12-lead ECG <sup>i</sup><br>(triplicate at Day 1 pre-dose) | X | Х | | | | | | X | | X | |
| CDC HIV-1 stage <sup>ff</sup> | X | Χ | | | | | | | | | |
| HIV Associated Conditions | | Χ | Χ | X | X | Χ | Χ | Х | Х | Χ | X |
| AEs, SAEs, Concomitant Medications | χi | Χ | X | X | X | Χ | X | Χ | Х | X | X |
| ISR Assessment for IM injection | | Х | X | X | X | X | X | X | X | X | X |
| Columbia Suicide Severity Rating Scale<br>(eC-SSRS) k | X | X | X | | X | | | X | | Х | |

| | sit a | | | | Maintenan | ice Phase | | | Extension<br>Phase | = x | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | ing Vis | | | | | Mont | th | | | Withdrawal | Long-Term<br>Follow-up z |
| | Screening Visit <sup>a</sup> | Day 1b | <b>1</b> º | 3 | 5 | 7 | 9 | 11 | Q2M after<br>Month 11 | Withdrawal<br>Assessments <sup>y</sup> | Long<br>Follo |
| Clinical chemistry and Hematology | X | Χ | X | X | X | Χ | Χ | X | Х | X | X |
| Pregnancy Testing | S | U | U | U | U | U | U | U | U | S | U |
| HIV-1 RNA and sample for storage (S) <sup>m</sup> | X | X | X | X | X | Х | Х | X | Х | X | X |
| HIV-1 RNA low copy sample | | X | | | | | | X | | ] | |
| CD4+ cell count | X | X | Χ | Х | Χ | X | X | X | X | X | X |
| CD8+ cell count | | X | | | X | | | X | | X | |
| Urinalysis <sup>n</sup> | | X | X | | X | | | X | | X | |
| Fasting Labs: Glucose, Cholesterol<br>(Total, HDL and LDL) and<br>Triglycerides <sup>o</sup> | | x | | | х | | | х | | ХР | |
| Hepatitis B (HBsAg), Anti-HBc, and<br>Anti-HBsAG, Hepatitis C (anti-HCV Ab) | X | | | | | | | | | | |
| PT/PTT/INR | X | X | | | | | | | | | |
| Whole Blood (Virology) | | X | | | X | | | X | | X | |
| CCI | | | | | | | | | | | |
| PBMCs q | | Χ | | | X | | | X | | X | |
| Insulin, HbA1c and renal, and bone<br>biomarker analytes (blood urine) <sup>r</sup> | | X | | | X | | | X | | Хx | |
| CCI | | | | | | | | | | | |
| Genetics sample t | | X | | | | | | | | | |
| PK sampling u(S)=Storage only | | | S | S | S | S | S | S | | Х | S |
| IM treatment administration | | Х | Х | Х | X | Х | Χ | Χ | Х | | |
| HIV TSQs <sup>cc</sup> | | X | | | X | | | X | | Xqq | |
| HIV TSQc∞ | | | | | | | | X | | Xqq | |
| CCI | | | | | | | | | | | |
| Preference <sup>∞</sup> | | | | | | | | X | | Xqq | |

| | Visit a | | | | Maintenan | ce Phase | Extension<br>Phase | | | E Z | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Procedure | | | | Month | | | | | | drawal<br>sment | g-Term |
| | Screening | Day 1⁵ | <b>1</b> º | | | | | | Q2M after<br>Month 11 | With | Long |
| PIN∞ | | | Χ | | Χ | | | X | | Xaa | |
| CCI | | | | | | | | | | | |
| History of Cosmetic procedures <sup>99</sup> | | | | | | | | X | | X | |

# Time and Events Table for BIK Participants:

| | Screening Visit <sup>a</sup> | | Maintenance Phase | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | ning \ | 4 | Month | | | | | | |
| | ** | Day 1b | 2 | 4 | 6 | 8 | 10 | 12 <sup>bb</sup> | Withdrawal<br>Assessments <sup>y</sup> |
| Written Informed Consent | Х | | | | | | | | |
| Eligibility Verification (Inclusion/<br>Exclusion Criteria) | Х | Χq | | | | | | | |
| Randomization | | X | | | | | | | |
| Demography | X | | | | | | | | |
| Medical History <sup>e</sup> | X | | | | | | | | |
| Cardiovascular risk assessmente | X | X | | | | | | X | |
| Medication History/ Prior ART history | Х | | | | | | | | |
| Syphilis serology + reflex Rapid Plasma Reagin (RPR) | X | X | | | | | | | |
| Symptom Directed Physical Exam and Medical<br>Assessment | Х | Х | X | x | X | X | X | X | X |
| Weight, Height and BMI9 | | Х | Х | Х | X | | | X | Х |
| Waist Circumference | | Х | X | Х | X | | | X | Х |
| Hip Circumference | | Х | X | Х | X | | | X | Х |
| Vital Signs (BP, HR, Temperature) <sup>h</sup> | Χ | X | X | X | Χ | | | X | X |
| 12-lead ECGi<br>(triplicate at Day 1 pre-dose) | X | X | | | | | | X | Х |
| CDC HIV-1 stage# | Х | X | | | | | | | ] |
| HIV Associated Conditions | | X | X | X | X | X | X | X | X |
| AEs, SAEs, Concomitant Medications | Χī | X | X | Χ | X | X | X | X | X |
| Columbia Suicide Severity Rating Scale (eC-SSRS) k | X | X | X | | X | | | X | X |
| Clinical chemistry and Hematology | Х | X | X | Х | X | X | X | X | X |
| Pregnancy Testing | S | U | U | U | U | U | U | U | S |
| HIV-1 RNA and sample for storage (S)m | Х | X | X | Χ | X | X | X | X | Х |
| HIV-1 RNA low copy sample | | X | | | | | | X | |

| | Maintenance Phase Month 2 4 6 8 10 12 <sup>bb</sup> | | | | | | | | Withdrawal<br>Assessments <sup>y</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | ning \ | 4 | Month | | | | | | |
| | Screen | Day 1b | 2 | 4 | 6 | 8 | 10 | 12 <sup>bb</sup> | Withdrawal |
| CD4+ cell count | X | X | Χ | Χ | X | Х | Х | Х | X |
| CD8+ cell count | | X | | | X | | | X | X |
| Urinalysis <sup>n</sup> | | Х | | | X | | | Х | X |
| Fasting Labs<br>Glucose, Cholesterol (Total, HDL and LDL) and<br>Triglycerides∘ | | х | | | х | | | х | Хр |
| Hepatitis B (HBsAg), Anti-HBc, and Anti-HBsAG,<br>Hepatitis C<br>(anti-HCV Ab) | X | | | | | | | | |
| PT/PTT/INR | X | X | | | | | | | |
| Whole Blood (Virology) | | X | | | X | | | X | X |
| CCI | | | | | | | | | |
| PBMCs q | | X | | | X | | | X | X |
| Insulin, HbA1c and renal, and bone biomarker analytes (blood urine) <sup>r</sup> | | X | | | X | | | X | Хх |
| Genetics sample t | | X | | | | | | | |
| BIK Dispensation | | X | X | X | X | X | X | Xaa | |
| IP accountability (Pill Counts) | | | Х | X | X | X | X | X | |
| HIV TSQs∞ | | X | | | X | | | X | Xqq |
| HIV TSQc∞ | | | | | | | | X | Xdd |
| CCI | | | | | | | | | |
| History of Cosmetic procedures <sup>99</sup> | | | | | | | | Х | X |

# Time and Events Table for BIK to Oral Lead In – Extension Phase:

| | | Exten | sion Phase | | ` | |
|---|---|---|---|---|---|---|
| Procedure | | | Month | | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| | 13 | 14 | 15 | Q2M After<br>Month 15 | With | Lon |
| Eligibility Verification (Inclusion/<br>Exclusion Criteria) | Χα | | | | | |
| Symptom Directed Physical Exam and Medical<br>Assessment <sup>f</sup> | X | X | X | X | X | х |
| Weight, Height and BMl | | | | | Х | |
| Waist Circumference | | | | | Х | |
| Hip Circumference | | | | | Х | |
| Vital Signs (BP, HR, Temperature) <sup>n</sup> | | | | | Х | |
| 12-lead ECG <sup>i</sup> | | | | | X | |
| HIV Associated Conditions | X | Х | X | Χ | X | Х |
| AEs, SAEs, Concomitant Medications | Х | Х | X | Х | X | X |
| ISR Assessment for IM injection | | Х | X | X | X | Х |
| Clinical chemistry and Hematology | X | Х | X | X | X | ) x |
| Pregnancy Testing | S | U | U | U | S | U |
| HIV-1 RNA and sample for storage (S) <sup>m</sup> | Х | Х | X | X | Х | χ |
| CD4+ cell count | | X | X | X | X | χ |
| CD8+ cell count | | | | | Х | |
| Urinalysis <sup>n</sup> | | Х | | | X | |
| Fasting Labs<br>Glucose, Cholesterol (Total, HDL and LDL) and<br>Triglycerides <sup>o</sup> | | х | | | X | |
| Whole Blood (Virology) | | | | | X | |
| CCI | | | | | | |
| PBMCs q | | | | | X | |

# CONFIDENTIAL

| | | | nsion Phase | | wal<br>ents <sup>y</sup> | E Z C |
|---|---|---|---|---|---|---|
| Procedure | | | Month | ndraw<br>ssme | T-Ter | |
| | 13 | 14 | 15 | Q2M After<br>Month 15 | Withdrawal<br>Assessment | Long-Term<br>Follow-up z |
| PK sampling <sup>u</sup><br>(S)=Storage only | | S | S | | х | S |
| Oral CAB and Oral RPV Dispensation v | X | | | | | |
| IP accountability (Pill Counts) | X | X | | | | |
| IM treatment administration w | | X | X | X | | |

# Time and Events Table for BIK to Direct to Injection – Extension Phase:

| | | Extension Ph | ase | | |
|---|---|---|---|---|---|
| Procedure | | Month | | Withdrawal<br>Assessments <sup>y</sup> | Long-Term<br>Follow-up z |
| | 13 | 14 | Q2M After Month<br>14 | With | Long |
| Eligibility Verification (Inclusion/<br>Exclusion Criteria) | Χq | | | | |
| Symptom Directed Physical Exam and Medical<br>Assessment <sup>r</sup> | X | X | x | X | х |
| Weight, Height and BMl⁰ | | | | X | |
| Waist Circumference | | | | X | |
| Hip Circumference | | | | X | |
| Vital Signs (BP, HR, Temperature) <sup>n</sup> | | | | X | |
| 12-lead ECGi | | | | x | |
| HIV Associated Conditions | X | X | X | X | X |
| AEs, SAEs, Concomitant Medications | X | Х | X | X | X |
| ISR Assessment for IM injection | X | X | X | Х | X |
| Clinical chemistry and Hematology | X | X | X | Х | X |
| Pregnancy Testing | S | U | U | 8 | U |
| HIV-1 RNA and sample for storage (S) <sup>m</sup> | X | X | X | Χ | X |
| CD4+ cell count | | X | X | Χ | X |
| CD8+ cell count | | | | Χ | |
| Urinalysis <sup>n</sup> | | Х | | X | |
| Fasting Labs Glucose, Cholesterol (Total, HDL and LDL) and Triglycerides <sup>o</sup> | | х | | х | |
| Whole Blood (Virology) | | | | X | |
| PBMCs q | | | | X | |

| Procedure | | Extension Phase | • | Irawal<br>:ments <sup>y</sup> | Long-Term<br>Follow-up z |
|---|---|---|---|---|---|
| Tiocedule | 13 | 14 | Q2M After Month<br>14 | Withdraw<br>Assessmer | Long |
| PK sampling <sup>u</sup><br>(S)=Storage only | | S | | Х | s |
| IP accountability (Pill Counts) | X | | | | |
| IM treatment administration w | X | X | X | | |

Safety Follow Up Visit: Conduct approximately 4 weeks after the last dose of IP. Required only if the participant has ongoing AEs or lab abnormalities at the last on-study visit. This visit may be conducted by telephone.

Note: BP – Blood pressure, HR – Heart Rate, BMI – Body Mass Index, HDL – High Density Lipoprotein, LDL – Low Density Lipoprotein, PT - Prothrombin Time, PTT - Partial Thromboplastin Time, INR - International normalized ratio, PBMC – peripheral blood mononuclear cell, RNA – Ribonucleic acid, HbA1c = Glycated hemoglobin, HBsAg = hepatitis B surface antigen, HCV = hepatitis C virus, HIV-1 = human immunodeficiency virus type 1.

- a. Complete all Screening assessments within 35 days. Participants may begin the Maintenance Phase as soon as all Screening assessments are complete. Participants may be rescreened once and will be assigned a new participant number.
- b. For participants who elect to participate in the oral lead in period, oral CAB 30 mg + RPV 25 mg will be administered and the oral lead will start on Day 1. For participants who choose to go directly into injections, the first loading dose will be administered on Day 1. Visits for participants on the BIK arm are expected to occur every 56 days as projected according to the Day 1 visit. There is a ±3 day visit window, from the projected visit date (Maintenance Phase of the study).
- c. For participants who elect to participate in the oral lead in period, the first loading dose will be administered and the oral lead in will end. For participants who choose to go directly into injections, the second loading dose will be administered.
- Confirmation of eligibility to continue the Maintenance Phase, and eligibility to enter the Extension Phase.
- e. Collect full routine medical history plus (report at Baseline visit): HIV risk factors (may be collected at a later study visit), cardiovascular risk factors (assessments include smoking status and history, family history of cardiac events), recent [≤6 months] illicit drug use, intravenous drug use, gastrointestinal disease, metabolic, psychiatric, renal, bone, and neurologic disorders. At Month 11 (D2I)/12 (OLI and BIK), assessments inclusive of smoking status, alcohol use and illicit drug use since the start of the study will be administered.
- f. Physical exams should be conducted as part of normal routine clinical care. Medical assessments include any decisions the study staff must make for participants management and/or care of participant.
- g. Height collected at Baseline Day 1 only. Recommended procedures to measure weight, waist and hip circumference can be found in protocol Section 10.10. Weight related measurements to be collected are weight, body fat %, total body water %, muscle mass, and bone mineral mass.
- h. Measure vital signs after about 5 minutes of rest in a semi-supine position.
- i. A 12-lead ECG will be performed after resting in a semi-supine position for at least 5 minutes. ECGs will be performed pre-dose. ECG pre-dose will be performed in triplicate at Day 1. A 2-hour post-dose ECG will also be performed at Day 1 (D2I), Month 1 (OLI) and Month 12 (OLI)/Month 11 (D2I) for participants receiving CAB LA + RPV LA with an allowable window of ± 30 minutes.
- Only SAEs related to study participation or to a concomitantly administered ViiV/GSK product will be collected between obtaining informed consent and administration of study drug at Day 1.
- k. On Day 1, the eC-SSRS is to be administered prior to randomization. The eC-SSRS will be completed at the beginning of the visit following administration of other PROs required prior to injections. The eC-SSRS is not required during the Withdrawal visit if withdrawal occurs during the Extension Phase.
- I. Women of childbearing potential only. S=serum, U=urine. Pregnancy events will be captured starting at Day 1 following initial exposure to study drug. Serum pregnancy test can substitute for urine pregnancy test if locally required but must be appropriately timed to confirm pregnancy status prior to randomization and first IM administration. If the urine test is positive, perform a serum test and do not administer injection. The frequency of pregnancy tests should be performed according to local legal requirements.
- m. Month 12 (OLI and BIK) and Month 11 (D2I) HIV-1 RNA retest (within 4 weeks) for results > 50 c/mL will be captured as unscheduled visit. Plasma for storage samples will be used for possible future analyses.
- A morning specimen is preferred. To assess biomarkers: urine albumin/creatinine ratio; urine protein/creatinine ratio; urine phosphate; beta-2-microglobulin; and retinol binding protein.
- An overnight fast is preferred; however, a minimum of a 6-hour fast is acceptable.
- p. Only collect if the Withdrawal visit occurs at Month 6 or Month 12 (OLI and BIK); Month 5 or Month 11 (D2I).
- q. Whole blood/PBMC collection samples may be used for virologic analyses. PBMCs will be collected at baseline Day 1, Month 6, Month 12, or Withdrawal if prior to Month 12 (OLI and BIK). PBMCs will be collected at baseline Day 1, Month 5, Month 11, or Withdrawal if prior to Month 11 (D2I)
- r. Blood sample for insulin, HbA1c, and renal and bone biomarker assessments: Renal: CystatinC; Beta-2-Microglobulin; Retinol Binding Protein (RBP); Bone: bone specific alkaline phosphatase, procollagen type 1-N-propeptide, type 1 collagen cross-linked C-telopeptide, osteocalcin, 25 hydroxy-Vitamin D.
- Blood sample force
- t. Informed consent for genetic research must be obtained before sample collection. Sample may be collected at any visit after signing informed consent, but preferably at the Day 1 visit
- u. One blood sample for CAB and RPV each to be collected at each PK timepoint. At Month 1, for participants who elected to participate in the Oral Lead in, and Month 14 for participants who were randomized to BIK and switched to CAB LA + RPV LA in the Extension Phase and will participate in the Oral Lead in, Pre dose PK samples are to be collected: PRIOR to the final oral dose of CAB + RPV. For pregnant participants (on CAB+RPV arm): two blood samples for CAB and one RPV sample at each PK timepoint. Refer to protocol Section 10.6.6.3.
- v. Participants who elected to participate in the Oral Lead in before switching to CAB LA + RPV LA injections, will take final dose of oral lead-in regimen in the clinic at the Month 1/Month 14 visit and begin injections.
- w. If possible, injections should be spaced approximately 2 cm from one another and from the site of any previous injection and or any injection site reaction. Bring RPV LA to approximately room temperature prior to injecting. Time and location of injection (right or left) as well as needle length used will be collected in the eCRF. The first injection can be performed before central lab results become available and safety parameters are reviewed.
- x. Collect sample for these assessments ONLY if the Withdrawal visit occurs at Months 6 and 12 (OLI and BIK); Month 5 and 11 (D2I).
- y. Refer to Section 7.1 of the protocol for additional information on performing withdrawal assessments
- z. Participants receiving one or more injections with CAB LA and/or RPV LA will be assessed with clinic visits at Months 3, 6, 9 and 12 during the Long-Term Follow-Up Phase
- aa. BIK dispensation (1-month supply) for participants who plan on entering into the Extension Phase. Participants who do not enter the Extension Phase or do not wish to transition to the commercial supply will not receive 1-month supply at M12.

- bb. Data from visit will be used to determine participant's eligibility to enter the Extension Phase of study. If participant elects to enter the Extension Phase, determine if the participant will elect to start injections immediately or start with oral lead in.
- cc. All PROs are recommended to be administered before other assessments and injections take place at each designated visit.
- dd. Only collected if Withdrawal visit occurs during the Maintenance Phase.
- ff. When assessing CDC stage at Screening/Baseline, consider only the latest available CD4 T-cell count, except when the participant had an active Stage 3 event 6 months prior to Screening.
- gg. At Month 11 (D2I)/ Month 12 (OLI or BIK) or withdrawal, (depending which is sooner) participants will be asked if any cosmetic procedures were performed during the conduct of the study.

# 16.3. Appendix 3: Assessment Windows

## 16.3.1. Definitions of Assessment Windows for Analyses

Unless otherwise noted, laboratory data, vital signs, ECGs, Health Outcomes assessments, and genotypic/phenotypic data will be assigned to assessment windows according to actual dates rather than the nominal visit labels as recorded on the eCRF or in the laboratory database.

In most cases the window around an assessment will include all dates from the midpoints between the target day and that of the previous and the proceeding visits. The target Study Day or target Injection Study Day for is defined in Section 16.3.2.

For parameters which are not scheduled to be assessed at a particular visit, the all-inclusive assessment windows will still be used; however, data summaries will only report scheduled visits. Assessments at unscheduled visits will be included for "any time" and "on-treatment" time points and in data listings, as well any algorithms that make use of additional data (e.g., snapshot).

Maintenance phase assessments are assigned based on the Maintenance Phase Study Day, respectively. Extension phase assessments are assigned based on the Maintenance Phase Study day for subjects continuing CAB LA + RPV LA dosing (Q2M) into the Extension Phase, and based on the Extension Phase Study Day for subjects switching from the BIK arm to CAB LA + RPV LA dosing (Switch Q2M) for the Extension phase. Long-term Follow-up phase assessments are assigned based on the LTFU study day. See Section 16.6.1 for derivation of Maintenance, Extension and LTFU Study Day.

# 16.3.2. Definitions of Assessment Windows for Data Other than Health Outcomes

# 16.3.2.1. Assessment Windows for Screening, Maintenance and Extension Phase Data – Q2M OLI Subjects

| All Parameters except for where noted ি | Analysis Window | Target<br>Study Day | Target<br>Injection<br>Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint<br>2 | Notes |
|---|---|---|---|---|---|---|
| | Study Day ≤ 1 | Study day of<br>the earliest<br>record | | Screening | Screening | Screening |
| | Last available recorded value up<br>to and including the date of first<br>Maintenance Phase dose of IP | 1 | | Maintenance<br>Baseline (Day 1) | Maintenance<br>Baseline (Day 1) | Maintenance<br>Baseline (Day 1) |
| Post-dose ECG | Value taken post-dose | 1 | | Day 1 (Post Dose) | Day 1(Post Dose) | Day 1(Post Dose) |
| Urinalysis | Injection Study Day ≤ 15 and Study Day ≥2 For those with OLI only: 2<= Study Day<= Study Day of Last Oral Dose +1 Injection Study Day ≤ 42 and Study Day ≥2 For those with OLI only: 2<= Study Day<= Study Day of Last Oral Dose +1 | 31 | 1 | Month 1 | Month 1 | Injection 1 |
| Post-dose ECG | Value taken post-dose Month 1<br>16 ≤ Injection Study Day ≤ 60 | 61 | 31 | Month 2 | Month 2 | Injection 2 |
| | 61 ≤ Injection Study Day ≤ 120 | 121 | 91 | Month 4 | Month 3/4 | Injection 3 |
| | 121 ≤ Injection Study Day ≤ 180 | | | | | , |
| Urinalysis <sup>[a]</sup> , CD8, CD4/CD8 ratio, fasting<br>glucose and lipids <sup>[a]</sup> , weight, height, BMI,<br>Waist and Hip Circumference, Vital<br>Signs [SCIIII], Insulin, HbA1c, HOMA-IR, | 121 ≤ Injection Study Day ≤ 192 | 181 | 151 | Month 6 | Month 5/6 | Injection 4 |

| All Parameters except for where noted <sup>[d]</sup> | Analysis Window | Target<br>Study Day | Target<br>Injection<br>Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint<br>2 | Notes |
|---|---|---|---|---|---|---|
| Renal, Bone and COI | | | | | | |
| - | 181 ≤ Injection Study Day ≤ 240 | 241 | 211 | Month 8 | Month 7/8 | Injection 5 |
| | 241 ≤ Injection Study Day ≤ 300 | 301 | 271 | Month 10 | Month 9/10 | Injection 6 |
| | 301 ≤ Injection Study Day ≤ 360 | | | | | |
| Urinalysis <sup>[a]</sup> , CD8, CD4/CD8 ratio, fasting glucose and lipids <sup>[b]</sup> , weight, height, BMI, Waist and Hip Circumference, Vital Signs, CCI , Insulin, HbA1c, Renal, Bone and CCI | 301 ≤ Injection Study Day ≤ 372 | 361 | 331 | Month 12 | Month 11/12 | Injection 7 |
| | 361 ≤ Injection Study Day ≤ 420 For those who did not continue to Extension after completing Maintenance Phase: 361 ≤ Injection Study Day ≤ Injection Study Day of: max(Last Injection Date + 67, Date of Last Oral Dose + 1) | 421 | 391 | Month 14 | Month 13/14 | Injection 8 |
| | (30*m - 59) ≤ Injection Study<br>Day ≤ (30*m) | 30*m + 1 | 30*m - 29 | Month 16, 18, etc. | Month m-1/m | Injection (m/2+1) |
| | If subject permar | nently discont | inued study tre | eatment: | • | • |
| | Subject received at least 1 injection of IP: Date > min(LTFU ART start date, max(Last Injection Date + 67, Date of Last Oral Dose + 1)) Subject received oral CAB/RPV only: Date > (Date of Last oral CAB/RPV Dose +1) | | | Follow-up | Follow-up | Follow-up |

#### NOTES:

- Analysis windows are applied after data has been assigned to the Maintenance Phase and Extension Phase as defined in Section 16.4.1
- Study day and injection study day is defined in Section 16.6.1
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19 impact.
- Target Injection Study Day is only applicable to Q2M OLI subjects

[a] Urinalysis: All parameters provided by the central laboratory under the category of urinalysis.

[b] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
[c]Bone Markers: Bone-specific alkaline phosphatase, Procollagen type 1 N-propeptide, Type 1 collagen cross-linked C-telopeptide, Osteocalcin, 25 hydroxy-Vitamin D; Renal Markers: Cystatin C, Retinol Binding Protein, Beta-2-Microglobulin; CCI

[d] Analysis windows for parameters with sparse collection are noted.

# 16.3.2.2. Assessment Windows for Screening, Maintenance and Extension Phase Data – Q2M D2I Subjects

| All Parameters except for where notedে | Analysis Window | Target Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint 2 | Notes |
|---|---|---|---|---|---|
| | Study Day ≤ 1 | Study day of the earliest record | Screening | Screening | Screening |
| | Last available recorded value up<br>to and including the date of first<br>Maintenance Phase dose of IP | 1 | Maintenance<br>Baseline (Day 1) | Maintenance<br>Baseline (Day 1) | Injection 1 |
| post-dose ECG | Value taken post-dose | 1 | Day 1 (Post<br>Dose) | Day 1(Post Dose) | Injection 1 |
| | 2 ≤ Study Day ≤ 60 | 31 | Month 1 | Month 1 | Injection 2 |
| Urinalysis | 2 ≤ Study Day ≤ 72 | 31 | IWORLE I | IMONUT I | Injection 2 |
| | 61 ≤ Study Day ≤ 120 | 91 | Month 3 | Month 3/4 | Injection 3 |
| | 121 ≤ Study Day ≤ 180 | | | | |
| Urinalysis <sup>[3]</sup> , CD8, CD4/CD8 ratio, fasting glucose and lipids <sup>[3]</sup> , weight, height, BMI, Waist and Hip Circumference, Vital Signs, COL, Insulin, HbA1c, Renal, Bone and CCI | 121 ≤ Study Day ≤ 192 | 151 | Month 5 | Month 5/6 | Injection 4 |
| | 181 ≤ Study Day ≤ 240 | 211 | Month 7 | Month 7/8 | Injection 5 |
| | 241 ≤ Study Day ≤ 300 | 271 | Month 9 | Month 9/10 | Injection 6 |
| | 301 ≤ Study Day ≤ 360 | | | | |
| Urinalysis <sup>[a]</sup> , CD8, CD4/CD8 ratio, fasting glucose and lipids <sup>[b]</sup> , weight, height, BMI, Waist and Hip Circumference, Vital Signs, color Insulin, HbA1c, Renal, Bone and color | 301 ≤ Study Day ≤ 372 | 331 | Month 11 | Month 11/12 | Injection 7 |

| All Parameters except for where noted <sup>[c]</sup> | Analysis Window | Target Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint 2 | Notes |
|---|---|---|---|---|---|
| | 361 ≤ Study Day ≤ 420 For those who did not continue to Extension after completing Maintenance Phase: 361 ≤ Study Day ≤ max(Last Injection Date + 67, Date of Last Oral Dose + 1)) | 391 | Month 13 | Month 13/14 | Injection 8 |
| | (30*m - 29) ≤ Study Day ≤<br>(30*m + 30) | 30*m + 1 | Month 15, 17,<br>etc. | Month m/m+1 | Injection ((m+3)/2) |
| If subject permanently discontinued study treatment: | | | | | |
| | Date > min(LTFU ART start<br>date, max(Last Injection Date +<br>67, Date of Last Oral Dose + 1)) | | Follow-up | Follow-up | Follow-up |

#### NOTES:

- Analysis windows are applied after data has been assigned to the Maintenance Phase and Extension Phase as defined in Section 16.4.1
- Study day is defined in Section 16.6.1
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19 impact.

[a] Urinalysis: All parameters provided by the central laboratory under the category of urinalysis.

[b] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides [c]Bone Markers: Bone-specific alkaline phosphatase, Procollagen type 1 N-propeptide, Type 1 collagen cross-linked C-telopeptide, Osteocalcin, 25 hydroxy-Vitamin D; Renal Markers: Cystatin C, Retinol Binding Protein, Beta-2-Microglobulin; CCI

[d] Analysis windows for parameters with sparse collection are noted.

# 16.3.2.3. Assessment Windows for Screening and Maintenance Phase Data -BIK

| All Parameters except for where<br>noted <sup>[ৱ]</sup> | Analysis Window | Target Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint 2 | Notes |
|---|---|---|---|---|---|
| | Study Day ≤ 1 | Study day of the earliest record | Screening | Screening | |
| | Last available recorded value up<br>to and including the date of first<br>Maintenance Phase dose of IP | 1 | Maintenance<br>Baseline (Day<br>1) | Maintenance<br>Baseline (Day 1) | |
| post-dose ECG | Value taken post-dose | 1 | Day 1 (Post<br>Dose) | Day 1(Post Dose) | |
| | 2 ≤ Study Day ≤ 84 | 57 | Month 2 | Month 2 | |
| | 85 ≤ Study Day ≤ 140 | 113 | Month 4 | Month 3/4 | |
| | 141 ≤ Study Day ≤ 196 | | | | |
| Urinalysis, CD8, CD4/CD8 ratio, fasting glucose and lipids, weight, height, BMI, Waist and Hip Circumference, Vital Signs, CCIII, Insulin, HbA1c, Renal, Bone and | 141 ≤ Study Day ≤ 210 | 169 | Month 6 | Month 5/6 | |
| | 197 ≤ Study Day ≤ 252 | 225 | Month 8 | Month 7/8 | |
| | 253 ≤ Study Day ≤ 308 | 281 | Month 10 | Month 9/10 | |
| | 309 ≤ Study Day ≤ 350 | | | | |
| Urinalysis <sup>[a]</sup> , CD8, CD4/CD8 ratio, fasting glucose and lipids <sup>[b]</sup> , weight, height, BMI, Waist and Hip Circumference, Vital Signs, CCIII, Insulin, HbA1c, Renal, Bone and | 309 ≤ Study Day ≤ 378 | 337 | Month 12 | Month 11/12 | |
| | 351 ≤ Study Day ≤ Study Day of<br>Last Maintenance BIK Dose +1 | 365 | Month 13 | Month 13/14 | |
| | If subject permar | ently discontinued study treat | ment: | | |
| | Date> (Date of Last BIK Dose<br>+1) | | Follow-up | Follow-up | |

<sup>80</sup> 

- Note for the BIK arm, the "every two months" are implemented as "every 56 days", therefore the analysis windows are adjusted according to the actual visit schedules instead
  of nominal.
- Study day is defined in Section 16.6.1
- Follow-up will be derived only for participants who permanently discontinued study treatment.

[a] Urinalysis: All parameters provided by the central laboratory under the category of urinalysis.

[b] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides

[c]Bone Markers: Bone-specific alkaline phosphatase, Procollagen type 1 N-propeptide, Type 1 collagen cross-linked C-telopeptide, Osteocalcin, 25 hydroxy-Vitamin D; Renal

Markers: Cystatin C, Retinol Binding Protein, Beta-2-Microglobulin; Col

[d] Analysis windows for parameters with sparse collection are noted.

# 16.3.2.4. Assessment Windows for Extension Phase Data – BIK subjects Switching to CAB LA + RPV LA (Switch Q2M) and choose OLI (Switch OLI)

| All Parameters except for where noted <sup>[c]</sup> | Analysis Window | Target<br>Extension<br>Study Day | Target Extension Injection Study Day | Analysis<br>Timepoint 1 | Analysis Timepoint 2 | Notes |
|---|---|---|---|---|---|---|
| | Last available recorded value up to and including the date of first Extension Phase dose of CAB/RPV | 1 | | Extension<br>Baseline<br>(Month 13) | Extension Baseline<br>(Month 13) | |
| Urinalysis <sup>[a]</sup> , fasting<br>glucose and lipids <sup>[b]</sup> | Extension Injection Study Day ≤ 15 and Extension Study day ≥2 For those with Ext OLI only: 2<= Extension Study Day<= Extension Study Day of Last Extension Oral Dose +1 Extension Injection Study Day ≤ 42 and Extension Study day ≥2 For those with Ext OLI only: 2<= Extension Study Day<= Extension Study Day of Last Extension Oral Dose +1 | 31 | 1 | Month 14 | Month 14 | Extension Injection 1 |
| | 16 ≤ Extension Injection Study Day ≤ 60 | 61 | 31 | Month 15 | Month 15 | Extension Injection 2 |
| | 61 ≤ Extension Injection Study Day ≤ 120 | 121 | 91 | Month 17 | Month 16/17 | Extension Injection 3 |
| | 121 ≤ Extension Injection Study Day ≤ 180 | 181 | 151 | Month 19 | Month 18/19 | Extension Injection 4 |
| | $(30*(m-14) - 29) \le$ Extension Injection Study Day $\le (30*(m-14)+30)$ | 30*(m-13) + 1 | 30*(m-14) + 1 | Month 21, 23, etc. | Month m-1/m | Extension Injection (m-11)/2 |
| | If subject permar | nently discontir | nued study treat | ment: | | |
| | Subject received at least 1 injection of IP: Date > min(LTFU ART start date, max(Last Injection Date + 67, Date of Last Oral Dose + 1)) Subject received oral CAB/RPV only: Date> (Date of Last oral Dose +1) | | - | Follow-up | Follow-up | |

# NOTES:

- Analysis windows are applied after data has been assigned to the Extension Phase as defined in Section 16.4.1
- Extension Study day and Extension Injection Study Day is defined in Section 16.6.1
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19 impact.
- Target Extension Injection Study Day is only applicable to Switch Q2M subjects who choose OLI during the Extension Phase
- [a] **Urinalysis:** All parameters provided by the central laboratory under the category of urinalysis.
- [b] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- [c] Analysis windows for parameters with sparse collection are noted.

# 16.3.2.5. Assessment Windows for Extension Phase Data –BIK subjects Switching to CAB LA + RPV LA (Switch Q2M) and choose D2I (Switch D2I)

| All Parameters except for where noted <sup>[c]</sup> | Analysis Window | Target Extension Study Day | Analysis<br>Timepoint 1 | Analysis<br>Timepoint 2 | Notes |
|---|---|---|---|---|---|
| | Last available recorded value up to and including the date of first Extension Phase dose of CAB/RPV | 1 | Extension<br>Baseline<br>(Month 13) | Extension Baseline<br>(Month 13) | Extension Injection 1 |
| Urinalysis <sup>[a]</sup> , fasting<br>glucose and lipids <sup>[b]</sup> | $2 \le \text{Study Day} \le 60$<br>$2 \le \text{Study Day} \le 72$ | 31 | Month 14 | Month 14 | Extension Injection 2 |
| | 61 ≤ Study Day ≤ 120 | 91 | Month 16 | Month 16/17 | Extension Injection 3 |
| | 121 ≤ Study Day ≤ 180 | 151 | Month 18 | Month 18/19 | Extension Injection 4 |
| | $(30*(m-13) - 29) \le Study Day \le (30*(m-13) + 30)$ | 30*(m-13) + 1 | Month 20, 22,<br>etc. | Month m/m+1 | Extension Injection (m-10)/2 |
| | If subject perman | ently discontinued study trea | tment: | | |
| | Date > min(LTFU ART start date, max(Last Injection Date + 67, Date of Last Oral Dose + 1)) | , | Follow-up | Follow-up | |

#### NOTES:

- Analysis windows are applied after data has been assigned to the Extension Phase as defined in Section 16.4.1
- Extension Study day is defined in Section 16.6.1
- Follow-up will be derived only for participants who permanently discontinued study treatment.
- Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19 impact.
- [a] Urinalysis: All parameters provided by the central laboratory under the category of urinalysis.
- [b] Lipids: Cholesterol, HDL Cholesterol Direct, LDL Cholesterol Calculation, LDL Cholesterol Direct, Total Cholesterol/HDL Cholesterol Ratio, Triglycerides
- [c] Analysis windows for parameters with sparse collection are noted.

# 16.3.2.6. Assessment Windows for Summary of Snapshot Data - Data assigned to Maintenance Phase Only

| Snapshot Analysis<br>(If no on-treatment viral load data in defau | | Analysis | Analysis |
|---|---|---|---|
| Default <sup>[a]</sup> | Expanded +6 Week Upper Window | Timepoint 1 | Timepoint 2 |
| Last available recorded value up to and including the date of first<br>Maintenance Phase dose of IP | Last available recorded value up to and including the date of first Maintenance Phase dose of IP | Maintenance<br>Baseline (Day 1) | Maintenance<br>Baseline (Day 1) |
| CAB LA + RPV LA (OLI) | | | |
| Injection Study Day ≤ 15 and Study Day ≥2 For those with OLI only: 2<= Study Day<= 45 | Injection Study Day ≤ 42 and Study Day ≥2 For those with OLI only: 2<= Study Day<= Study Day of Last Oral Dose +1 | Month 1 | Month 1 |
| 16 ≤ Injection Study Day ≤ 60 | 16 ≤ Injection Study Day ≤ 72 | Month 2 | Month 2 |
| 61 ≤ Injection Study Day ≤ 120 | 61 ≤ Injection Study Day ≤ 132 | Month 4 | Month 3/4 |
| 109 ≤ Injection Study Day ≤ 192 | 109 ≤ Injection Study Day ≤ 192 | Month 6 | Month 5/6 |
| 181 ≤ Injection Study Day ≤ 240 | 181 ≤ Injection Study Day ≤ 252 | Month 8 | Month 7/8 |
| 241 ≤ Injection Study Day ≤ 300 | 241 ≤ Injection Study Day ≤ 312 | Month 10 | Month 9/10 |
| 289 ≤ Injection Study Day ≤ 372 | 289 ≤ Injection Study Day ≤ 372 | Month 12 | Month 11/12 |
| CAB LA + RPV LA (D2I) | | | |
| 2 ≤ Study Day ≤ 60 | 2 ≤ Study Day ≤ 72 | Month 1 | Month 1 |
| 61 ≤ Study Day ≤ 120 | 61 ≤ Study Day ≤ 132 | Month 3 | Month 3/4 |
| 109 ≤ Study Day ≤ 192 | 109 ≤ Study Day ≤ 192 | Month 5 | Month 5/6 |
| 181 ≤ Study Day ≤ 240 | 181 ≤ Study Day ≤ 252 | Month 7 | Month 7/8 |
| 241 ≤ Study Day ≤ 300 | 241 ≤ Study Day ≤ 312 | Month 9 | Month 9/10 |
| 289 ≤ Study Day ≤ 372 | 289 ≤ Study Day ≤ 372 | Month 11 | Month 11/12 |
| BIK Arm | | | |
| 2 ≤ Study Day ≤ 84 | 2 ≤ Study Day ≤ 98 | Month 2 | Month 2 |
| 85 ≤ Study Day ≤ 140 | 85 ≤ Study Day ≤ 154 | Month 4 | Month 3/4 |
| 127 ≤ Study Day ≤ 210 | 127 ≤ Study Day ≤ 210 | Month 6 | Month 5/6 |
| 197 ≤ Study Day ≤ 252 | 197 ≤ Study Day ≤ 266 | Month 8 | Month 7/8 |
| 253 ≤ Study Day ≤ 308 | 253 ≤ Study Day ≤ 322 | Month 10 | Month 9/10 |
| 295 ≤ Study Day ≤ 378 | 295 ≤ Study Day ≤ 378 | Month 12 | Month 11/12 |

- o An on-treatment viral load assessment may be assigned to more than one snapshot analysis window.
  - a.  $\pm$  6 Week window is always used at key analysis timepoints (Month 5/6 and Month 11/12). For other analysis timepoints, if no viral load data in default window, expand upper bound to +6 weeks.

# 16.3.2.7. Assessment Windows for Summaries of Long-Term Follow Up Phase Data

| Analysis Window | Analysis<br>Timepoint | Target LTFU Study Day of Window |
|---|---|---|
| 1 ≤ LTFU Study Day ≤ 135 | LTFU Month 3 | 90 |
| 136 ≤ LTFU Study Day ≤ 225 | LTFU Month 6 | 180 |
| 226 ≤ LTFU Study Day ≤ 315 | LTFU Month 9 | 270 |
| 316 ≤ LTFU Study Day ≤ 405 | LTFU Month 12 | 360 |
| (30*m - 44) ≤ LTFU Study Day≤ (30*m + 45) | LTFU Month m | 30*m |
| | m = 15, 18,21, | |

#### NOTES:

- Analysis windows are applied after data has been assigned to the LTFU Phase as defined in Section 16.4.1.
- Long-Term Follow-Up (LTFU) Study day is defined in Section 16.6.1
- An assessment may be slotted to both LTFU and Maintenance/Extension Phase

#### 16.3.3. Assessment Window for Study Conclusion

The study conclusion and Phase conclusion records in disposition data will be slotted based on Section 16.3.1 for Maintenance and Extension Phase conclusion records. However, if the discontinuation date is post-treatment (based on Section 16.4.3), then the discontinuation will be slotted to the participant's last attained on-treatment analysis visit across all assessments (e.g. analysis visit corresponding to the last on-treatment lab assessment), rather than follow up.

#### 16.3.4. Assessment Window for Health Outcome Data

#### 16.3.4.1. HIVTSQs/HIVTSQc/PINICOL

Assessments will be assigned to analysis visits as follows:

- Maintenance Baseline (Day 1) will be defined as last available recorded value up
  to and including the date of first Maintenance Phase dose of study treatment
  (expected to be collected at Day 1). Baseline is not applicable for PIN, HIVTSQc
  and other one-time questionnaires such as treatment preference.
- If the nominal visit identifier as captured in the source dataset corresponds to a
  scheduled collection per the Time and Events Schedule (see Section 16.2) and the
  assessment is collected in the Maintenance Phase (see Section 16.4.1.2), then the
  nominal visit identifier will be kept as the analysis visit (excluding Day 1 which
  will normally be assigned to Maintenance Baseline (Day 1).
- If the nominal visit identifier is unscheduled or withdrawal, then the following procedure will be used:
  - Assign the assessment to a study Phase according to Section 16.4.1.2.
     Proceed to step b if the assessment is assigned to the Maintenance Phase.

- Identify the 'last nominal visit' with the HO assessment performed prior to the unscheduled/withdrawal visit to be slotted.
- c. Unscheduled/withdrawal visits will be slotted to the planned nominal visit subsequent to the 'last nominal visit'. If the 'last nominal visits' does not exist (e.g. no records originate from a planned nominal visit), then the unscheduled/withdrawal visit will be slotted to the first planned nominal visit after Day 1. If there is already an original (planned) value for the subsequent visit, then the original value will be selected instead of an 'unscheduled' value.

Example 1, for HIVTSQs, for Q2M subjects with OLI, the planned nominal visits are Day 1, Month 6, and Month 12. If a participant has the 'last nominal visit' (with HIVTSQs assessment) at Month 6 prior to withdrawal at Month 8, the withdrawal assessment will be slotted to the subsequent planned nominal visit of Month 12.

Example 2, for HIVTSQs, for Q2M subjects with OLI if there is unscheduled visit between Month 6 and Month 12, this unscheduled visit will be slotted to Month 12. In this case, there are two assessments with analysis visit equal to Month 12 (i.e. the slotted value and the value at original nominal Month 12 visit). The original nominal value will be selected for summary per the rule below for multiple records—see Section 16.3.5.

Table 6 Planned Nominal Visit of Health Outcome Data

| Questionnaire | Day 1 | Month 1/2 | Month 5/6 | Month 11/12 |
|---|---|---|---|---|
| PIN | | X | X | X |
| HIVTSQs | X | | X | X |
| HIVTSQc | | | | X |
| CCI | | | | |
| NOTES: | | | | |
| Day 1 visits are recorded as "Baseline | " visits in the da | atabase. | | |



#### 16.3.4.3. Treatment Preference

The treatment preference questionnaire is taken at Month 11/12 and withdrawal. The nominal visit identifier will be kept as the analysis visit. Data will be reported separately for Month 11/12 and for withdrawal.

#### 16.3.5. Multiple assessments within an Analysis Window

If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:

For data other than health outcome:

- the assessment closest to the window target Study Day (or target Injection Study Day if injection study day is used for assessment window slotting);
- if there are multiple assessments equidistant from the target Study Day or target Injection Study Day, then the mean of these values will be used. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean. For post-dose ECG, the assessment closest to two-hour post injection will be used.

#### Health outcome assessments:

- if there are multiple assessments assigned to the same analysis visit, the assessment from the original planned nominal visit will be used for summary statistics.
- if there are multiple assessments assigned to the same analysis visit and none originate from a planned nominal visit (e.g. two unscheduled/withdrawal nominal visits), then
  - a. the assessment closest to the window target Study Day will be used;
  - b. if there are multiple assessments equidistant from the target Study Day, then the earliest assessment will be used.

Assessments not chosen for use in summary statistics by this algorithm will still be included in the associated listings. Also, all applicable assessments, irrespective of proximity to the target study day, will be used when categorizing values across visits, such as 'maximum grade' or 'at any time', and for any algorithm that has specific rules for which observation to use (e.g., snapshot algorithm or CVF identification, where applicable).

# 16.4. Appendix 4: Study Phases and Treatment State

# 16.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to the Treatment Start Date defined in Section 16.6.1.

AEs will be assigned to study phases as defined in Section 16.4.1.1.

Laboratory data (efficacy, safety, and virology), HIV associated/ AIDS-defining conditions, health outcomes assessments, vital signs, and ECGs will be assigned to study phases as defined as in Section 16.4.1.2. For example, assessments/events occurring up to and including start of extension phase IP/LTFU ART will be assigned to the Maintenance Phase.

Assessments/events are assigned to study phases sequentially, starting from the top of each table.

# 16.4.1.1. Study Phases for AEs

| Study Phase | Date range |
|---|---|
| Screen | Date < Maintenance Treatment Start Date |
| Maintenance | Q2M Arm (OLI and D2I): |
| | For participants continuing into Extension Phase: OLI: Maintenance Treatment Start Date ≤ Date < Date of Nominal Month 14 Injection Visit D2I: Maintenance Treatment Start Date ≤ Date < Date of Nominal Month 13 Injection Visit |
| | For participants <u>not</u> continuing into Extension Phase: Maintenance Treatment Start Date ≤ Date < LTFU ART Start Date (if applicable) |
| | Note: |
| | - For AEs leading to withdrawal and started on the same date as LTFU ART Start Date, Maintenance Phase, instead of Long-term Follow-up phase, will be assigned. |
| | - LTFU ART start date is not applicable for those who complete maintenance phase and transition to commercial supply. |
| | BIK Arm: For participants continuing into Extension Phase: Maintenance Treatment Start Date ≤ Date < min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) |
| | For participants <u>not</u> continuing into Extension Phase: |
| | Date ≥Maintenance Treatment Start Date |

| Study Phase | Date range |
|---|---|
| Extension | Participants continuing maintenance CAB LA + RPV LA into Extension Phase OLI: Date of Nominal Month 14 Injection Visit ≤ Date < LTFU ART Start Date (if applicable) |
| | <b>D2I:</b> Date of Nominal Month 13 Injection Visit ≤ <b>Date</b> < LTFU ART Start Date (if applicable) |
| | Participants Switching from Maintenance BIK Arm to CAB LA + RPV LA: |
| | min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) ≤ <b>Date</b> < LTFU ART Start Date (if applicable) |
| | Note: LTFU ART start date is not applicable for those who transition to commercial supply. |
| • <b>Date</b> = A | AE Start date |
| • Mainten | ance Treatment Start Date: refer to Treatment Start Date in Section 16.6.1 |

# 16.4.1.2. Study Phases for Lab assessments, ECG, Vital Signs, Health Outcomes, Protocol Deviations, and HIV associated/AIDS-defining conditions

| Study Phase | Date range |
|---|---|
| Screen | Date ≤ Maintenance Treatment Start Date |
| Maintenance | Q2M Arm: |
| | For participants continuing into Extension Phase: |
| | <b>OLI:</b> Maintenance Treatment Start Date < <b>Date</b> ≤ Date of Nominal Month 14 Injection Visit |
| | <b>D2I:</b> Maintenance Treatment Start Date < <b>Date</b> ≤ Date of Nominal Month 13 Injection Visit |
| | For participants <u>not</u> continuing into Extension Phase: |
| | Maintenance Treatment Start Date < <b>Date</b> ≤ LTFU ART Start Date (if applicable) |
| | Note: LTFU ART start date is not applicable for those who complete maintenance phase and transition to commercial supply. |

| Study Phase | Date range |
|---|---|
| | BIK Arm: For participants continuing into Extension Phase: Maintenance Treatment Start Date < Date ≤ min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) For participants not continuing into Extension Phase: |
| | Date > Maintenance Treatment Start Date |
| Extension | Participants continuing maintenance CAB LA + RPV LA into Extension Phase OLI: Date of Nominal Month 14 Injection Visit < Date ≤ LTFU ART Start Date (if applicable) D2I: Date of Nominal Month 13 Injection Visit < Date ≤ LTFU ART Start Date (if applicable) |
| | Participants Switching from Maintenance BIK arm to CAB LA + RPV LA: min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) < Date ≤ LTFU ART Start Date (if applicable) Note: LTFU ART start date is not applicable for those who transition to commercial supply. |

- Date = start or assessment date
- Maintenance Treatment Start Date: refer to Treatment Start Date in Section 16.6.1

# 16.4.1.3. Long-Term Follow-Up Phase

| Study Phase | Date range |
|---|---|
| Long-Term | Date > max (Last CAB/RPV Injection Date, Last Oral Bridging End Date) |
| Follow-Up | |

- Date = Assessment/Start Date
- Only applicable to subjects who have received at least 1 injection
- LTFU phase is not applicable for those who transition to commercial supply. Last oral Bridging may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19.

Note that the long-term follow-up Phase and Maintenance/Extension Phases are not necessarily mutually exclusive and are to be defined with separate Phase variables in the datasets.

# 16.4.1.4. Study Phases for Concomitant medication/ART

| Study Phase | Date range |
|---|---|
| Prior | Medication Taken < Maintenance Treatment Start Date |
| Maintenance <sup>[a]</sup> | Q2M Arm (OLI and D2I): |
| | For participants continuing into Extension Phase: |
| | <b>OLI:</b> Maintenance Treatment Start Date ≤ <b>Medication Taken</b> < Date of |
| | Nominal Month 14 Injection Visit |
| | <b>D2I:</b> Maintenance Treatment Start Date ≤ <b>Medication Taken</b> < Date of Nominal Month 13 Injection Visit |
| | For participants <u>not</u> continuing into Extension Phase: Maintenance Treatment Start Date ≤ Medication Taken < LTFU ART Start Date (if applicable) |
| | Note: LTFU ART start date is not applicable for those who transition to commercial supply. |
| | BIK Arm: |
| | For participants continuing into Extension Phase: |
| | Maintenance Treatment Start Date ≤ <b>Medication Taken</b> < min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) |
| | For participants <u>not</u> continuing into Extension Phase: |
| | Medication Taken ≥Maintenance Treatment Start Date |
| Extension <sup>[b]</sup> | Participants continuing maintenance CAB LA + RPV LA into Extension |
| | <pre>Phase OLI: Date of Nominal Month 14 Injection Visit ≤ Medication Taken &lt; LTFU ART Start Date (if applicable)</pre> |
| | <b>D2I:</b> Date of Nominal Month 13 Injection Visit ≤ <b>Medication Taken</b> < LTFU ART Start Date (if applicable) |
| | Participants Switching from Maintenance BIK Arm to CAB LA + RPV LA: |
| | min (Start Date of Extension Phase CAB/RPV oral lead-in, Date of first Extension Phase CAB/RPV injection) ≤ <b>Medication Taken</b> < LTFU ART Start Date (if applicable) |
| | Note: LTFU ART start date is not applicable for those who transition to commercial supply. |

| Study Phase | Date range |
|---|---|
| Long-Term | For participants who received at least one CAB and/or RPV Injection: |
| Follow-Up | |
| | Medication Taken ≥ LTFU ART Start Date |
| | Notes I TELL above to and conflicted from the conduction of the conflicted from the conduction of the |
| | Note: LTFU phase is not applicable for those who transition to commercial supply. |
| [a]: ART stopped on the start date of Maintenance Treatment will be considered a prior medication and will not be considered concomitant during the Maintenance Phase. If the stop date of ART medication is completely missing and this medication is recorded in eCRF as prior, it will be considered a prior medication and will not be considered concomitant during the Maintenance phase. | |
| [b]: ART stopped on the start date of Extension Phase IP will not be assigned to the Extension Phase. | |

If a partial date for medication/ART is recorded in the eCRF, the following convention will be used to assign the medication:

- if the partial date is a start date, a '01' will be used for missing days and 'Jan' will be used for missing months;
- if the partial date is a stop date, a '28/29/30/31' will be used for the missing day (dependent on the month and year) and 'Dec' will be used for the missing month; for medications recorded separately in the eCRF as prior ART, the earlier of this imputed date or the day before IP start will be used.

# 16.4.2. Study Periods

Certain displays will be produced for data collected during the oral-lead-in. These period variables are defined in the tables below and will be reflected in the datasets with separate variables.

# 16.4.2.1. Oral Lead-in Period for AE Data

| Study Period | Date range |
|---|---|
| Maintenance | Q2M OLI subjects only: |
| Phase Oral | |
| Lead-in | For participants receiving at least one Injection: Maintenance Treatment Start Date ≤ Date < Date of First Maintenance Phase CAB/RPV Injection |
| | For participants withdrawing prior to first Injection: Date ≥ Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |
| Extension<br>Phase Oral | Switch Q2M OLI subjects only: |
| Lead-in | For participants receiving at least one Extension Phase Injection: Extension Oral CAB/RPV Start Date ≤ Date < Date of First Extension Phase CAB/RP injection |
| | For participants withdrawing prior to first Extension Phase Injection: Date ≥ Extension Phase Oral CAB/RPV Start Date |

# 16.4.2.2. Oral Lead-in Period for Lab assessments

| Study Period | Date range |
|---|---|
| Maintenance<br>Phase Oral | Q2M OLI subjects only: |
| Lead-in | For participants receiving at least one Injection: Maintenance Treatment Start Date < Date ≤ Date of First Maintenance Phase CAB/RPV Injection |
| | For participants withdrawing prior to first Injection: Date > Maintenance Treatment Start Date |
| | Note that the oral lead-in period is only applicable to the participants who received at least one dose of study treatment during the oral lead-in period in the study. Oral lead-in period is within the maintenance phase. |

| Extension | Switch Q2M OLI subjects only: |
|---|---|
| Phase Oral | |
| Lead-in | For participants receiving at least one Extension Phase Injection: Extension Oral CAB/RPV Start Date < Date ≤ Date of First Extension Phase CAB/RP injection |
| | For participants withdrawing prior to first Extension Phase Injection: Date > Extension Oral CAB/RPV Start Date |

# 16.4.3. Treatment State

Within each treatment study phase (i.e. Maintenance, and Extension—based on assignment of study phase described in Section 16.4.1), only those assessments which occur within the ranges shown below will be considered 'on-treatment' for the given phase. Note "on-treatment" criteria will not be implemented for adverse event summaries.

Table 7 Treatment State within Study Phases

| Study Phase <sup>a</sup> | Treatment State | Date Range |
|---|---|---|
| Screen | Pre-treatment | All assessments/events within Phase |
| Maintenance | On-treatment | Q2M Arm: |
| | | <b>Date</b> ≤ max (Date of Last Injection Dose + 67, Date of Last Oral Dose + 1) |
| | | BIK Arm: |
| | | Date ≤ Maintenance ART Stop Date + 1 |
| | Post-treatment | Q2M Arm: |
| | | Date > max (Date of Last Injection Dose + 67, Date of Last Oral Dose + 1) |
| | | BIK Arm: |
| | | Date > Maintenance ART Stop Date + 1 |
| Extension | On-treatment | Date ≤ max (Date of Last IP Injection Dose + 67,<br>Date of Last Oral Dose + 1) |
| | Post-treatment | Date > max (Date of Last IP Injection Dose + 67,<br>Date of Last Oral Dose + 1) |
| Long-Term<br>Follow-up | On-treatment | Date ≤ min (LTFU ART start date, max (Date of Last IP Injection Date + 67, Date of Last Oral Dose + 1)) |
| | Post-treatment | Date > min (LTFU ART start date, max (Date of Last IP Injection Date + 67, Date of Last Oral Dose + 1)) |
| Noto: | | |

#### Note:

• Treatment State is determined after data has been assigned to the study Phases as defined in Section 16.4.1

- The upper bound with last IP injection / last oral dose /Maintenance ART Stop Date should only be applied to participants who permanently discontinue from study treatment
- Date = Assessment/Start Date.
- Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19.

# 16.4.4. Combining Treatment Phases and States

On-treatment and Post-treatment assessments and events will be classified as occurring during the Maintenance Phase, Extension, or Long-term follow up Phase.

# 16.5. Appendix 5: Data Display Standards & Handling Conventions

# 16.5.1. Reporting Process

#### Software

- The currently supported versions of SAS software or R/RStudio will be used.
- The specific versions of SAS or R packages used to generate the analyses will be detailed in the ADRG.

# **Reporting Area**

| HARP Server | : us1salx00259 |
|---------------|--------------------------------|
| HARP Compound | : \ARPROD\GSK1265744\mid213500 |

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 & ADaM IG Version 1.2).
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for reporting efforts described in the RAP.

# 16.5.2. Reporting Standards

#### General

- The current GSK Statistical Display Standards in the GSK Standards Library (IDSL) will be applied for reporting, unless otherwise stated (Library Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include participant level listings in the main body of the GSK Clinical Study Report. All
  participant level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK Statistical Display Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the GSK Standard Statistical Display Principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:

- If space permits, planned and actual time relative to study drug dosing will be shown in listings (Refer to GSK Standard Statistical Display Principle 5.05.1).
- Unscheduled or unplanned readings will be presented within the participant's listings.

#### **Unscheduled Visits**

- Unscheduled visits will be slotted to analysis time points as per Section 16.3.
- However, data summaries will only report visits that are planned assessment time points for each parameter (according to the Time and Events table).
- Assessments at unscheduled visits will be included for 'any time On-treatment' time points and in data listings, as well any algorithms that make use of additional data (e.g., Snapshot and PDVF identification).
- All unscheduled visits will be included in listings.

| Descriptive Summary Statistics | |
|---|---|
| Continuous Data | Refer to GSK Standard Statistical Display Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Graphical Displays | |
| Refer to GSK Standard Statistical Display Principals 7.01 to 7.13. | |

# CONFIDENTIAL

213500

- 16.6. Appendix 6: Derived and Transformed Data
- 16.6.1. **General**

#### Multiple Measurements at One Analysis Time Point

- If after window assignment there are multiple valid assessments of a parameter within the same window, then the following hierarchy will be used to determine the value to be used for summary statistics of observed values:
  - the assessment closest to the window target Study Day (or target Injection Study Day if injection study day is used for assessment window slotting);
  - if there are multiple assessments equidistant from the target Study Day or target Injection Study Day, then for continuous variables the mean of these values will be used and for categorical variables the worse assessment. For HIV-1 RNA, the geometric mean of the number of copies will be used as opposed to the arithmetic mean
- Assessments not chosen for use in summary statistics by this algorithm will still appear in the
  associated listings. Also, such valid assessments will be used when determining values of potential
  clinical concern for the 'any time ' time point, and for any algorithm that has specific rules for which
  observation to use (e.g., Snapshot).

#### **Treatment Start Date**

Treatment start date is defined as follows:

- Maintenance Phase
  - For participants randomized to Q2M: Date of first dose of CAB + RPV (oral or injection) entered in the IP exposure CRF form.
  - For participants randomized to BIK: BIK regimen start date entered in the Maintenance Phase IP exposure CRF
- Extension Phase
  - For participants continuing CAB LA + RPV LA (Q2M):
    - for Q2M OLI: Date of the nominal Month 14 injection date
    - for Q2M D2I: Date of the nominal Month 13 injection date
    - For participants switching from BIK to Q2M:

      Date of the nominal Month 13 Q2M injection date (BIK to D2I) or the oral CAB + RPV start date entered in the Extension Phase IP exposure CRF (BIK to OLI)

#### Study Day

The Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the Maintenance Phase start date of study treatment as follows:

if date of event ≥ start date of study treatment, then

Study Day = Date of Event – Start Date of Maintenance Phase IP + 1

if date of event < start date of study treatment, then

Study Day = Date of Event – Start Date of Maintenance Phase IP

Note that the start date of study treatment on Maintenance Phase is considered to be on Study Day 1 and the day before this is Study Day -1; i.e., there is no Study Day 0.

Injection Study Day (Maintenance Phase) (Only applicable to Q2M OLI subjects)

The Injection Study Day of an event will be derived as the number of days between the date of the event and the date of first Maintenance Phase injection as follows:

if date of event ≥ first Maintenance Phase injection, then

Injection Study Day = Date of Event – Date of First Maintenance Phase CAB/RPV Injection + 1

if date of event < first Maintenance Phase injection, then

Injection Study Day = Date of Event – Date of First Maintenance Phase CAB/RPV Injection

Note that the date of first Maintenance Phase injection is considered to be on Injection Study Day 1 and the day before this is Injection Study Day -1; i.e., there is no Injection Study Day 0.

#### **Extension Study Day**

The Extension Phase Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the initial start date of Extension Phase IP as follows:

if date of event ≥ start date of Extension Phase IP, then

Extension Study Day = Date of Event – Start Date of Extension Phase IP + 1

if date of event < start date of Extension Phase IP, then

Extension Study Day = Date of Event – Start Date of Extension Phase IP

Note that the start date of Extension Phase IP is considered to be on Extension Phase Study Day 1 and the day before this is Extension Phase Study Day -1; i.e., there is no Extension Phase Study Day 0.

#### Extension Injection Study Day (Only applicable to Extension Switch OLI subjects)

The Extension Phase Injection Study Day of an event (e.g., lab assessment, vital sign, ECG, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the initial start date of Extension Phase injection as follows:

if date of event ≥ date of first Extension Phase injection, then

 Extension Injection Study Day = Date of Event – Date of First Extension Phase CAB/RPV Injection + 1

if date of event < date of first Extension Phase injection, then

 Extension Injection Study Day = Date of Event – Date of First Extension Phase CAB/RPV Injection

Note that the date of first Extension Phase Injection is considered to be on Extension Injection Study Day 1 and the day before this is Extension Injection Study Day -1; i.e., there is no Extension Phase Injection Study Day 0.

#### Long-Term Follow Up Study Day

The Long-Term Follow Up (LTFU) Study Day of an event (e.g., lab assessment, start date of AE or HIV associated/AIDS-defining condition) will be derived as the number of days between the date of the event and the end of IP treatment [i.e max (Last IM Injection Date, Last Oral Bridging End Date)] as follows:

If the onset of event falls in Long-term Follow up Phase, then

LTFU Study Day = Date of Event – End Date of IP

# 16.6.2. Study Population

#### **Demographics and Baseline Characteristics**

#### Age

- Age, in whole years, will be calculated with respect to the participant's Screening visit.
- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
- Any participant with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.
- Completely missing dates of birth will remain as missing, with no imputation applied. Consequently, the age of the participant will not be calculated and will remain missing.

#### **Body Mass Index (BMI)**

• BMI is calculated as Weight (kg) / Height (m)<sup>2</sup>. Height is only collected at Baseline Day 1.

#### **Hepatitis Status**

- Hepatitis status at entry will be based on the assessments prior to/on the start of the study treatment.
- A participant will be considered positive for hepatitis B virus (HBV) if they have a positive surface antigen or detectable HBV DNA result. "HBV DNA DETECTED" in the lab comment takes precedence over HBV DNA test result for positive hepatitis B status, for example, if a participant has HBV test result below level of detection, however, the lab comment shows that HBV DNA detected, this participant will be considered positive for hepatitis B. If HBV DNA result is available, it will be used to qualify hepatitis B status as positive or negative (positive if ≥ limit of quantification); otherwise Hepatitis B status will be determined using the surface antigen result (i.e. "REACTIVE").
- Hepatitis C status will be determined using antibody (IgM or IgG) and/or hepatitis C virus (HCV) RNA assessments performed during screening or during the conduct of the study. If both antibody and virus RNA assessments are available, then the latter will take precedence and positive/negative status will be based on whether HCV RNA is detectable (i.e., ≥ limit of quantification) or not. In the absence of an HBV RNA result, Hepatitis C antibody of "REACTIVE" or "BORDERLINE" will qualify as Hep C positive.

#### Framingham Risk Equation

• The predicted probability,  $\hat{p}$ , of having a cardiovascular disease (CVD) within the next 10-years according to the Framingham formula [D'Agostino, 2008] is

#### For females:

```
\hat{p}_F = 1 - S_0(t) \exp\{2.32888 \times \log(\text{age}) + 1.20904 \times \log(TC) - 0.70833 \times \log(HDL) + 2.76157 \times \log(SBPu) + 2.82263 \times \log(SBPt) + 0.52873 \times I_S + 0.69154 \times I_d - 26.1931\}.
```

#### For males:

```
\hat{p}_{M} = 1 - S_{0}(t) \exp\{3.06117 \times \log(\text{age}) + 1.12370 \times \log(TC) - 0.93263 \times \log(HDL) + 1.93303 \times \log(SBPu) + 1.99881 \times \log(SBPt) + 0.65451 \times I_{s} + 0.57367 \times I_{d} - 23.9802\},
```

#### **Demographics and Baseline Characteristics**

Where

$$S_0(t) = \begin{cases} 0.95012, \text{ females} \\ 0.88936, males \end{cases}$$

$$I_s = \begin{cases} 1, \text{ current smoker} \\ 0, & otherwise \end{cases}$$

$$I_d = \begin{cases} 1, & \text{diabetic} \\ 0, & otherwise \end{cases}$$

TC = total serum cholesterol (mg/dL),

HDL = serum HDL cholesterol (mg/dL),

SBPu = systolic blood pressure (mmHg) if participant is not treated for high blood pressure (note that if a participant is treated for high blood pressure then log(SBPu) = 0)

SBPt = systolic blood pressure (mmHg) if participant is treated for high blood pressure (note that if a participant is not treated for high blood pressure then log(SBPt) = 0)

- A participant will be considered as treated for high blood pressure if during screening it has specified
  that is suffering from hypertension. A participant is classified as diabetic if current or past is indicated
  in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or if baseline (Day 1) fasting
  glucose ≥7.00 mmol/L (126 mg/dL) and HbA1C >6.5%.
- Smoking status is collected in the eCRF at Day 1. A current smoker is defined as currently smoking/using tobacco or has smoked/used tobacco within the previous 6 months; a former smoker is defined as previously smoked/used tobacco products and has not smoked/used tobacco products within the previous 6 months.
- This calculation will not be performed for participants who have indicated current or past myocardial
  infarction conditions on the eCRF. These participants will not be included in summary statistics of
  risk, but they will be counted in the highest category of risk in the summary by category.
- Framingham Risk will also be calculated at Month 6 and Month 12.
  - Baseline smoking status will be used for the Month 6 calculation. Smoking status collected at Month 12 will be used for the Month 12 calculation.
  - Diabetic status is defined as:
    - 1. Current or past is indicated in the medical conditions eCRF for Type 1 or Type 2 diabetes mellitus, or
    - At any time prior to and including the analysis timepoint:
       2a. fasting glucose ≥7.00 mmol/L (126 mg/dL) and HbA1C >6.5%, or
    - 2b. an adverse event is collected as having "type 1 or type 2 diabetes mellitus"
  - ° "Treated for high blood pressure" at Month 6 and Month 12 is defined as
    - 1. hypertension at baseline or
    - 2. use of medication treating hypertension which started prior to and including the analysis time point

#### **Lipid-modifying Agents**

- The following ATC codes correspond to lipid-modifying agents:
  - o ATC Level 2: C10
  - o ATC Level 3: C10A, C10B (if Level 2 is not available)

#### **Demographics and Baseline Characteristics**

- ATC Level 4: C10AA, C10AB, C10AC, C10AD, C10AX, C10BA, C10BX (if level 2, 3 are not available)
- Participants are considered to have used a lipid-modifying agent at baseline if they are taking the medication at the time of their baseline fasting lipid testing date.
- Participants are also considered to have used a lipid-modifying agent at baseline if they stopped their lipid modifying medication within 12 weeks prior to their baseline fasting lipid testing date.

#### **Treatment Compliance**

 For defining protocol deviation (i.e. treatment non- compliance) leading to exclusion from the Per Protocol population, the total non-compliance days will be calculated (see details in Section 16.1).
 The percentage of the total number of non-compliant days to the Exposure ('overall exposure' for CAB+RPV treatment) will be used to define protocol deviation leading to exclusion from PP Population for the Month 12 analysis due to study treatment non-compliance (i.e. >10%).

#### Adherence to CAB/RPV Injection Schedule

Timeliness of Injections relative to Date of Projected Dosing Visits are assessed by using "actual injection visit date - projected visit date from first injection". The injections of interest in adherence analysis are those after first injection. For participants who choose oral lead-in (Q2M OLI), the first injection is planned at Month 1. For Q2M D2I participants, the first injection is planned at Day 1. Each injection visit is counted only once. Individual CAB and RPV injections administered at the same visit are not counted twice. "Extra" unscheduled injections are excluded from all derivations. For example, if during a scheduled visit a participant receives 2 ml of injection instead of 3 ml due to a dosing error, but this participant returns one week later for the remaining 1 ml injection, then the additional visit is excluded. If a participant receives an extra injection at an unscheduled visit by mistake, this visit will also be excluded.

The categories of Timeliness of Injections relative to date of Projected Dosing Visits for summary are listed below:

```
< -14 days
```

-14 to - 8 days

-7 to - 4 days

-3 to -2 days

-1 day

0 day

1 day

2 to 3 days

4 to 7 days

8 to 14 days

>14 days

Missed Injection without Oral Bridging

Missed Injection with Oral Bridging

Missed Injection with CAB+RPV Oral Bridging

Missed Injection with SOC Oral Bridging

# 16.6.3. Efficacy



#### Target Detected / Target Non-Detected/ Super Low Viral Load Testing

- When a measurement of plasma HIV-1 RNA is below the limit of quantification (i.e. 40 c/mL) and is
  qualitatively observable that will be denoted as a "Target Detected" measure, while HIV-1 RNA
  below the limit of quantification that is not qualitatively observable that will be denoted as "Target Not
  Detected". Any measurements <40 c/mL characterised as "Target Not Detected" or "Target
  Detected" will be captured in the database.</li>
- SuperLow viral load will also be tested by BioMONTR Labs for viral loads below the limit of quantification at Day 1 and Month 11/12.

#### Confirmed Virologic Failure

 The definition of CVF is provided in the Protocol, Section 7.1.6 – Definition of Protocol-Defined Virologic Failure

#### Treatment (TRDF) and Efficacy Related (ERDF) Discontinuation = Failure

 The analysis of time to confirmed virologic failure (CVF) or discontinuation due to treatment related reasons (i.e., drug-related AE, intolerability of injections, protocol defined safety stopping criteria, or lack of efficacy) will censor participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than those related to treatment. This will be the Treatment Related Discontinuation = Failure (TRDF) data.

#### HIV-1 RNA

- Participants who have not met CVF criteria and are ongoing in the study, or who have discontinued for reasons other than lack of efficacy, will be censored in the analysis of the Efficacy Related Discontinuation = Failure (ERDF) data.
- Proportion of Participants without virologic (ERDF) or tolerability (TRDF) failure will be estimated
  using the Kaplan-Meier nonparametric method based on the time to ERDF or TRDF. The estimated
  proportion at time point of interest will be presented by treatment group, along with estimated
  difference in proportions between treatment groups and its associated two-sided 95% CI. The
  estimate of the standard error used to derive confidence intervals will be based on Greenwood's
  formula [Kalbfleisch, 1980].
- See Appendix 10: Variables Defined for Time to Event Analysis for additional details

#### Delay in IP Injection

IM dosing is expected to occur every 2 months starting from the third injection and onwards. The Delay in IP injection (days) will be calculated as:

For the second injection:

Delay in IP injection(days) = Injection date - date of preceding injection - 31

For other injections:

Delay in IP injection(days) = Injection date – date of preceding injection - 62

Delay in IP injection will be grouped into: ≤1, 2-3, 4-7, >7 days.

- The proportion of participants with HIV-1 RNA≥50 c/mL at Month 12 will be summarized by last delay in IP Injection. The last delay in IP injection will be the delay in IP injection at Month 11(D2I) or Month 12(OLI), or the delay in last IP injection prior to Month 11/Month 12 if a participant does not receive their Month 11/12 injection (i.e. missing visit or withdrawal).
- Delays are defined as more than 31 or 62 days for the second and the subsequent injections, respectively.
- If there are subjects who did not receive any injection or received only one injection, then add the "No injection or only 1 injection" category.
#### 16.6.4. Safety

#### **Adverse Events**

#### **DAIDS Grading**

 Clinical adverse events will be graded based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events Version 2.1, March 2017, as specified in the protocol Appendix 4.

#### Potential QTc Interval Prolonging Events of Interest

Potential QTc Interval Prolonging Events of Interest will be identified based on Standardised MedDRA Query (SMQ) for Torsade de pointes/QT prolongation, broad (MedDRA). The terms per this reference are listed below.

| AE preferred term |
|----------------------------------------------|
| Electrocardiogram QT interval abnormal |
| Electrocardiogram QT prolonged |
| Long QT syndrome |
| Long QT syndrome congenital |
| Torsade de pointes |
| Ventricular tachycardia |
| Cardiac arrest |
| Cardiac death |
| Cardiac fibrillation |
| Cardio-respiratory arrest |
| Electrocardiogram repolarisation abnormality |
| Electrocardiogram U wave inversion |
| Electrocardiogram U wave present |
| Electrocardiogram U-wave abnormality |
| Loss of consciousness |
| Sudden cardiac death |
| Sudden death |
| Syncope |
| Ventricular arrhythmia |
| Ventricular fibrillation |
| Ventricular flutter |
| Ventricular tachyarrhythmia |

#### **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will

be used to determine how much to add or subtract in order to impute the corresponding numeric value. If a character value starting with "<=x", then the numeric value will be x.

- Example 1: 2 Significant Digits = '< x ' becomes x 0.01</li>
- Example 2: 1 Significant Digit = '> x' or '>=x' becomes x + 0.1
- Example 3: 0 Significant Digits = '< x' becomes x 1

#### Estimate of Glomerular Filtration Rate (GFR) (Levey, 2012)

 Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation [Levey, 2012]. be used by the central laboratory to provide an estimate of GFR, in mL/min per 1.73 m², as follows:

$$GFR = 141 \times \min \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{\alpha} \times \max \left(\frac{CRT_{mg/dL}}{\kappa}, 1\right)^{-1.209} \times 0.993^{Age} \times [1.018 \text{ if Female}] \times [1.159 \text{ if Black}]$$

Abbreviations / Units:

eGFR (estimated glomerular filtration rate) = mL/min/1.73 m<sup>2</sup>

age = years at time of assessment

 $\kappa = 0.7$  (if female) or 0.9 (if male)

 $\alpha$  = -0.329 (if female) and -0.411 (if male)

min() = the minimum of CRT/ $\kappa$  or 1

max() = the maximum of CRT/ $\kappa$  or 1

CRTmg/dL = serum creatinine concentration in mg/dL. The serum creatinine concentration in mg/dL is obtained from GSK standard units of  $\mu$ mol/L as CRTmg/dL =0.0113x CRT $\mu$ mol/L.

#### **Lab Toxicities**

- Toxicities will be based on the Division of AIDS (DAIDS) grading system, Version 2.1, March 2017, as specified in the protocol of Appendix 4. Toxicity grades provided by the central laboratory do not distinguish between abnormally high or low criteria, when both are relevant for a particular parameter.
- When summarising toxicity grades for such parameters, they will be categorised as to whether they are above or below the midpoint of normal range.

| Parameter | Below Midpoint for those ≥Grade 1 | Above Midpoint for those ≥Grade 1 |
|---|---|---|
| Fasted glucose | Hypoglycemia | Hyperglycemia |
| Sodium | Hyponatremia | Hypernatremia |
| Potassium | Hypokalemia | Hyperkalemia |

#### National Cholesterol Education Program (NCEP) Lipid Categories

• In addition to DAIDS toxicity grades (see protocol), lipid values will be categorized according to the 2001 NCEP Adult Lipid Guidelines [Grundy, 2001]

| Parameter | Value Range (mmol/L) | Value Range (mg/dL) | Category |
|---|---|---|---|
| Triglycerides | <1.70 | <150 | Normal |
| | 1.70 to <2.26 | 150 to <200 | Borderline High |
| | 2.26 to <5.65 | 200 to <500 | High |
| | ≥5.65 | ≥500 | Very High |
| Total Cholesterol | <5.18 | <200 | Desirable |
| | 5.18 to <6.21 | 200 to <240 | Borderline High |
| | ≥6.21 | ≥240 | High |
| HDL Cholesterol | <1.04 | <40 | Low |
| | 1.04 to <1.56 | 40 to <60 | Normal |
| | ≥1.56 | ≥60 | High |
| LDL Cholesterol | <2.59 | <100 | Optimal |
| | 2.59 to <3.37 | 100 to <130 | Near/Above Optimal |
| | 3.37 to <4.14 | 130 to <160 | Borderline High |
| | 4.14 to <4.92 | 160 to <190 | High |
| | ≥4.92 | ≥190 | Very High |

#### **Total Cholesterol / HDL Cholesterol Ratio**

• When both total cholesterol and HDL cholesterol results are available from the same date for a participant, then the ratio will be calculated by dividing the total cholesterol result by the HDL cholesterol result. The ratio can be classified as follows:

| Parameter | Value Range |
|-------------------|--------------|
| Total Cholesterol | < 3.5 |
| / HDL Ratio | 3.5 to < 4.4 |
| | 4.4 to < 5 |
| | ≥5 |

| Percentage change for lipids | |
|---|---|
| The percentage change from Baseline* is ca | Iculated as: |
| % Change from BL = | Value at Month X – BL value X 100 % |
| | BL value |
| *Maintenance or Extension | |
| Other Safety Endpoints | |
| Extent of Exposure | |
| <ul> <li>Exposure to CAB+RPV (oral lead-in), CA pages.</li> </ul> | AB LA+RPV LA, BIK will be calculated from the IP eCRF |
| Maintenance Phase: Q2M | |
| Exposure to CAB + RPV (oral lead-in) = * Q2M OLI subjects only | Oral lead-in CAB/RPV Stop Date – Oral lead-in CAB/RPV Start Date +1 |
| Exposure to CAB LA + RPV LA = | Number of IP injections received during Maintenance<br>Phase up to and include the Month 12 (OLI) or the Month<br>11 (D2I) injection |
| Overall Exposure to IP (Q2M OLI) = | min [Date of latest Maintenance Phase visit up to and including Month 14 (OLI), max (Date of last CAB LA + RPV LA injection +67, Date of last oral CAB/RPV dose) ] – Oral lead-in CAB/RPV Start Date +1 |
| Overall Exposure to IP (Q2M D2I) = | min [Date of latest Maintenance Phase visit up to and including Month 13(D2I), max (Date of last CAB LA + RPV LA injection +67, Date of last oral CAB/RPV dose) ] – CAB LA + RPV LA Start Date +1 |
| Overall Exposure to Study Treatment (OLI) = min [Date of latest Maintenance Phase visit up to an including Month 14, max (Date of last CAB LA + RP\(\text{injection}\) injection +67, Date of last oral CAB/RPV dose, Date last oral SOC bridging) ] – Oral lead-in CAB/RPV States | |
| Overall Exposure to Study Treatment (D2I) = | min [Date of latest Maintenance Phase visit up to and including Month 13, max (Date of last CAB LA + RPV LA injection +67, Date of last oral CAB/RPV dose, Date of last oral SOC bridging) ] – CAB LA + RPV LA Start Date +1 |
| Maintenance Phase: BIK arm | |
| Exposure = Min (Date of latest Maintenance Phase visit up to and including Month 13, Maintenance Phase Treatment Stop Date, Date of Maintenance Phase Discontinuation) – Maintenance Treatment Start Date + 1 | |
| <ul> <li>Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19</li> <li>Last CAB LA + RPV LA injection / last oral dose is only applicable to participants who permanently discontinue from study</li> </ul> | |

#### Corrected QT (QTc)

When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fridericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

If RR interval (in msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{RR/1000}} \qquad \qquad QTcF = \frac{QT}{\sqrt[3]{RR/1000}}$$

where uncorrected QT interval is also measured in msec.

If RR interval is not provided directly and one of QTcB or QTcF has been entered, then RR interval can be obtained from the above formulas and used to calculate the other correction method value; i.e.,

$$QTcB = \sqrt{\frac{QTcF^3}{QT}} \qquad \qquad QTcF = \sqrt[3]{QT \cdot QTcB^2}$$

#### **QTc Values by Category**

The following categories for QTc will be used:

- For absolute QTc values:
- ≤450
- >450 to ≤480
- >480 to ≤500
- >500
- For change from baseline in QTc values:
- ≤30
- >30 to ≤60
- >60

#### Columbia Suicide Severity Rating Scale (C-SSRS) (Posner, 2007)

Missing data will not have any imputation performed (Nilsson, 2013)

#### Homeostatic model assessment-Insulin Resistance (HOMA-IR)

- HOMA-IR = (fasting plasma insulin (mU/L) \* fasting plasma glucose (mmol/L)) / 22.5.
- HOMA-IR categories will be categorised as follows for the shift table analysis:
- 1. <2
- 2. 2 to <3
- 3. 3 to <4
- 4. >=4

All HOMA-IR analyses will be based on fasting values and only patients with post-baseline values will be included in analyses (i.e. patients with missing post-baseline HOMA-IR will not be included in summary tables or figures).

The following subjects will be excluded from the HOMA-IR analysis:

- diabetic as captured on the medical history or have taken an anti-diabetic medication (ATC code "A10" (<u>DRUGS USED IN DIABETES</u>)) up to screening
- fasting glucose >126mg/dl and HbA1C >6.5% at Day 1
- have had a cosmetic procedure including liposuction/liposculpture of the thighs, buttocks, hips and/or abdomen

#### **Metabolic Syndrome**

- Diagnosis of Metabolic Syndrome is defined as follows per joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity.
- Three abnormal findings out of the following five qualifies a person for the metabolic syndrome:
  - Elevated waist circumference
     Males: ≥102 cm (≥40 in)
     Females: ≥88 cm (≥35 in)
  - Elevated triglycerides≥150 mg/dL (1.7 mmol/L)
  - Reduced HDL-C
     Males: < 40 mg/dL (1.0 mmol/L)</li>
     Females: < 50 mg/dL (1.3 mmol/L)</li>
  - Elevated blood pressure (meeting either or both criteria)
     Systolic ≥130 and/or diastolic ≥ 85 mm Hg
  - Elevated fasting glucose
     ≥ 100 mg/dL

#### BMI (For Shift Table)

The following categories will be used for BMI shift tables:

<Normal: <18.5 kg/m²
Normal: 18.5 - <25 kg/m²
Overweight: 25 - <30 kg/m²
Obese: >= 30 kg/m²

#### 16.6.5. Pharmacokinetic

N/A.

#### 16.6.6. Health Outcomes

# HIVTSQs CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded. Treatment Satisfaction Score

- Total Treatment Satisfaction Score is computed with items 1-11. Items 1-11 are summed to produce a score with a possible range of 0 to 66.
- Item 12 will not be included in Total Treatment Satisfaction Score. Instead, it will be treated
  as a stand-alone item only.
- Higher scores represent greater treatment satisfaction as compared to the past few weeks.
- A maximum of 5 items can be missing, which can be imputed to reflect the mean of the completed item scores. If 6 or more items are missing, then the treatment satisfaction scale score should not be computed.

#### Individual Item Scores

- Items are rated as 6 ccl
  - CCI
- Higher scores represent greater satisfaction with each aspect of treatment
- For individual item scores outputs, missing scores will not be computed (according to Page)





| Lower scores represent worse perception of injection | |
|---|---|
| <ul> <li>For individual item scores outputs, missing scores will not be computed.</li> <li>CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected</li> </ul> | |
| by third party copyright laws and therefore have been excluded. | naide or indices, which are protected |
| CCI | |





#### 16.6.7. Viral Genotype and Phenotype

#### Genotype

#### **Amino Acid Changes**

- A mutation is considered present whenever the encoded amino acid residue differs from the amino acid that would have been encoded by the wild-type (e.g., HXB2, NL43) comparator gene; e.g., Q148K.
- If the encoded amino acid is seen as a mixture of wild-type and mutant amino acid, e.g., Q148Q/K, the mutated amino acid is considered present at the codon of interest.
- If the encoded amino acid is seen as a mixture of two or more amino acids, which may or
  may not include wild type, e.g., Q184K/H or Q184K/H/Q, etc., for the purposes of calculating
  the number of mutated amino acids, only one mutation is considered to be present at the
  codon of interest.

#### Representation of Amino Acid Changes

| Mutations | Amino acid change |
|---|---|
| T69S | Single mutation from amino acid 'T' (vendor reference) to 'S' (sample) at codon '69' |
| Q148H/K/R | Mixture of amino acid mutations 'H', 'K' and 'R' (sample) from amino acid 'Q' (vendor reference) at codon '148' |
| _69_1T | First insertion of amino acid 'T' (sample) at codon '69' |
| _69_2S | Second insertion of amino acid 'S' (sample) at codon '69' |
| _69_3S/A | Third insertion of a mixture of amino acids 'S' and 'A' (sample) at codon '69' |
| L74L/- | Mixture of amino acid 'L' (sample) and a deletion at codon '74' |
| V75- | Single deletion of amino acid (sample) at codon '75' |

#### Resistance Associated Mutations

 Known INI mutations associated with the development of resistance to BIC, RAL, EVG, CAB or DTG:

| HIV Integrase for<br>Analysis | H51Y, T66A/I/K, E92Q/V/G, Q95K, T97A, G118R, F121C/Y, E138A/K/T, G140A/C/R/S, Y143C/H/R/K/S/G/A, P145S, Q146P, S147G, Q148H/K/R/N, V151L/A, S153F/Y, N155H/S/T, E157Q, G163R/K, S230R, D232N, R263K, L68V/I*, L74I/M*, E138D*, V151I*, G193E* |
|---|---|

Notes:

- Draft listing; may be modified in case of additional substantive data availability.
- INI mutations listed taken from Stanford HIV Resistance Database (http://hivdb.stanford.edu/DR/cgi-bin/rules\_scores\_hivdb.cgi?class=INI cited 22Feb2021)
- INI substitutions listed above in bold had a score of =60.
   \*Denotes additional INI mutations added as they were identified during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (ING112574).
- Major resistance mutations to other classes (i.e., NRTI, NNRTI, PI) as defined by the International Antiviral Society-USA (IAS-USA). The most up to date IAS-USA guidelines available at the time of DBF will be used in the analysis [Wensing, 2019].

| | are an area area area area area area are |
|---|---|
| Class | Mutations |
| NRTIs | M41L, A62V, K65R/E/N, D67N, 69 insert, K70E/R, L74V, V75I, F77L, Y115F, F116Y, |
| | Q151M, M184V/I, L210W, T215Y/F, K219Q/E |
| NNRTIs | L100I, K101E/P, K103N/S, V106A/M, V108I, E138/A/G/K/Q/R, V179L, |
| | Y181C/I/V, Y188C/L/H, G190S/A, H221Y, P225H, F227C, M230I/L, |
| Pls | D30N,V32I , M46I/L, I47A/V, G48V, I50V/L, I54M/L/V, Q58E, T74P, L76V, |
| | V82A/T/F/L/S, N83D, I84V, N88S,L90M |

Note: List generated from IAS\_USA Guideline, [Wensing. 2019]

- The pre-specified INI Mutations are identified as below:
  - Per the IAS-USA list of mutations (both minor and major) associated with resistance to Bictegravir, Cabotegravir, Dolutegravir, Elvitegravir, or Raltegravir (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019): T66A/I/K, L74M, E92Q/G, T97A, G118R, F121Y, E138A/K/T, G140A/C/R/S, Y143C/H/R, S147G, Q148H/K/R, S153F/Y, N155H, R263K
  - Observed mutations during in vitro passage of DTG or seen in a previous DTG study in INI-experienced subjects (study ING112574): H51Y, L74I, L68V/I, E92V, Q95K, E138D, Y143K/S/G/A, P145S, Q146P, V151I/L/A, N155S/T, E157Q, G163R/K, G193E, S230R
  - Mutations per FDA request for Study 201584: Q146L, T124A
- The NNRTI resistance associated mutations (RAMs) are identified per IAS-USA NNRTI mutations (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019):
  - V90I, A98G, L100I, K101E/H/P, K103N/S, V106A/I/M/T, V108I, E138A/G/K/Q/R, V179D/F/L/T, Y181C/I/V, Y188C/H/L, G190A/E/S, H221Y, P225H, F227C/L/R, M230I/L, L234I
- The RPV RAMs are identified per IAS-USA NNRTI mutations (IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019):
  - L100I, K101E/P, E138A/G/K/Q/R, V179L, Y181C/I/V, Y188L, H221Y, F227C, M230I/L
- The NRTI major mutations associated with resistance to BIKTARVY (Emtricitabine and Tenofovir, IAS-USA 2019 resistance mutations update volume 27 issue 3, 2019):
  - K65R/E/N, K70E, M184V/I

#### Phenotype

#### Phenotypic Susceptibility

Phenotypic susceptibility to all licensed antiretroviral drugs and CAB will be determined using PhenoSense HIV assays from Monogram Inc. and will be reported as fold change (FC) in IC50

- relative to wild-type control virus NL4-3, i.e., FC of sample virus = IC50 of sample virus/IC50 of control virus.
- Since the maximum assay limit for FC for each ART varies from assay to assay, FC values that are greater than the maximum assay limit (e.g., '>100') will be interpreted as having a value equal to the smallest maximum assay limit for that ART in the study population for data analysis. Censored values will be presented 'as is' in the listings. Phenotypic susceptibilities will be categorised according to FC as shown in Table below (based on Monogram PhenoSense assay). Clinical cutoffs (where available) or biological cutoffs by PhenoSense will be used to define the phenotypic susceptibility of background treatment by Monogram. PHENOTYP dataset from Monogram contains the phenotypic susceptibility information derived from the cutoff listed below. Thus, phenotypic susceptibility (i.e. full sensitivity and partial sensitivity) will not be re-derived in our analysis.
- Replication capacity is generated as part of standard phenotypic assays

**PhenoSense Algorithm** 

| Drug | Abbreviation | Class | PhenoSense cutoff |
|---|---|---|---|
| Abacavir | ABC | NRTI | (4.5 – 6.5) <sup>a</sup> |
| Lamivudine | 3TC | NRTI | 3.5 a |
| Didanosine | ddl | NRTI | (1.3 – 2.2) a |
| Stavudine | d4T | NRTI | 1.7 a |
| Zidovudine | AZT (ZDV) | NRTI | 1.9 |
| Emtricitabine | FTC | NRTI | 3.5 |
| Tenofovir | TDF | NRTI | (1.4 – 4) a |
| Delavirdine | DLV | NNRTI | 6.2 |
| Efavirenz | EFV | NNRTI | 3 |
| Nevirapine | NVP | NNRTI | 4.5 |
| Etravirine | ETR | NNRTI | (2.9-10) a |
| Rilpivirine | RPV | NNRTI | 2.0 |
| Doravirine | DOR | NNRTI | 3.0 |
| Fosamprenavir/r | FPV/r | PI | (4-11) a |
| Atazanavir | ATV | PI | 2.2ª |
| Atazanavir/r | ATV/r | PI | 5.2ª |
| Indinavir/r | IDV/r | PI | 10 a |
| Lopinavir/r | LPV/r | PI | (9 – 55) a |
| Nelfinavir | NFV | PI | 3.6 |
| Saquinavir/r | SQV/r | PI | (2.3 – 12) a |
| Tipranavir/r | TPV/r | PI | (2 – 8) a |
| Darunavir/r | DRV/r | PI | (10 – 90) a |
| Ritonavir | RTV | PI | 2.5 |
| Enfuvirtide | T20 | FI | 6.48 |
| Cabotegravir | CAB | INI | 2.5 |
| Raltegravir | RAL | INI | 1.5 |
| Elvitegravir | EVG | INI | 2.5 |
| Dolutegravir | DTG | INI | (4-13) a |
| Bictegravir | BIC | INI | (2.5- 10) |
| a. clinical cutoff (lower | cutoff – higher cutoff). | | |

Phenotypic susceptibility to each drug in a subject's background regimen will be determined by applying drug-associated cutoffs as defined by the PhenoSense algorithm to the phenotypic fold resistance to that drug at a certain timepoint (e.g. Screening or Baseline).

#### **Full Sensitivity**

| Fold Change | Interpretation |
|--------------------------------------------|----------------|
| > clinical lower cutoff or biologic cutoff | resistance |
| ≤ clinical lower cutoff or biologic cutoff | sensitive |

#### **Partial Sensitivity**

| Fold Change | Interpretation |
|------------------------------------------------------|---------------------|
| > clinical higher cutoff | resistance |
| ≤ clinical higher cutoff and > clinical lower cutoff | partially sensitive |
| ≤ clinical lower cutoff | sensitive |

#### **Genotypic and Net Assessment Susceptibility**

Genotypic and Net assessment susceptibility to all licensed antiretroviral drugs and CAB will be determined from Monogram Inc. Net assessment susceptibility will be reported with the categories of 'resistant', 'partially sensitive', and 'sensitive' as what will be performed for phenotypic susceptibility. Genotypic susceptibility will be reported with the categories of 'resistant', 'resistance possible' and 'sensitive'. Genotypic and Net assessment susceptibility will be assessed at time of CVF using plasma sample, Genotypic susceptibility may be assessed at baseline using PBMC.

# 16.7. Appendix 7: Reporting Standards for Missing Data

# 16.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Participants are considered to have completed the study if they remain on therapy (i.e., have not permanently discontinued IP) and satisfy one of the following: <ul> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Month 11/12 visits (with or without Month 11/12 study treatment) and did not enter the Extension Phase;</li> <li>Randomly assigned to either treatment group, completed the randomized Maintenance Phase including Month 13, entered and completed the Extension Phase (defined as remaining on study until commercial supplies of the CAB LA + RPV LA Q8W regimen become locally available or development of CAB LA + RPV LA is terminated).</li> </ul> </li> </ul> |
| | Participants who withdraw from CAB LA + RPV LA and go into the Long-Term Follow Up Phase will be considered to have prematurely withdrawn from the study, even if they complete the 52-week follow-up Phase. |
| | In addition to the 52-week Follow-Up phase required for participants who receive one or more injections with CAB LA or RPV LA, an in-clinic Follow-Up visit will be conducted approximately 4 weeks after the last dose of study medication for participants who withdraw during the oral lead-in phase and who were randomized to BIK with ongoing AEs, serious adverse events (SAEs) and any laboratory abnormalities that are considered to be AEs or potentially harmful to the participant, at the last on-study visit. Assessments at the Follow-up visit should reflect any ongoing complaints (e.g., blood draws to follow a laboratory abnormality). Follow-Up visits are not required for successful completion of the study. |
| | <ul> <li>Withdrawn subjects were not replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |
| | <ul> <li>Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be<br/>summarised as withdrawal visits.</li> </ul> |

# 16.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in participant listing displays.</li> </ul> |
| | Unless all data for a specific visit are missing in which case the data is excluded from the table. |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 16.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in participant listing displays. |
| Adverse Events | Partial dates will be displayed as captured in participant listing displays. The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment State. Missing Stop Day: Last day of the month will be used, unless this is after the last contact date; in this case the last contact date will be used. Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be |
| | missing. |
| Concomitant<br>Medications/Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>For medications recorded in the eCRF as prior ART, the earlier of this imputed date or the day before Screening date will be used.</li> </ul> </li> <li>For medications with completely missing start date, they will be considered started prior to the maintenance phase treatment start date.</li> <li>For medications with completely missing stop date, they will be considered ongoing unless recorded in eCRF as prior.</li> <li>For ART booster medications, the start and stop dates are not recorded in the database (i.e. missing), the dates will be imputed to be the same as the dates of their parent medications.</li> <li>The recorded partial or missing date will be displayed in listings.</li> </ul> |
| Health outcomes | For the summary of individual item scores outputs, missing scores will not be computed. |

# 16.7.2.2. Handling of Missing data for Statistical Analysis

| Element | Reporting Detail |
|---|---|
| Snapshot | <ul> <li>In the Snapshot dataset, participants without HIV-1 RNA data in the assessment<br/>window for the visit of interest (due to missing data or discontinuation of IP prior to<br/>the visit window) do not belong to 'HIV-1 RNA &lt; 50 c/mL (or &lt;200 c/mL)'. The nature<br/>of this missing data will be further classified in Snapshot summaries as either 'HIV-1<br/>RNA≥50' or 'No Virologic Data at Week X'. See Appendix 9: Snapshot Algorithm<br/>Details.</li> </ul> |
| Lipid<br>Evaluable | <ul> <li>For subjects with lipid-modifying agent use, lipid assessments will be considered<br/>non-evaluable (equal to missing) after initiation without any imputation.</li> </ul> |
| | <ul> <li>If participants take lipid modifying agents within 12 weeks prior to the start of the<br/>study treatment, all the post-baseline values will be non-evaluable.</li> </ul> |
| | The lipid evaluability rules will be used for the following displays: Summary of Fasting TC/HDL ratio Change from Baseline Summary of Fasting Lipids Percentage Changes from Baseline Summary of Chemistry Changes from Baseline |
| | <ul> <li>All other displays of lipids (i.e. toxicity tables and NCEP tables) will use observed<br/>fasting data, without considering lipid evaluability.</li> </ul> |
| | <ul> <li>The same rule of "lipid evaluable" will be applied to anthropometric parameters as<br/>specified in Section 8.5.3:</li> </ul> |
| | <ul> <li>Weight, Height and BMI</li> <li>Waist circumferences</li> <li>Hip circumference</li> </ul> |
| | Tanita scale parameters (total body fat percent, total body water percent, muscle mass, and bone mineral mass). |

# 16.8. Appendix 8: Values of Potential Clinical Importance

| Element | Reporting Detail |
|---|---|
| Laboratory<br>Values and<br>Adverse Events | <ul> <li>The DAIDS grading for severity of laboratory toxicities and clinical adverse events is included in the protocol.</li> <li>The central laboratory will flag lab parameter toxicities directly in the provided</li> </ul> |
| | datasets. |
| ECG values | • Defined as QTc > 500 msec or increase from baseline in QTc ≥ 60 msec |

#### 16.9. Appendix 9: Snapshot Algorithm Details

o HIV-1 RNA < 50 c/mL o HIV-1 RNA  $\geq$  50 c/mL

#### **Detailed Algorithm Steps**

- Consider an analysis visit window for Month X as defined in Section 16.3.1
- The HIV-1 RNA threshold of 50, 200 copies/mL will be analysed, respectively, in this study.

Data in window not below threshold

• The COVID-19 pandemic presents significant logistical challenges for many clinical sites around the world, with variable restrictions being placed on site resources and operations, and on an individual participant's ability to attend clinic visits. The snapshot algorithm is modified to allow for the presentation of full scope of COVID-19 relatedness. The analysis window 'Week 48' and HIV-1 RNA threshold of '50 c/mL' are used for the purpose of illustration. A participant's Snapshot response and reason at Week 48 are categorized as below.

```
Non-COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below threshold
         Change in background therapy*
     COVID-19 related
         Discontinued for lack of efficacy
         Discontinued for other reason while not below threshold
         Change in background therapy*
o No Virologic Data at Week 48 Window
     Non-COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reasons
         Not evaluated or discontinued due to confirmed pregnancy**
         On study but missing data in window
        COVID-19 related
         Discontinued study due to AE or death
         Discontinued study for other reason
```

On study but missing data in window

- Note: since permanent changes in ART are not permitted in this protocol, all such participants who permanently change ART will be considered 'HIV-1 RNA ≥ 50 c/mL' if the change is made prior to an analysis timepoint. Participants with protocol permitted oral bridging treatment, CAB+RPV or SOC (during COVID-19 pandemic due to the unavailability of the CAB/RPV IM injections and oral CAB+RPV), or a temporary change in ART by mistake prior to an analysis timepoint (e.g. participant took the ART different from study treatment during oral lead-in by mistake for a short period of time and then went back to the study treatment) will not be considered 'HIV-1 RNA ≥ 50 c/mL' due to 'change in ART'.
- The steps in determining response and reasons are indicated in Table below, in the order stated.
- \*Background therapy is not given to participants while on study. The "change in background therapy" in detailed steps below refers to the "change in ART" in this study.
- \*\* This category is not needed if no subject on the Q2M arm becomes pregnant and continues in the study.

#### **Detailed steps**

Please note that the following scenarios will NOT be penalized per Snapshot algorithm (i.e. please exclude these scenarios from Conditions 1-4).

- Dose reduction, dropping a component, or change in formulation (e.g. 'Tivicay + Kivexa' to 'Triumeq' with the identical ingredients)
- Protocol permitted temporary oral bridging, or temporary change in ART by mistake

| Condition ('Week 48' indicates Week 48 window) | Response | Reasons |
|---|---|---|
| 1. If non-permitted change in background therapy prior to Week 48 | | |
| o not due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (non-COVID-19 related) |
| o due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
| 2. If permitted change <sup>[a]</sup> in background therapy prior to Week 48 AND the la study) | test on-treatment VL prior to/on the | e date of change is ≥ 50 c/mL (NA to this |
| o not due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (non-COVID-19 related) |

| o due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
|---|---|---|
| 3. If non-permitted change in background therapy during Week 48 | | |
| <ul> <li>○ Last on-treatment VL during Week 48 prior to/on the date of change ≥</li> <li>50 c/mL</li> </ul> | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| <ul> <li>Last on-treatment VL during Week 48 prior to/on the date of change &lt;</li> <li>50 c/mL</li> </ul> | HIV-1 RNA < 50 | |
| <ul> <li>No VL during Week 48 prior to/on the date of change and the change in<br/>background therapy is not due to COVID-19</li> </ul> | HIV-1 RNA ≥ 50 | Change in background therapy (Non-COVID-19 related) |
| <ul> <li>No VL during Week 48 prior to/on the date of change and the change in<br/>background therapy is due to COVID-19</li> </ul> | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
| 4. If permitted change <sup>[a]</sup> in background therapy during Week 48 AND the last on-trea study) | tment VL prior to/on th | ne date of change is ≥ 50 c/mL (NA to this |
| 4.1 This last on-treatment VL occurs prior to Week 48 | | |
| The change in background therapy is not due to COVID-19 | HIV-1 RNA ≥ 50 | Change in background therapy (non-COVID-19 related) |
| <ul> <li>The change in background therapy is due to COVID-19</li> </ul> | HIV-1 RNA ≥ 50 | Change in background therapy (COVID-19 related) |
| 4.2 This last on-treatment VL occurs during Week 48 but prior to/on the date of change | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| 5. If none of the above conditions met | <u> </u> | |
| 5.1 On-treatment VL available during Week 48 | | |
| <ul> <li>Last on-treatment VL during Week 48 ≥ 50 c/mL</li> </ul> | HIV-1 RNA ≥ 50 | Data in window not below 50 |
| Last on-treatment VL during Week 48 < 50 c/mL | HIV-1 RNA < 50 | |
| 5.2 No on-treatment VL during Week 48 | | |
| 5.2.1 If participants are still on study, i.e. a participant has not permanently discontinued the study treatment yet, or if a participant permanently discontinued | | |

| the study treatment and the upper bound of analysis snapshot window is prior to t | h | |
|---|---|---|
| following date: | | |
| For Q2M arm: Min[max(Date of last CAB/RPV LA Dose + 67, Date of last oral dose+1), withdrawal date] | | |
| For BIK arm: Min (BIK Stop Date + 1, withdrawal date) | | |
| Note: | | |
| <ul> <li>Last oral dose: may be CAB/RPV or SOC ART Oral Bridging where<br/>CAB/RPV is not available due to COVID-19 impact.</li> </ul> | | |
| Withdrawal Date: date the participant failed to complete per corresponding conclusion form | | |
| 5.2.1.1 If no on-treatment VL during Week 48 is not due to COVID-19 | | |
| If no on-treatment VL is not due to confirmed pregnancy | No virologic data at<br>Week 48 Window | On study but missing data in window (Non-COVID-19 related) |
| <ul> <li>If no on-treatment VL is due to confirmed pregnancy ("while on-<br/>treatment": data not evaluable)</li> </ul> | No virologic data at<br>Week 48 Window | Not evaluated or discontinued due to confirmed pregnancy(Non-COVID-19 related) |
| 5.2.1.2 If no on-treatment VL during Week 48 is due to COVID-19 | No virologic data at<br>Week 48 Window | On study but missing data in window (COVID-19 related) |
| 5.2.2 If participants withdraw before/during Week 48 due to | | |
| 5.2.2.1 Non-COVID-19 related safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc, as recorded in eCRF Conclusion form) | No virologic data at<br>Week 48 Window | Disc due to AE/death (Non-COVID-19 related) |
| <u>'</u> | | |

| 5.2.2.2 COVID-19 related safety reasons (e.g. AE/death, liver chemistry stopping criteria, renal toxicity withdrawal criteria, QTc withdrawal criteria etc, as recorded in eCRF Conclusion form) | No virologic data at<br>Week 48 Window | Disc due to AE/death (COVID-19 related) |
|---|---|---|
| 5.2.2.3 Non-safety and Non-COVID-19 related reasons (e.g. Lack of efficacy, protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc, as recorded in eCRF Conclusion Form) | | |
| <ul> <li>Last on-treatment VL &lt;50 c/mL OR no on-treatment VL</li> </ul> | | |
| available during study • Withdrew not due to pregnancy | No virologic Data at<br>Week 48 Window | Disc for other reasons (Non-COVID-19 related) |
| Withdrew due to pregnancy | No virologic Data at<br>Week 48 Window | Not evaluated or discontinued due to confirmed pregnancy(Non-COVID-19 related) |
| ° Last on-treatment VL ≥ 50 c/mL AND withdrawal due to | HIV-1 RNA ≥ 50 | Disc. for lack of efficacy (Non-COVID- |
| Lack of efficacy | | 19 related) |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND withdrawal due to<br/>all other non-safety related reasons</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for other reason while not below 50 (Non-COVID-19 related) |
| 5.2.2.4 Non-safety and COVID-19 related reasons (e.g. protocol deviation, withdrew consent, loss to follow-up, study closed/terminated, investigator discretion etc., as recorded in eCRF Conclusion Form) | | |
| Last on-treatment VL <50 c/mL OR no on-treatment VL available during study | No virologic Data at<br>Week 48 Window | Disc for other reasons (COVID-19 related) |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND withdrawal due to Lack<br/>of efficacy</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for lack of efficacy (COVID-19 related) |
| <ul> <li>Last on-treatment VL ≥ 50 c/mL AND withdrawal due to all<br/>other non-safety related reasons</li> </ul> | HIV-1 RNA ≥ 50 | Disc. for other reason while not below 50 (COVID-19 related) |

#### **Examples from FDA guidance**

#### Data in Window

Virologic outcome should be determined by the last available measurement while the patient is on treatment and continued on trial within the time window:

HIV-RNA = 580 copies/mL at Day 336, HIV-RNA below 50 copies/mL on Day 350. This should be categorized as HIV-RNA below 50 copies/mL.

#### No Data in Window

Discontinued study due to Adverse Event or Death:

- Any patient who discontinues because of an AE or death before the window should be classified as Discontinued due to AE or Death (as appropriate), regardless
  of the HIV-RNA result, even if the HIV-RNA is below 50 copies/mL at the time of discontinuation.
- However, if a patient has an HIV-RNA value in the time window and also discontinues in the time window, the viral load data should be used to classify the patient's response. This is the Virology First hierarchy:
- HIV-RNA below 50 copies/mL at Day 336 and discontinues because of AE or even dies on Day 360 this person is categorized as having HIV-RNA below 50 copies/mL.
- HIV-RNA is 552 copies/mL on Day 336 and the patient discontinues on Day 360, the patient is categorized as having HIV-RNA greater than or equal to 50 copies/mL.

#### Discontinued for Other Reasons:

- Only patients who have achieved virologic suppression can be counted as *Discontinued for Other Reasons*.
- If a patient discontinues the study before the time window because of *lack of efficacy* then the patient should be included in the HIV-RNA greater than or equal to 50 row and not in the Discontinued for Other Reasons row.
- If a patient discontinues because of *subject withdrew consent* and his or her HIV-1 RNA result at the time of discontinuation was equal to or above 50 copies/mL, then he or she should be categorized as HIV-RNA greater than or equal to 50 and NOT as Discontinued for Other Reasons.
- If a patient discontinued because of *Lost to Follow-Up* and the last HIV-RNA result was 49 copies/mL, then the patient can be categorized as Discontinued for Other Reasons.
- If patients changed background treatment not permitted by protocol— they should be considered an efficacy failure and captured in the HIV-RNA greater than or equal to 50 copies/mL row.

#### On study but missing data in window:

• If there are no data during Days 294 to 377, but there is an HIV-RNA below 50 copies/mL on Day 380, this patient should be considered *On Study but Missing Data in Window.* 

#### CONFIDENTIAL

213500

• If there are no data during Days 294 to 377, but there is an HIV-RNA equal to or above 50 copies/mL on Day 280, this patient also should be classified as On Study but Missing Data in Window.

Not evaluated due to confirmed pregnancy:

Q2M subjects who became pregnant on study will be allowed to continue study treatment whereas BIK subjects will be withdrawn. HIV-1 RNA data will be treated as non-evaluable after confirmed pregnancy date as recorded on the eCRF, if a pregnant Q2M subject is allowed to continue.

# 16.10. Appendix 10: Variables Defined for Time to Event Analysis

| Programming Instructions for the Kaplan-Meier a | nalysis of treatme | nt-related discontinuation equals failure (TRDF) |
|---|---|---|
| Condition | Censor Status | Event Description/AVAL |
| Participant met CVF event criteria during the Maintenance Phase (based on derived CVF) | CNSR=0 | EVNTDESC=CVF AVAL=Study Day of SVF* *immediately preceding CVF |
| 2. Participant with Maintenance Phase withdrawal due to 'Lack of Efficacy', 'Treatment Related AE', 'Intolerability due to Injection', or 'Protocol Defined Safety Stopping Criteria' during Maintenance Phase Note: primary reason and/or standardized subreason for discontinuation based on Maintenance Conclusion form in the eCRF. 'Protocol Defined Safety Stopping Criteria' includes GSK defined liver chemistry stopping criteria, renal toxicity criteria and QTc withdrawal criteria. Treatment Related AE' is defined as participants who have primary reason for withdrawal =AE and who have at least one AE considered drug related and leading to withdrawal/permanent discontinuation of investigational product. | CNSR=0 | For Q2M arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, Study day of Starting LTFU HAART if applicable, max(Study Day of Last Maintenance Q2M IM Dose + 67, Study Day of Last Maintenance Oral Dose + 1)] For BIK arm: AVAL= min [Study Day of Maintenance Phase Discontinuation, Study Day of Maintenance IP Stop Date + 1] Note: Last Q2M IM / last oral dose/ Maintenance IP Stop Date only applies to subjects who permanently discontinue from study treatment. Date of Maintenance Phase discontinuation is from the Maintenance Phase Conclusion form in the eCRF. |
| If none of the above conditions met | | |
| Participant with Maintenance Phase withdrawal due to other reasons | CNSR=1 | EVNTDESC='Censored due to Study Discontinuation for Other Reasons' AVAL will be defined as the same as above 2 |
| Participant who did not have premature withdrawal from the Maintenance Phase | CNSR=1 | EVNTDESC='Censored due to data cutoff for analysis' |

| Condition | Censor Status | analysis of treatment-related discontinuation equals failure (TRDF) Censor Status Event Description/AVAL |
|---|---|---|
| | | AVAL = Study Day of last on-treatment date during the maintenance phase, which is defined as follows: |
| | | For Q2M arm: min [Study Day of Month 13(D2I)/14(OLI) Visit, Study Day of Starting LTFU HAART, Study Day of Last Contact Date at time of analysis, max(Study Day of Last Maintenance Q2M IM Dose + 67, Study Day of Last Maintenance oral dose + 1)] |
| | | For BIK arm: min [Study Day of Month 13 Visit, Day of Last Contact at time of analysis, Study Day of Maintenance IP stop Date + 1] |
| | | Note: • Last Q2M IM / last oral dose/ Maintenance IP Stop Date only applies to subjects who permanently discontinue from study treatment |

<sup>\*</sup>Last oral dose may be CAB/RPV or SOC ART Oral Bridging where CAB/RPV is not available due to COVID-19 impact.

Note that last injection and last oral dose mentioned above are only applied to participants who permanently discontinued from the study treatment.

The similar approach will be used to derive for Kaplan-Meier analysis of efficacy-related discontinuation equals failure (ERDF), except that the reason of withdrawal in Condition 2 will be restricted to 'Lack of Efficacy'.

# 16.11. Appendix 11: Identification of Adverse Events of Special Interest (AESI)

The adverse events of special interest are identified based on MedDRA coded values and/or AE data available in the study database. The PT terms and codes below are from MedDRA 24.1. SMQs use narrow terms unless otherwise specified. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. Additional events may be added based on the blinded review of AE data collected on study prior to the database freeze.

#### 16.11.1. Hepatic Safety Profile

#### Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions (SMQ)

| PT | PT Code |
|----------------------------------------------------|----------|
| Acquired hepatocerebral degeneration | 10080860 |
| Acute hepatic failure | 10000804 |
| Acute on chronic liver failure | 10077305 |
| Acute yellow liver atrophy | 10070815 |
| Ascites | 10003445 |
| Asterixis | 10003547 |
| Bacterascites | 10068547 |
| Biliary cirrhosis | 10004659 |
| Biliary fibrosis | 10004664 |
| Cardiohepatic syndrome | 10082480 |
| Cholestatic liver injury | 10067969 |
| Chronic hepatic failure | 10057573 |
| Coma hepatic | 10010075 |
| Cryptogenic cirrhosis | 10063075 |
| Diabetic hepatopathy | 10071265 |
| Drug-induced liver injury | 10072268 |
| Duodenal varices | 10051010 |
| Flood syndrome | 10084797 |
| Gallbladder varices | 10072319 |
| Gastric variceal injection | 10076237 |
| Gastric variceal ligation | 10076238 |
| Gastric varices | 10051012 |
| Gastric varices haemorrhage | 10057572 |
| Gastrooesophageal variceal haemorrhage prophylaxis | 10066597 |
| Hepatectomy | 10061997 |
| Hepatic atrophy | 10019637 |
| Hepatic calcification | 10065274 |
| Hepatic cirrhosis | 10019641 |

| PT | PT Code |
|------------------------------------|----------|
| Hepatic encephalopathy | 10019660 |
| Hepatic encephalopathy prophylaxis | 10066599 |
| Hepatic failure | 10019663 |
| Hepatic fibrosis | 10019668 |
| Hepatic hydrothorax | 10067365 |
| Hepatic infiltration eosinophilic | 10064668 |
| Hepatic lesion | 10061998 |
| Hepatic necrosis | 10019692 |
| Hepatic steato-fibrosis | 10077215 |
| Hepatic steatosis | 10019708 |
| Hepatitis fulminant | 10019772 |
| Hepatobiliary disease | 10062000 |
| Hepatocellular foamy cell syndrome | 10053244 |
| Hepatocellular injury | 10019837 |
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Immune-mediated cholangitis | 10083406 |
| Immune-mediated hepatic disorder | 10083521 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Nonalcoholic fatty liver disease | 10082249 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |

| PT | PT Code |
|---------------------------------------|----------|
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Sugiura procedure | 10083010 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |
| Hepatic cytolysis | 10049199 |
| Spontaneous bacterial peritonitis | 10061135 |

# Hepatitis, non-infectious (SMQ)

| PT | PT Code |
|--------------------------------------------|----------|
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |

| PT | PT Code |
|-------------------------------|----------|
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |
| Hepatic cytolysis | 10049199 |

# 16.11.2. Hypersensitivity Reactions (HSR)

# Drug reaction with eosinophilia and systemic symptoms syndrome (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Pseudolymphoma | 10037127 |
| Granulomatous T-cell pseudolymphoma | 10084214 |

# PTs (select)

| PT | PT Code |
|-----------------------------------|----------|
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |
| Periorbital swelling | 10056647 |
| Swelling of eyelid | 10042690 |
| Polymers allergy | 10086347 |

16.11.3. Rash

# Severe cutaneous adverse reactions (SMQ)

| PT | PT Code |
|-------------------------------------------------------|----------|
| Acute generalised exanthematous pustulosis | 10048799 |
| Bullous haemorrhagic dermatosis | 10083809 |
| Cutaneous vasculitis | 10011686 |
| Dermatitis bullous | 10012441 |
| Dermatitis exfoliative | 10012455 |
| Dermatitis exfoliative generalised | 10012456 |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 |
| Epidermal necrosis | 10059284 |
| Erythema multiforme | 10015218 |
| Erythrodermic atopic dermatitis | 10082985 |
| Exfoliative rash | 10064579 |
| Oculomucocutaneous syndrome | 10030081 |
| SJS-TEN overlap | 10083164 |
| Skin necrosis | 10040893 |
| Stevens-Johnson syndrome | 10042033 |
| Target skin lesion | 10081998 |
| Toxic epidermal necrolysis | 10044223 |
| Toxic skin eruption | 10057970 |
| Generalised bullous fixed drug eruption | 10084905 |
| Severe cutaneous adverse reaction | 10085778 |

# PTs (Select)

| PT | PT Code |
|----------------------|----------|
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |

| PT | PT Code |
|---------------------|----------|
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

# 16.11.4. Prolongation of the Corrected QT Interval of the ECG in Supratherapeutic Doses

# Torsade de pointes/QT prolongation (SMQ)

| PT | PT Code |
|----------------------------------------|----------|
| Electrocardiogram QT interval abnormal | 10063748 |
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |

# PTs (Selective)

| PT | PT Code |
|----------------------------------------------|----------|
| Electrocardiogram repolarisation abnormality | 10052464 |

#### 16.11.5. Suicidal Ideation/Behaviour

### Suicide/self-injury (SMQ)

| PT | PT Code |
|-------------------------------------------------|----------|
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |

| PT | PT Code |
|---------------------------|----------|
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |
| Suspected suicide | 10082458 |
| Suspected suicide attempt | 10081704 |

# 16.11.6. Depression

# Depression (excl suicide and self injury) (SMQ)

| PT | PT Code |
|-----------------------------------------------------------|----------|
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depression rating scale score increased | 10084390 |
| Depressive symptom | 10054089 |
| Discouragement | 10084257 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

# 16.11.7. Bipolar Disorder

# **HLGT Manic and Bipolar mood disorders and disturbances**

| PT | PT Code |
|----------------------|----------|
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |
| Manic symptom | 10084119 |

# 16.11.8. Psychosis

# Psychosis and psychotic disorders (SMQ)

| PT | PT Code |
|---------------------------------------------------|----------|
| Acute psychosis | 10001022 |
| Alcoholic psychosis | 10001632 |
| Alice in wonderland syndrome | 10001666 |
| Brief psychotic disorder with marked stressors | 10048549 |
| Brief psychotic disorder without marked stressors | 10056395 |
| Brief psychotic disorder, with postpartum onset | 10006362 |
| Charles Bonnet syndrome | 10063354 |
| Childhood psychosis | 10061040 |
| Clang associations | 10009232 |
| Cotard's syndrome | 10059591 |
| Delusion | 10012239 |
| Delusion of grandeur | 10012241 |
| Delusion of parasitosis | 10012242 |
| Delusion of reference | 10012244 |
| Delusion of replacement | 10012245 |
| Delusion of theft | 10084030 |
| Delusional disorder, erotomanic type | 10012249 |
| Delusional disorder, grandiose type | 10012250 |
| Delusional disorder, jealous type | 10012251 |
| Delusional disorder, mixed type | 10012252 |
| Delusional disorder, persecutory type | 10053195 |
| Delusional disorder, somatic type | 10012254 |
| Delusional disorder, unspecified type | 10012255 |
| PT | PT Code |
|-------------------------------------------------------|----------|
| Delusional perception | 10012258 |
| Dementia of the Alzheimer's type, with delusions | 10012295 |
| Depressive delusion | 10063033 |
| Derailment | 10012411 |
| Epileptic psychosis | 10059232 |
| Erotomanic delusion | 10015134 |
| Flight of ideas | 10016777 |
| Hallucination | 10019063 |
| Hallucination, auditory | 10019070 |
| Hallucination, gustatory | 10019071 |
| Hallucination, olfactory | 10019072 |
| Hallucination, synaesthetic | 10062824 |
| Hallucination, tactile | 10019074 |
| Hallucination, visual | 10019075 |
| Hallucinations, mixed | 10019079 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hysterical psychosis | 10062645 |
| Ideas of reference | 10021212 |
| Illusion | 10021403 |
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |

| PT | PT Code |
|------------------------------------------|----------|
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |
| Negative symptoms in schizophrenia | 10084992 |
| Pseudohallucination | 10066297 |

### 16.11.9. Mood Disorders

#### **HLGT Mood disorders and disturbances**

| PT | PT Code |
|----------------------------------|----------|
| Affect lability | 10054196 |
| Affective ambivalence | 10077173 |
| Affective disorder | 10001443 |
| Alexithymia | 10077719 |
| Anger | 10002368 |
| Apathy | 10002942 |
| Blunted affect | 10005885 |
| Boredom | 10048909 |
| Constricted affect | 10010778 |
| Crying | 10011469 |
| Diencephalic syndrome of infancy | 10012774 |
| Discouragement | 10084257 |
| Dysphoria | 10013954 |
| Emotional disorder | 10014551 |

| PT | PT Code |
|--------------------------------------------------|----------|
| Emotional distress | 10049119 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Flat affect | 10016759 |
| Frustration tolerance decreased | 10077753 |
| Inappropriate affect | 10021588 |
| Irritability | 10022998 |
| Laziness | 10051602 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Moaning | 10027783 |
| Mood altered | 10027940 |
| Mood disorder due to a general medical condition | 10027944 |
| Mood swings | 10027951 |
| Morose | 10027977 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Premenstrual dysphoric disorder | 10051537 |
| Premenstrual syndrome | 10036618 |
| Screaming | 10039740 |
| Seasonal affective disorder | 10039775 |
| Steroid withdrawal syndrome | 10042028 |
| Substance-induced mood disorder | 10072387 |
| Sibling rivalry disorder | 10086385 |

# 16.11.10. Anxiety

## **HLGT Anxiety disorders and symptoms**

| PT | PT Code |
|-------------------------|----------|
| Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10001084 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |

| PT | PT Code |
|-----------------------------------------------------|----------|
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Catastrophic reaction | 10082329 |
| Cibophobia | 10082413 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Cryophobia | 10082662 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of surgery | 10084519 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |

| PT | PT Code |
|------------------------------------------------------------------|----------|
| Haphephobia | 10067580 |
| Herpetophobia | 10081809 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosocomephobia | 10083993 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders associated with | |
| streptococcal infection | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Postpartum anxiety | 10082233 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |

| PT | PT Code |
|--------------------------------|----------|
| Post-traumatic stress disorder | 10036316 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |
| Aichmophobia | 10085292 |
| Olfactory reference syndrome | 10085053 |
| Frigophobia | 10086104 |
| Somniphobia | 10085856 |

# 16.11.11. Sleep Disorders

# **HLGT Sleep Disorders and Disturbances**

| PT | PT Code |
|-------------------------------------------------|----------|
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Exploding head syndrome | 10080684 |
| Hypersomnia | 10020765 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |

| PT | PT Code |
|-------------------------------------------------------------------|----------|
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Insomnia related to another mental condition | 10022443 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Nightmare | 10029412 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Parasomnia | 10061910 |
| Paradoxical insomnia | 10083337 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep attacks | 10040981 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Sopor | 10058709 |
| Stupor | 10042264 |

| PT | PT Code |
|----------------------------------|----------|
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |

# **HLGT Sleep disturbances (incl subtypes)**

| PT | PT Code |
|-------------------------------------------------|----------|
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Advanced sleep phase | 10001423 |
| Behavioural induced insufficient sleep syndrome | 10081938 |
| Behavioural insomnia of childhood | 10072072 |
| Breathing-related sleep disorder | 10006344 |
| Cataplexy | 10007737 |
| Central-alveolar hypoventilation | 10007982 |
| Circadian rhythm sleep disorder | 10009191 |
| Confusional arousal | 10067494 |
| Delayed sleep phase | 10012209 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Hypersomnia | 10020765 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Loss of dreaming | 10065085 |
| Microsleep | 10076954 |
| Middle insomnia | 10027590 |
| Narcolepsy | 10028713 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Shift work disorder | 10078088 |
| Sleep apnoea syndrome | 10040979 |
| Sleep deficit | 10080881 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |

| PT | PT Code |
|----------------------------------|----------|
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Sudden onset of sleep | 10050014 |
| Terminal insomnia | 10068932 |
| Upper airway resistance syndrome | 10063968 |
| Catathrenia | 10085704 |

### 16.11.12. Injection Site Reactions (ISR)

ISR data available in the database, i.e. data collected from non-serious ISR AE eCRF form and collected serious adverse events with 'STUDY DRUG INJECTION SITE' included in the AE term.

#### 16.11.13. Seizures and Seizure-like Events

#### Convulsions (SMQ)

| PT | PT Code |
|-----------------------------------------------------------------|----------|
| 1p36 deletion syndrome | 10082398 |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Alpers disease | 10083857 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| CEC syndrome | 10083749 |
| CDKL5 deficiency disorder | 10083005 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Congenital bilateral perisylvian syndrome | 10082716 |
| Convulsion in childhood | 10052391 |

| PT | PT Code |
|-----------------------------------------------------------------|----------|
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epilepsy with myoclonic-atonic seizures | 10081179 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Faciobrachial dystonic seizure | 10084187 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Gelastic seizure | 10082918 |
| Generalised onset non-motor seizure | 10083376 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| GM2 gangliosidosis | 10083933 |
| Grey matter heterotopia | 10082084 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Jeavons syndrome | 10084303 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |

| PT | PT Code |
|---------------------------------------------------|----------|
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Neonatal epileptic seizure | 10082068 |
| Neonatal seizure | 10082067 |
| Partial seizures | 10061334 |
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Transient epileptic amnesia | 10081728 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |
| Hemiconvulsion-hemiplegia-epilepsy syndrome | 10085010 |
| Juvenile absence epilepsy | 10085031 |
| Parietal lobe epilepsy | 10085326 |
| Epilepsy of infancy with migrating focal seizures | 10086114 |
| Photosensitive seizure | 10086294 |
| PURA syndrome | 10085882 |
| Epilepsia partialis continua | 10015034 |

#### PTs (Selective)

| PT | PT Code |
|----------------------------------|----------|
| Confusional state | 10010305 |
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

#### 16.11.14. Weight Gain

### **HLT General nutritional disorders NEC (Selective)**

| PT | PT Code |
|----------------------|----------|
| Abdominal fat apron | 10077983 |
| Overweight | 10033307 |
| Abnormal weight gain | 10000188 |
| Central obesity | 10065941 |
| Obesity | 10029883 |

### PTs (Select) - Physical examination procedures and organ system status

| PT | PT Code |
|-------------------------------|----------|
| Weight abnormal | 10056814 |
| Weight increased | 10047899 |
| Waist circumference increased | 10064863 |
| Body mass index abnormal | 10074506 |
| Body mass index increased | 10005897 |

#### PTs (Select) - General Signs and Symptoms

| PT | PT Code |
|----------------------|----------|
| Fat tissue increased | 10016251 |
| Sarcopenic obesity | 10083992 |

### 16.11.15. Rhabdomyolysis

# Rhabdomyolysis/myopathy (SMQ)

| PT | PT Code |
|---------------------------|----------|
| Muscle necrosis | 10028320 |
| Myoglobin blood increased | 10028625 |
| Myoglobin blood present | 10059888 |
| Myoglobin urine present | 10028631 |
| Myoglobinaemia | 10058735 |
| Myoglobinuria | 10028629 |
| Myopathy | 10028641 |
| Myopathy toxic | 10028648 |
| Necrotising myositis | 10074769 |
| Rhabdomyolysis | 10039020 |
| Thyrotoxic myopathy | 10081524 |
| Muscle infarction | 10086278 |

## PTs (Selective) - Muscle Disorders

| PT | PT Code |
|----------|----------|
| Myalgia | 10028411 |
| Myositis | 10028653 |

#### 16.11.16. Pancreatitis

## Acute pancreatitis (SMQ)

| РТ | PT Code |
|------------------------------------|----------|
| Cullen's sign | 10059029 |
| Grey Turner's sign | 10075426 |
| Haemorrhagic necrotic pancreatitis | 10076058 |
| Immune-mediated pancreatitis | 10083072 |
| Ischaemic pancreatitis | 10066127 |
| Oedematous pancreatitis | 10052400 |
| Pancreatic abscess | 10048984 |
| Pancreatic cyst drainage | 10082531 |
| Pancreatic haemorrhage | 10033625 |
| Pancreatic phlegmon | 10056975 |
| Pancreatic pseudoaneurysm | 10081762 |
| Pancreatic pseudocyst | 10033635 |
| Pancreatic pseudocyst drainage | 10033636 |
| Pancreatic pseudocyst haemorrhage | 10083813 |
| Pancreatic pseudocyst rupture | 10083811 |
| Pancreatitis | 10033645 |
| Pancreatitis acute | 10033647 |
| Pancreatitis haemorrhagic | 10033650 |
| Pancreatitis necrotising | 10033654 |
| Pancreatitis relapsing | 10033657 |
| Pancreatorenal syndrome | 10056277 |
| Subacute pancreatitis | 10084554 |
| Walled-off pancreatic necrosis | 10085347 |

### 16.11.17. Impact on Creatinine

## Acute renal failure (SMQ)

| PT | PT Code |
|-------------------------------|----------|
| Acute kidney injury | 10069339 |
| Acute phosphate nephropathy | 10069688 |
| Anuria | 10002847 |
| Azotaemia | 10003885 |
| Continuous haemodiafiltration | 10066338 |
| Dialysis | 10061105 |
| Foetal renal impairment | 10078987 |
| Haemodialysis | 10018875 |

| PT | PT Code |
|---------------------------|----------|
| Haemofiltration | 10053090 |
| Neonatal anuria | 10049778 |
| Nephropathy toxic | 10029155 |
| Oliguria | 10030302 |
| Peritoneal dialysis | 10034660 |
| Prerenal failure | 10072370 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Subacute kidney injury | 10081980 |

# Renal Failure and Impairment

| PT | PT Code |
|--------------------------------------|----------|
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |

| PT | PT Code |
|--------------------------|----------|
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |

## 16.11.18. Safety in Pregnancy

Use AE terms co-reported in pregnancy exposures to CAB and/or RPV.

#### 16.12. Appendix 12: Identification of COVID-19 Adverse Events

COVID-19 adverse events are identified based on MedDRA coded values and/or AE referenced in the COVID-19 Coronavirus Infection assessment. PT terms and codes below are from MedDRA 24.1. In case there is a change to the version of MedDRA at time of reporting, the coded values based on the MedDRA version at the time of reporting will be used. Additional events may be added based on the blinded review of AE data collected on study prior to the database freeze.

| PT | PT Code |
|-----------------------------------------------|----------|
| Asymptomatic COVID-19 | 10084459 |
| COVID-19 | 10084268 |
| COVID-19 pneumonia | 10084380 |
| Suspected COVID-19 | 10084451 |
| SARS-CoV-2 carrier | 10084461 |
| SARS-CoV-2 test positive | 10084271 |
| Multisystem inflammatory syndrome | 10086091 |
| Multisystem inflammatory syndrome in adults | 10085850 |
| Multisystem inflammatory syndrome in children | 10084767 |
| SARS-CoV-2 viraemia | 10084640 |
| Post-acute COVID-19 syndrome | 10085503 |
| Coronavirus infection | 10051905 |
| Coronavirus test positive | 10070255 |
| Coronavirus pneumonia | 10084381 |

#### 16.13. Appendix 13: Data Handling for Pregnant Subjects

The SOLAR study allows pregnant subjects on the Q2M arm to continue CAB LA + RPV LA treatment, while those who became pregnant on the BIK arm will be withdrawn. To minimize bias, for summary tables, if Q2M subjects continue while being pregnant, data after date of confirmed pregnancy (as recorded in the eCRF EOS pregnancy form) will not be evaluable for pregnant Q2M subjects with documented evidence confirming pregnancy unless the confirmation occurs prior to or on the same day as termination of pregnancy (as recorded on the EOS pregnancy form and the AE form, respectively) within the same time period between two study visits. The above data handling strategy will not be implemented on the following:

- All adverse events
- ECG/QTc analysis
- Vital signs
- eC-SSRS
- CCI
- Health Outcomes
- Virology

Note all observed data collected for all pregnant subjects will be included in the listings.

For study outcomes based on the FDA snapshot algorithm, an additional sub-category will be added under "No Virologic Data": Not evaluated or discontinued due to confirmed pregnancy. Viral load after confirmed pregnancy of a Q2M subject will not be evaluated for snapshot outcomes (See Appendix 9: Snapshot Algorithm Details).

Sensitivity analysis including all data (all data as observed) will be provided for the following snapshot-based analysis is applicable:

- Summary of Study Outcomes (50 c/mL threshold)
- Summary of Analysis for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL (or <50 c/ml)</li>
- Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL (or <50 c/ml) by Visit

If no Q2M subject became pregnant on study, then the "while on-treatment" strategy will not be necessary and therefore no sensitivity analysis will be performed, and the additional sub-category mentioned above will not be needed.

# 16.14. Appendix 14: Abbreviations & Trade Marks

### 16.14.1. Abbreviations

| Abbreviation | Description |
|--------------|---------------------------------------------------------------|
| 3TC | Lamivudine, EPIVIR |
| ABC | Abacavir, ZIAGEN |
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| AIC | Akaike's Information Criteria |
| AIDS | Acquired immunodeficiency syndrome |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| A&R | Analysis and Reporting |
| BIK | Bictegravir/emtricitabine/tenofovir alafenamide Single Tablet |
| | Regimen |
| BMI | Body Mass Index |
| BP | Blood Pressure |
| CAB | Cabotegravir |
| CAB LA | Cabotegravir long-acting |
| CD4 | Cluster of Differentiation 4 |
| CD8 | Cluster of Differentiation 8 |
| CDC | Centers for Disease Control and Prevention |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CKD-EPI | Chronic Kidney Disease Epidemiology Collaboration |
| CMH | Cochran-Mantel Haenszel |
| COVID-19 | Coronavirus Disease 2019 |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CS | Clinical Statistics |
| CSR | Clinical Study Report |
| C-SSRS | Columbia Suicide Severity Rating Scale |
| CTR | Clinical Trial Register |
| CVF | Confirmed Virologic Failure |
| mCVF | Modified Confirmed Virologic Failure |
| c/mL | Copies/milliliter |
| D2I | Direct to Inject |
| DAIDS | Division of Acquired Immunodeficiency Syndrome |
| DBF | Database Freeze |
| DBR | Database Release |
| DNA | Deoxyribonucleic acid |
| DOB | Date of Birth |
| DP | Decimal Places |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Record Form |

| Abbreviation | Description |
|--------------|------------------------------------------------------------|
| eGFR | Estimated Glomerular Filtration Rate |
| EMA | European Medicines Agency |
| ERDF | Efficacy Related Discontinuation Failure |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure |
| | Requirements |
| GSK | GSK |
| HAART | Highly active antiretroviral therapy |
| HBV | Hepatitis B virus |
| HbA1c | Glycated hemoglobin |
| HbsAg | Hepatitis B surface Antigen |
| HCV | Hepatitis C virus |
| HDL | High density lipoprotein |
| HIV | Human Immunodeficiency Virus |
| HIVTSQc | Change Version of HIV Treatment Satisfaction Questionnaire |
| IDMC | Independent Data Monitoring Committee |
| IDSL | Integrated Data Standards Library (GSK Standards Library) |
| IM | Intramuscular |
| IMMS | International Modules Management System |
| INI | Integrase Inhibitor |
| INR | International normalized ratio |
| INSTI | Integrase strand transfer inhibitor |
| IP | Investigational Product |
| ISR | Injection Site Reaction |
| ITT | Intent-To-Treat |
| ITT-E | Intent-To-Treat Exposed |
| mITT-E | Modified Intent-To-Treat Exposed |
| LA | Long Acting |
| LDL | Low density lipoprotein |
| LPV | Lopinavir |
| LPV/r | Lopinavir-ritonavir |
| LTFU | Long-Term Follow-Up |
| MMRM | Mixed Model Repeated Measures |
| NNRTI | Non-nucleoside Reverse Transcriptase Inhibitor |
| NRTI | Nucleoside Reverse Transcriptase Inhibitor |
| OLI | Oral Lead In |
| PBMC | Peripheral Blood Mononuclear Cell |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PI | Protease Inhibitor |
| PIN | Perception of Injection |
| PK | Pharmacokinetic |

| Abbreviation | Description |
|--------------|--------------------------------------------------|
| PopPK | Population PK |
| PP | Per Protocol |
| PRO | Protease |
| PTT | Partial Thromboplastin Time |
| PSRAE | Possible suicidality-related adverse event |
| Q2M | Every 2 Months |
| QC | Quality Control |
| QTcF | Frederica's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| RAL | Raltegravir |
| RAMOS | Randomization & Medication Ordering System |
| RAP | Reporting & Analysis Plan |
| RBP | Retinol Binding Protein |
| RNA | Ribonucleic acid |
| RPR | Rapid plasma reagin |
| RPV | Rilpivirine, Edurant |
| RPV LA | Rilpivirine long-acting |
| RT | Reverse transcriptase |
| RTV | Ritonavir |
| SAE | Serious Adverse Event |
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SMQ | Standardised MedDRA Query |
| SOC | System Organ Class or Standard of Care |
| SOP | Standard Operation Procedure |
| SRM | Study Reference Manual |
| TDF | Tenofovir disoproxil fumarate |
| TFL | Tables, Figures & Listings |
| TRDF | Treatment Related Discontinuation Failure |
| ULN | Upper limit of normal |

#### 16.14.2. Trademarks

| Trademarks of the GSK Group of Companies |
|------------------------------------------|
| EPIVIR |
| EPZICOM/KIVEXA |
| TRIUMEQ |
| TRIZIVIR |
| ZIAGEN |

| Trademarks not owned by the GSK<br>Group of Companies |
|-------------------------------------------------------|
| Biktarvy |
| Edurant |
| GenoSure |
| Monogram Biosciences |
| PhenoSense |
| SAS |

#### 16.15. Appendix 15: List of Data Displays

#### 16.15.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|-------------|-------------|
| Study Population | 1.1 to 1.n | 1.1 to 1.n |
| Efficacy | 2.1 to 2.n | 2.1 to 2.n |
| Safety | 3.1 to 3.n | 3.1 to 3.n |
| Pharmacokinetic* | 4.1 to 4.n | 4.1 to 4.n |
| Health Outcomes | 6.1 to 6.n | 6.1 to 6.n |
| Virology | 7.01 to 7.n | 7.01 to 7.n |
| Section | Listings | |
| ICH Listings | 1 to x | |
| Other Listings | y to z | |

<sup>\*</sup> For the Month 12 analysis, only listings will be provided for the Pharmacokinetic section. The numbers for Table/Figures are reserved for future reports if applicable.

#### 16.15.2. Mock Example Shell Referencing

Nonstandard specifications will be referenced as indicated and if required example mockup displays will be provided in Appendix 16: Example Mock Shells for Data Displays or in a separate document:

| Section | Description |
|---------|---------------------------------------|
| HL | Headline |
| M6 | Month 6 (OLI and BIK)/Month 5 (D2I) |
| M12 | Month 12 (OLI and BIK)/Month 11 (D2I) |

#### 16.15.3. Deliverables

| Delivery [Priority] [1,3] | Description |
|---|---|
| Month 6 | Interim analysis when all participants have completed their Month 6 (OLI |
| | and BIK)/Month 5 (D2I) visit[2] |
| Month 12 | Primary analysis when all participants have completed their Month 12 (OLI |
| | and BIK)/Month 11 (D2I) visit |
| EOS | Final End of Study analysis |

#### NOTES:

- 1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort
- 2. Will not be shared with any participant and with most investigators. See Section 3.1 for details.
- 3. The Month 6(OLI and BIK)/Month 5(D2I) and the Month 12(OLI and BIK)/Month 11(D2I) analyses may also be referred to as the "Month 6" and "Month 12" analysis, respectively.

## 16.15.4. Study Population Tables

Note analysis population below has been updated to reflect the M12 analysis plan. In the Month 6 analysis, ITT-E was used prior to this amendment.

| Stud | y Population T | <b>Tables</b> | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Subj | ect Dispositio | n | | | |
| 1.1. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failures | | M6, M12 |
| 1.2. | Enrolled | NS1 | Summary of Number of Subjects<br>Enrolled by Country and Site ID | Only include "no treatment" if there is any enrolled but not randomized. Column Header style 2. | M6, M12 |
| 1.3. | mITT-E | Shell POP_T1 | Summary of Subject Accountability:<br>Study and Phase Conclusion Record | See 207966/primary_15/T1.3 Include the sections: "Outcome of Adverse Events Which Led to Study Withdrawal" (Fatal and Non-Fatal); "Type of Adverse Events Which Led to Study Withdrawal" (COVID-19 and Non-COVID-19) | HL, M6,<br>M12, EOS |
| 1.4. | mITT-E | Shell POP_T4 | By Phase Summary of Subject<br>Disposition | 201584/primary_07/T1.14 | M12, EOS |
| 1.5. | mITT-E | HIV_ES1 | Summary of Reasons for Withdrawals by Visit (Maintenance Phase) | 201584/ primary_07/T1.9 | M6, M12 |
| 1.6. | mITT-E | ES1 | Summary of Study Drug<br>Discontinuation | mid207966/primary_15/T1.10. Include the sections for fatal/non-fatal, COVID/Non-COVID | M6, M12,<br>EOS |

| Stud | y Population <sup>-</sup> | <b>Tables</b> | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| Proto | col Deviation | | | | |
| 1.7. | mITT-E | Shell POP_T2 | Summary of Important Protocol Deviations | ICH E3 | M6, M12,<br>EOS |
| 1.8. | mITT-E | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | Header Style 1 | M6, M12 |
| Popu | lation Analys | ed | | | |
| 1.9. | Screened | Shell POP_T3 | Summary of Study Populations | | HL, M6,<br>M12, EOS |
| 1.10. | mITT-E | Shell POP_T2 | Summary of Protocol Deviations<br>Leading to Exclusion from the Per-<br>Protocol Population - (Month X<br>Analysis) | [X =12 or 6] Add footnote: Month 6 Analysis: Month 6 (OLI and BIK)/Month 5 (D2I) or Month 12 Analysis: Month 12 (OLI and BIK)/Month 11 (D2I) | M6, M12 |
| Dem | ographic and | Baseline Characteristics | | | |
| 1.11. | mITT-E | mid207966/primary_15/T1.16 | Summary of Demographic Characteristics | | HL, M6,<br>M12 |
| 1.12. | Screened | mid207966/primary_15/T1.17 | Summary of Age Ranges | Including a column for No treatment | M6, M12 |
| 1.13. | mITT-E | DM6 | Summary of Race and Racial Combinations Details | | M6, M12 |
| 1.14. | mITT-E | mid207966/primary_15/T1.20 | Summary of Hepatitis Status at Entry | | M6, M12 |
| 1.15. | mITT-E | CDC1 | Summary of CDC Stages of HIV Infection at Maintenance Baseline | | M6, M12 |

| Stud | y Population <sup>-</sup> | Tables | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable [Priority] |
| 1.16. | mITT-E | mid207966/primary_15/T1.23 | Distribution of CD4+ Cell Count<br>Results at Screening and<br>Maintenance Baseline | | M6, M12 |
| 1.17. | mITT-E | mid207966/primary_15/T1.25 | Summary of HIV Risk Factors | | M6, M12 |
| Prior | and Concom | itant Medications | | | |
| 1.18. | mITT-E | MH1 | Summary of Current and Past Medical Conditions | Combine the current and past displays, by adding section headers: "Current", "Past" | M6, M12 |
| 1.19. | mITT-E | MH4 | Summary of Current and Past<br>Cardiac, Gastrointestinal, Metabolism<br>and Nutrition, Psychiatric, Renal and<br>Urinary, Nervous System Conditions,<br>and Hepatobiliary Disorders | Combine the two displays, by adding section headers: "Current", "Past" | M6, M12 |
| 1.20. | mITT-E | CA3 | Summary of Prior ART Medications | | M6, M12 |
| 1.21. | mITT-E | CM8 | Summary of Concomitant Non-ART<br>Medication Ingredient Combinations -<br>Maintenance Phase | | M6, M12 |
| 1.22. | mITT-E | mid207966/primary_15/T1.33 | Summary of Lipid Modifying Agent Use at Baseline and During Maintenance Phase | Combine the two displays, by adding a section header: "Maintenance Baseline", "Started During Maintenance Phase" | M6, M12 |
| 1.23. | mITT-E | mid207966/primary_15/T1.35 | Summary of Substance and Illicit Drug Use at Entry | | M6, M12 |
| COV | ID-19 Pande | mic Impact | | | |
| 1.24. | mITT-E | PAN4 | Summary of Visits impacted by COVID-19 Pandemic | | M6, M12,<br>EOS |

#### 16.15.5. Efficacy Tables

Note: For subgroup analyses, include randomization strata, all demographic and baseline characteristic subgroups as mentioned in EMA Subgroup Category 2 in Section 5.4.2 if applicable, unless otherwise specified.

Note analysis population below has been updated to reflect the M12 analysis plan. In the Month 6 analysis, ITT-E and CVF were used prior to this amendment.

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prima | ary Efficacy A | nalyses | | | |
| 2.1. | mITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA >=50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis - mITT-E | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | HL, M6, M12 |
| 2.2. | PP | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA >=50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis – Per Protocol | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | HL, M6, M12 |
| 2.3. | ITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA >=50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis – ITT-E (Efficacy<br>Sensitivity) | | M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.4. | mITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA >=50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis - mITT-E (All Data<br>as Observed) | Only required if there is any confirmed pregnancy on the Q2M arm. | M6, M12 |
| 2.5. | mITT-E | Shell EFF_T1 | Summary of Study Outcomes (50 c/mL<br>Threshold) at Month 12 (OLI and<br>BIK)/Month 11 (D2I) - Maintenance<br>Phase - Snapshot Analysis – Overall<br>and by subgroup | For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". Add section header for "Overall" and "Subgroup:xx:xx" | HL (overall<br>only), M6,<br>M12 |
| 2.6. | ITT-E | Shell EFF_T1 | Summary of Study Outcomes (50 c/mL<br>Threshold) at Month 12 (OLI and<br>BIK)/Month 11 (D2I) - Maintenance<br>Phase - Snapshot Analysis – ITT-E<br>(Efficacy Sensitivity) | Overall only | M12 |
| 2.7. | mITT-E | Shell EFF_T1 | Summary of Study Outcomes (50 c/mL<br>Threshold) at Month 12 (OLI and<br>BIK)/Month 11 (D2I) - Maintenance<br>Phase - Snapshot Analysis (All Data<br>as Observed) | Only required if there is any confirmed pregnancy on the Q2M arm. | M6, M12 |
| 2.8. | mITT-E | SNAPSHOT3A | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA >=50 c/mL at Month 12 (OLI and BIK)/Month 11 (D2I) - Maintenance Phase - Snapshot Analysis | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". For code refer to mid207966/primary_15/T2.10 | M12 |

| Effica | acy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.9. | mITT-E | SNAPSHOT5 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA >=50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) by Subgroup - Maintenance<br>Phase - Snapshot Analysis | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". For code refer to mid207966/primary_15/T2.5 | M12 |
| Seco | ndary Efficacy | / Analyses | | | |
| 2.10. | mITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA < 50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis - mITT-E | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | HL, M6, M12 |
| 2.11. | PP | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA < 50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis – Per Protocol | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | HL, M6, M12 |
| 2.12. | ITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA < 50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis – ITT-E (Efficacy<br>Sensitivity) | | M12 |
| 2.13. | mITT-E | Shell EFF_T3 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA <50<br>c/mL at Month 12 (OLI and BIK)/Month<br>11 (D2I) - Maintenance Phase -<br>Snapshot Analysis - mITT-E (All Data<br>as Observed) | Only required if there is any confirmed pregnancy on the Q2M arm. | M6, M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.14. | mITT-E | SNAPSHOT3A | Treatment by Strata Tests of Homogeneity for Proportion of Subjects with Plasma HIV-1 RNA < 50 c/mL at Month 12 (OLI and BIK)/Month 11 (D2I) - Maintenance Phase - Snapshot Analysis | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | M12 |
| 2.15. | mITT-E | SNAPSHOT5 | Summary of Analysis for Proportion of<br>Subjects with Plasma HIV-1 RNA < 50<br>c/mL at Month 12 (OLI and BIK) and<br>Month 11 (D2I) by Subgroup -<br>Maintenance Phase - Snapshot<br>Analysis | Q2M vs BIK. For Month 6/5 deliverable: replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)". | M12 |
| 2.16. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA ≥50 c/mL by Visit<br>(Maintenance Phase) – Snapshot<br>Analysis | For code refer to mid207966/primary_15/T2.13 | M6, M12 |
| 2.17. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA ≥50 c/mL by Visit | Only required if there is any confirmed pregnancy on the Q2M arm. | M6, M12,<br>EOS |
| 2.18. | mITT-E | SNAPSHOT6 | Proportion of Subjects with Plasma<br>HIV-1 RNA >=50 c/mL by Subgroup<br>and Visit (Maintenance Phase) –<br>Snapshot Analysis | For code refer to mid207966/primary_15/T2.14 | M12 |
| 2.19. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA <50 c/mL by Visit<br>(Maintenance Phase) – Snapshot<br>Analysis | | M6, M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.20. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA <50 c/mL by Visit | | M6, M12,<br>EOS |
| 2.21. | mITT-E | SNAPSHOT6 | Proportion of Subjects with Plasma<br>HIV-1 RNA <50 c/mL by Subgroup and<br>Visit (Maintenance Phase) – Snapshot<br>Analysis | | M12 |
| 2.22. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA <200 c/mL by Visit<br>(Maintenance Phase) – Snapshot<br>Analysis | | M6, M12 |
| 2.23. | mITT-E | SNAPSHOT4 | Proportion of Subjects with Plasma<br>HIV-1 RNA >=200 c/mL by Visit<br>(Maintenance Phase) – Snapshot<br>Analysis | | M6, M12 |
| 2.24. | mITT-E | Shell EFF_T1 | Summary of Study Outcomes (200 c/mL Threshold) at Month 12 (OLI and BIK)/Month 11 (D2I) (Maintenance Phase) – Snapshot Analysis | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" No subgroup needed | M6, M12 |
| 2.25. | mITT-E | mid207966/primary_15/2.19 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Month 12 (OLI and BIK) /Month 11 (D2I) - Treatment Related Discontinuation = Failure | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" | M6, M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.26. | mITT-E | mid207966/primary_15/T<br>2.20 | Summary of Kaplan-Meier Estimates of Proportion of Subjects Without Confirmed Virologic Failure at Month 12 (OLI and BIK) /Month 11 (D2I) - Efficacy Related Discontinuation = Failure | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" | M6, M12 |
| 2.27. | mITT-E | mid207966/primary_15/T2.21 | Proportion of Subjects with HIV-1 RNA<br>>=50 c/mL at Month 12 (OLI and<br>BIK)/Month 11 (D2I) (Snapshot) by<br>Last Delay in IP Injection (Maintenance<br>Phase) | | M6, M12 |
| 2.28. | mITT-E | mid207966/primary_15/T2.38 | Summary of Change from<br>Maintenance Baseline (Day 1) in<br>Plasma HIV-1 RNA (log10 c/mL) by<br>Visit | | M6, M12,<br>EOS |
| 2.29. | mITT-E | mid207966/primary_15/T2.23 | Cumulative Proportion of Subjects<br>Meeting Confirmed Virologic Failure<br>Criteria by Visit During | Up to Month 13/14 | HL, M6, M12,<br>EOS |
| 2.30. | mCVF | mid207966/primary_15/T2.25 | By Phase Distribution of Quantitative<br>Plasma HIV-1 RNA Results at<br>Suspected and Confirmation of<br>Confirmed Virologic Failure | | M6, M12,<br>EOS |
| 2.31. | mITT-E | mid207966/primary_15/T2.28 | Summary of Viral Load Category by Visit (Maintenance Phase) | Q2M and BIK only | M12 |

| Effica | Efficacy: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 2.32. | mITT-E | Shell EFF_T2 | Summary of Change from<br>Maintenance Baseline (Day 1) in CD4+<br>Cell Count (cells/mm^3) by Visit -<br>Overall | | M6, M12,<br>EOS |
| 2.33. | mITT-E | Shell EFF_T2 | Summary of Change from<br>Maintenance Baseline (Day 1) in CD8+<br>Cell Count (cells/mm^3) by Visit -<br>Maintenance Phase | Baseline, M5/6, M11/12<br>No subgroup | M6, M12 |
| 2.34. | mITT-E | Shell EFF_T2 | Summary of CD4+/CD8+ Cell Count<br>Ratio by Visit – Maintenance Phase | Baseline, M5/6, M11/12<br>No subgroup | M6, M12 |
| 2.35. | mITT-E | CDC2 | By Phase Summary of Stage-3 HIV-1<br>Associated Conditions | Add section header for "Including Recurrences" and<br>"Excluding Recurrences" | M6, M12.<br>EOS |

## 16.15.6. Efficacy Figures

Note analysis population below has been updated to reflect the M12 analysis plan. In the Month 6 analysis, ITT-E was used prior to this amendment.

| Effica | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Prima | ary Efficacy A | nalyses | | | |
| 1. | mITT-E | mid207966/primary_15/F2.1 | Proportion (95% CI) of Subjects with HIV-1 RNA ≥50 c/mL by Visit (Maintenance Phase) – Snapshot Analysis | | M6, M12 |
| 2. | mlTT-E | mid207966/primary_15/F2.2 | Unadjusted Treatment Difference in<br>Proportion (95% CI) of Subjects with<br>HIV-1 RNA ≥50 c/mL at Month 12 (OLI<br>and BIK)/Month 11 (D2I) by Subgroup –<br>Snapshot Analysis | | M12 |
| Seco | ndary CCI | Efficacy Analyses | 3 | | |
| 3. | mITT-E | mid207966/primary_15/F2.3 | Proportion (95% CI) of Subjects with<br>HIV-1 RNA <50 c/mL by Visit<br>(Maintenance Phase) – Snapshot<br>Analysis | | M6, M12 |
| 4. | mlTT-E | mid207966/primary_15/F2.4 | Unadjusted Treatment Difference in<br>Proportion (95% CI) of Subjects with<br>HIV-1 RNA <50 c/mL at Month 12 (OLI<br>and BIK)/Month 11 (D2I) by Subgroup –<br>Snapshot Analysis | | M12 |
| 5. | CVF | mid207966/primary_15/F2.7 | c/mL) Profiles by Visit for CVF Subjects | | M6, M12,<br>EOS |

| Effica | Efficacy: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6. | ITT-E | mid207966/primary_15/F2.8 | Individual complete Individual complete Individual complete Individual complete Individual Individu | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" | M6, M12 |

#### 16.15.7. Safety Tables

Note: For the Month 6 analysis, remove "By Phase" in the title if applicable and add to the end "(Maintenance Phase)", unless otherwise noted.

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expos | Exposure | | | | |
| 3.1. | Safety | Shell SAF_T2a and<br>SAF_T2b | By Phase Summary of Extent of Exposure to Study Treatment including SOC Oral Bridging | ICH E3 | M6, M12,<br>EOS |
| 3.2. | Safety | Shell SAF_T3 | Summary of Needle Length and Gauge for<br>CAB and RPV Injections (Maintenance<br>Phase) | | M6, M12 |
| 3.3. | Safety | mid207966/primary_15/T3.5 | Summary of Adherence to CAB/RPV Injection Dosing Schedule (Maintenance Phase) | | M6, M12 |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adver | Adverse Events | | | | |
| 3.4. | Safety | Shell SAF_T1a and SAF_T1b | <b>By Phase</b> Summary of All Adverse Events by System Organ Class and Preferred Term | ICH E3 | M6, M12 |
| 3.5. | Safety | Shell SAF_T4a and Shell<br>SAF_T4b | <b>By Phase</b> Summary of All Adverse Events by System Organ Class, Preferred Term and Maximum Toxicity | ICH E3 Include Unknown column if at last 1 AE exists with a missing/unknown toxicity grade mid207966/primary_15/T3.7 | HL, M6, M12,<br>EOS |
| 3.6. | Safety | Shell SAF_T4a and Shell<br>SAF_T4b | <b>By Phase</b> Summary of All Adverse Events Excluding Injection Site Reactions by System Organ Class, Preferred Term and Maximum Grade Toxicity | | HL, M6, M12,<br>EOS |
| 3.7. | Safety | AE3 | By Phase Summary of Common Adverse<br>Events (>=5%) by Overall Frequency | ICH E3<br>mid207966/primary_15/T3.11 | M6, M12,<br>EOS |
| 3.8. | Safety | AE3 | By Phase Summary of Common Grade 2-5<br>Adverse Events (>=1%) by Overall<br>Frequency | ICH E3<br>mid207966/primary_15/T3.12 | M6, M12,<br>EOS |
| 3.9. | Safety | Shell SAF_T1a and<br>SAF_T1b | <b>By Phase</b> Summary of All Drug-Related<br>Adverse Events by System Organ Class<br>and Preferred Term | ICH E3 | M6, M12 |
| 3.10. | Safety | Shell SAF_T4a and Shell<br>SAF_T4b | By Phase Summary of All Drug-Related<br>Adverse Events by System Organ Class,<br>Preferred Term and Maximum Toxicity | ICH E3 | HL, M6, M12,<br>EOS |
| 3.11. | Safety | Shell SAF_T4a and Shell<br>SAF_T4b | By Phase Summary of All Drug-Related<br>Adverse Events Excluding Injection Site<br>Reactions by System Organ Class,<br>Preferred Term and Maximum Toxicity | ICH E3 For Month 6: remove "By Phase" and add "(Maintenance Phase)" to the end | HL, M6, M12,<br>EOS |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | Safety | AE3 | By Phase Summary of All Drug-Related<br>Grade 2-5 Adverse Events by Overall<br>Frequency | mid207966/primary_15/T3.17 | M6, M12,<br>EOS |
| Serio | us and Other | Significant Adverse Events | | | |
| 3.13. | Safety | Shell SAF_T1a and<br>SAF_T1b | By Phase Summary of Serious Adverse<br>Events by System Organ Class and<br>Preferred Term | ICH E3 | HL, M6, M12,<br>EOS |
| 3.14. | Safety | Shell SAF_T1a and SAF_T1b | By Phase Summary of Drug-Related<br>Serious Adverse Events by System Organ<br>Class and Preferred Term | | M6, M12,<br>EOS |
| 3.15. | Safety | AE3 | <b>By Phase</b> Summary of Non-Fatal Serious<br>Adverse Events by Overall Frequency | mid207966/primary_15/T3.23 | M6, M12 |
| 3.16. | Safety | AE3 | <b>By Phase</b> Summary of Drug-Related Non-<br>Fatal Serious Adverse Events by Overall<br>Frequency | mid207966/primary_15/T3.24 | M6, M12,<br>EOS |
| 3.17. | Safety | Shell SAF_T1a and<br>SAF_T1b | By Phase Summary of Adverse Events Leading to Withdrawal/Permanent Discontinuation of Investigational Product by System Organ Class and Preferred Term | | HL, M6, M12,<br>EOS |
| 3.18. | Safety | AE3 | Summary of Common (>=5%) Non-Serious<br>Adverse Events by System Organ Class<br>and Preferred Term (Maintenance Phase) | | M6, M12 |
| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.19. | Safety | AE15 | Summary of Subjects and Number of<br>Occurrences of Common (>=5%) Non-<br>Serious Adverse Events by System Organ<br>Class and Preferred Term (Maintenance<br>Phase) | mid207966/primary_15/T3.28 | M6, M12 |
| 3.20. | Safety | AE16 | By Phase Summary of Subjects and<br>Number of Occurrences of SAEs, Fatal<br>SAEs, and Drug-related SAEs by System<br>Organ Class and Preferred Term | mid207966/primary_15/T3.29 | M6, M12,<br>EOS |
| 3.21. | Safety | Shell SAF_T5 | Summary of Cumulative Adverse Events by Preferred Term and Visit (Maintenance Phase) | mid207966/primary_15/T3.30 | M6, M12 |
| Inject | ion Site React | ion Adverse Events | | | |
| 3.22. | Safety | 207966/primary_15/T3.31 | By Phase Event-level Summary of Injection<br>Site Reaction Adverse Events by Preferred<br>Term | Include Overall ISR as a Preferred Term D2I, OLI and Q2M | HL, M6, M12.<br>EOS |
| 3.23. | Safety | 207966/primary_15/T3.33 | Summary of Overall and Common Subject-<br>level Characteristics of Injection Site<br>Reaction Adverse Events by Preferred<br>Term (Maintenance Phase) | Include Overall ISR as a Preferred Term D2I, OLI and Q2M Common ISR includes pain, induration, nodules and any other ISR with ≥5% subjects among randomized Q2M arm | M6, M12 |
| 3.24. | Safety | 207966/primary_15/T3.36<br>and T3.40 | Event-level Summary of Drug-Related Injection Site Reaction Adverse Events by Investigational Product and Preferred Term (Maintenance Phase) | Include Overall ISR as a Preferred Term D2I, OLI and Q2M Investigational Product: "CAB LA" or "RPV LA", "CAB/RPV LA" | M6, M12 |

| Safety | /: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.25. | Safety | 207966/primary_15/T3.37<br>and T3.41 | Summary of Overall and Common Subject-<br>level Characteristics of Drug-Related<br>Injection Site Reaction Adverse Events by<br>Investigational Product and Preferred<br>Term (Maintenance Phase) | Include Overall ISR as a Preferred Term D2I, OLI and Q2M Investigational Product: "CAB LA" or "RPV LA", "CAB/RPV LA" | M6, M12 |
| 3.26. | Safety | 207966/primary_15/T3.35 | Summary of Overall and Common Injection<br>Site Reaction Adverse Events by Preferred<br>Term, Visit, and Maximum Severity<br>(Maintenance Phase) | Include Overall ISR as a Preferred Term D2I, OLI and Q2M | M6, M12 |
| 3.27. | Safety | 207966/primary_15/T3.38<br>and T3.42 | Summary of Overall and Common Drug-<br>Related Injection Site Reaction Adverse<br>Events by Investigational Product,<br>Preferred Term, Visit and Maximum<br>Severity(Maintenance Phase) | Include Overall ISR as a Preferred Term D2I, OLI and Q2M Investigational Product: "CAB LA" or "RPV LA", "CAB/RPV LA" | M6, M12 |
| 3.28. | Safety | 207966/primary_15/T3.39<br>and T3.43 | Summary of Maximum Drug-Related Injection Site Reaction Adverse Event Grade by Investigational Product, Preferred Term and Needle Length (Maintenance Phase) - Common ISRs | Do not include Overall ISR as a Preferred Term D2I, OLI and Q2M Investigational Product: "CAB LA" or "RPV LA" | M6, M12 |
| Labora | atory: Chemisti | ry and Hematology | | | |
| 3.29. | Safety | Shell SAF_T6 | Summary of Chemistry Changes from Baseline by Visit | ICH E3 | M6, M12,<br>EOS |
| 3.30. | Safety | Shell SAF_T7 | By Phase Summary of Maximum Emergent<br>Chemistry Toxicities | 207966/primary_15/T3.48 | M6, M12,<br>EOS |
| 3.31. | Safety | Shell SAF_T6 | Summary of Hematology Changes from Baseline by Visit | ICH E3 | M6, M12,<br>EOS |

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.32. | Safety | Shell SAF_T7 | By Phase Summary of Maximum Emergent Hematology Toxicities | 207966/primary_15/T3.50 | M6, M12,<br>EOS |
| Labor | atory: Urinaly | rsis | | | |
| 3.33. | Safety | 207966/primary_15/T3.39<br>and T3.52 | Summary of Urinalysis Dipstick Results by Visit (Maintenance Phase) | | M6, M12 |
| 3.34. | Safety | Shell SAF_T6 | Summary of Urine Concentrations<br>Changes from Baseline by Visit<br>(Maintenance Phase) | 207966/primary_15/ T3.53 | M6, M12 |
| 3.35. | Safety | 207966/primary_15/ T3.53 | Summary of Changes in Proteinuria Baseline Laboratory Result to Maximum Post-Baseline Laboratory Result (Maintenance Phase) | | M6, M12 |
| Labor | atory: Lipids | | | | |
| 3.36. | Safety | 207966/primary_15/ T3.55 | Summary of Changes from Maintenance Baseline (Day 1) NCEP Fasting Lipid Category to Maximum Maintenance Phase Category – Triglycerides | | M6, M12 |
| 3.37. | Safety | 207966/primary_15/ T3.56 | Summary of Changes from Maintenance<br>Baseline (Day 1) NCEP Fasting Lipid<br>Category to Maximum Maintenance Phase<br>Category – Total Cholesterol | | M6, M12 |
| 3.38. | Safety | 207966/primary_15/ T3.57 | Summary of Changes from Maintenance<br>Baseline (Day 1) NCEP Fasting Lipid<br>Category to Minimum Maintenance Phase<br>Category – HDL Cholesterol | | M6, M12 |

| Safety | r: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.39. | Safety | 207966/primary_15/ T3.58 | Summary of Changes from Maintenance<br>Baseline (Day 1) NCEP Fasting Lipid<br>Category to Maximum Maintenance Phase<br>Category – LDL Cholesterol | | M6, M12 |
| 3.40. | Safety | 207966/primary_15/ T3.59 | Summary of Fasting Lipids Percentage<br>Changes from Baseline by Visit ( Lipid<br>Evaluable) - Maintenance Phase | | M6, M12 |
| 3.41. | Safety | 207966/primary_15/ T3.60 | Summary of Fasting TC/HDL Ratio<br>Changes from Maintenance Baseline (Day<br>1) (Maintenance Phase) – Lipid Evaluable | | M6, M12 |
| Labor | atory: Hepato | biliary (Liver) | | | |
| 3.42. | Safety | LIVER1 | By Phase Summary of Liver<br>Monitoring/Stopping Event Reporting | GSK Statistical Display Standard<br>207966/primary_15/ T3.61 | M6, M12,<br>EOS |
| 3.43. | Safety | 207966/primary_15/ T3.62 | By Phase Summary of Subjects Meeting<br>Hepatobiliary Abnormality Criteria | GSK Statistical Display Standard<br>Include 2 sections: OLI, Maintenance(See SAF_T7 for<br>section headers) | M6, M12,<br>EOS |
| Bone, | Renal, Inflam | mation, Insulin Resistance | Markers and CCI | | |
| 3.44. | Safety | SAF_T8 | Summary of Changes from Maintenance<br>Baseline (Day 1) - Bone, Renal,<br>Inflammation and Insulin Resistance<br>Markers (Maintenance Phase) | Ass section header: Bone Markers/Renal Markers/ COL // Insulin Resistance Markers HOMA-IR for insulin resistance marker Q2M vs. BIK | M12 |
| 3.45. | Safety | SAF_T11 | Summary of Shift in HOMA-Insulin<br>Resistance Categories from Baseline by<br>Visit (Maintenance Phase) | | M12 |

| Safety | afety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.46. | Safety | SAF_T9 | Statistical Analysis of Log-Transformed<br>Ratio to Baseline in HOMA-Insulin<br>Resistance - MMRM | 201584 primary_16/T6.08 | M12 |
| 3.47. | Safety | SAF_T10 | Statistical Analysis of Proportion of<br>Subjects with HOMA-IR ≥2, >=3 and >=4<br>at M12 (OLI and BIK) /M11(D2I) – Logistic<br>Regression | See Section 8.5.4 for details. Note: Subjects with evidence of pre-study diabetes (via medical history or prior medications) are excluded. | M12 |
| 3.48. | Safety | SAF_T9 | Statistical Analysis of Log-Transformed<br>Ratio to Baseline in Bone Markers - MMRM | 201584 primary_16/T6.08 | M12 |
| 3.49. | Safety | SAF_T9 | Statistical Analysis of Log-Transformed<br>Ratio to Baseline in Renal Markers- MMRM | 201584 primary_16/T6.08 | M12 |
| 3.50. | Safety | SAF_T9 | Statistical Analysis of Log-Transformed Ratio to Baseline in CCI MMRM | 201584 primary_16/T6.08 | M12 |
| 3.51. | Safety | SAF_T8 | Summary of Change from Baseline in by Visit | Include baseline | M12 |
| ECG | | | | | |
| 3.52. | Safety | EG1 | Summary of ECG Findings (Maintenance Phase) | 207966/primary_15/T3.64 | M12 |
| 3.53. | Safety | EG2 | Summary of Change from Baseline in ECG<br>Values by Visit (Maintenance Phase) | | M12 |

| Safety | y: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.54. | Safety | EG10 | Summary of QTc Values by Category (Maintenance Phase) | 207966/primary_15/T3.66 | M12 |
| 3.55. | Safety | EG10 | Summary of Change from Baseline QTc<br>Values by Category (Maintenance Phase) | 207966/primary_15/T3.67 | M12 |
| Vital | Signs and Ant | hropometric Profile | | | |
| 3.56. | Safety | VS1 | By Phase Summary of Change from Baseline in Vital Signs by Visit | Q2M and BIK only | M6, M12,<br>EOS |
| 3.57. | Safety | SAF_T12 | Summary of Shift in BMI Categories from<br>Baseline by Visit ( <b>Overall and By Strata</b> ) –<br>Maintenance Phase | Q2M and BIK only 207966/primary_15/T3.70 Month 5/6 and Month 11/12 For month 6 remove " by visit" Only include Gender, as BMI is already one of the stratification factors (M12) | M6, M12 |
| 3.58. | Safety | SAF_T13 | Summary of Change from Baseline in<br>Weight and BMI by Gender, Baseline BMI,<br>Race and by Visit (Maintenance Phase) | Q2M and BIK only 207966/primary_15/T3.71 Month 5/6 and Month 11/12 For month 6 remove " by visit". Do not need overall | M6, M12 |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.59. | Safety | SAF_T14 | Summary of Percent Change from Baseline in Weight (Maintenance Phase) | Q2M and BIK only | M6. M12 |
| 3.60. | Safety | VS1 | Summary of Anthropometric Parameters by Visit (Lipid Evaluable) | Q2M and BIK only. Include all planned visits Include: weight, height, BMI, waist and hip circumference, cell and Tanita scale measurements (total body Fat %, bone mass, musl mass, TBW%) | М6 |
| 3.61. | Safety | VS1 | Summary of Anthropometric Parameters by<br>Visit Excluding Subjects with Cosmetic<br>procedures (Lipid Evaluable) | Q2M and BIK only add footnote: Cosmetic procedures include procedures of the torso/thighs (exclude face/neck) including but not limited to liposuction/liposculpture/implants. | M12 |
| 3.62. | Safety | VS1 | Summary of Change from Baseline in<br>Anthropometric Parameters by Visit (Lipid<br>Evaluable) | Q2M and BIK only<br>Same parameters as 3.60 | М6 |

| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| 3.63. | Safety | VS1 | Summary of Change from Baseline in<br>Anthropometric Parameters by Visit<br>Excluding Subjects with Cosmetic<br>Procedures (Lipid Evaluable) | Q2M and BIK only add footnote: Cosmetic procedures include procedures of the torso/thighs (exclude face/neck) including but not limited to liposuction/liposculpture/implants. | M12 |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Metab | oolic Syndrom | ie | | | |
| 3.64. | Safety | SAF_T15 | Summary of Percent of Subjects with<br>Metabolic Syndrome and Risk Factors<br>(Maintenance Phase) | Q2M and BIK only In addition to Metabolic syndrome, also include percentage for each of the 5 factors: Elevated waist circumference; Elevated triglycerides; Reduced HDL-C; Elevated blood pressure; Elevated fasting glucose | M6, M12 |
| 3.65. | Safety | SAF_T12 | Summary of Shift in Metabolic Syndrome and Risk Factors at M12 (OLI and BIK) /M11(D2I) from Baseline | Update to M5/6 for M6 RE. Q2M and BIK only. Shift table from baseline to M5/6 or M11/12, Yes/No/Missing | M6, M12 |
| 3.66. | Safety | SAF_T10 | Statistical Analysis of Proportion of<br>Subjects with Metabolic Syndrome at M12<br>(OLI and BIK) /M11(D2I) – Logistic<br>Regression | | M6, M12 |

| Safety | afety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Cardio | ardiovascular Risk and Substance Use | | | | |
| 3.67. | Safety | 207966/primary_15/T1.22 | Summary of Cardiovascular Risk<br>Assessments by Visit (Maintenance Phase) | Add section header for each visit. For month 6, only calculate Framingham equation For month 12, also include smoking status Q2M vs. BIK | M6, M12 |
| 3.68. | Safety | SAF_T17 | Summary of Substance and Illicit Drug Use (Maintenance Phase) | Q2M vs. BIK | M12 |
| eC-SS | C-SSRS | | | | |
| 3.69. | Safety | CSSRS1 | By Phase Summary of Subjects with eC-<br>SSRS Suicidal Ideation or Behaviour | 207966/primary_15/T3.72<br>Q2M and BIK | M6, M12 |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| AEs o | AEs of Special Interest (AESI) | | | | |
| 3.70. | Safety | 207966/primary_15/T3.73 | By Phase Summary of Depression, Anxiety and Suicidal Ideation/Behaviour Adverse Events by System Organ Class, Preferred Term, Maximum DAIDS Toxicity Grade, and Prior History (Depression, Anxiety or Suicidal Ideation) at Screening | 3 Layers of section headers: Phase: Oral Lead-In Period(Maintenance)/Maintenance Treatment: Q2M, OLI(Q2M), D2I(Q2M), BIK Subjects has: yes/no prior history of depression, yes/or prior history of anxiety, yes/or prior history of suicidal ideation | M6, M12,<br>EOS |
| | | | | For Oral Lead-In period, only need to present the OLI(Q2M) groups | |
| 3.71. | Safety | SAF_T16a and<br>SAF_T16b | By Phase Summary of Adverse Events of<br>Special Interest by AESI Category,<br>System Organ Class and Preferred Term<br>(Number of Subjects and Occurrence) | 207966/primary_15/T3.75 | M6, M12,<br>EOS |
| 3.72. | Safety | 207966/primary_15/T3.109 | By Phase Summary of Characteristics of Adverse Events of Special Interest | Add footnote: AESIs with at least 1 event are included in the summary. | M6, M12,<br>EOS |
| 3.73. | Safety | 207966/primary_15/T3.111<br>and T3.112 | By Phase Summary of Syncope and Presyncope Adverse Events | | M6, M12,<br>EOS |
| COVII | D-19 Assessm | nents | | | |
| 3.74. | Safety | 207966 primary 15/Table<br>3.113 | Summary of COVID-19 Adverse Events by<br>System Organ Class, Preferred Term and<br>Maximum Toxicity (Maintenance Phase) | Q2M and BIK only | M6, M12 |

| Safety | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard/ Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.75. | Safety | PAN1 / PAN1A | Summary of COVID-19 Assessments for Subjects with COVID-19 Adverse Events | Q2M and BIK only | M6, M12 |
| 3.76. | Safety | PAN3 / PAN3A | Summary of COVID-19 Symptoms for Subjects with COVID-19 Adverse Events | Q2M and BIK only | M6, M12 |
| Additio | onal Analysis | | | | |
| 3.77. | Safety | Shell SAF_T6 | Summary of Absolute and Change from<br>Baseline Values by Visit (Maintenance<br>Phase) – Creatinine and GFR (Excluding<br>Samples Impacted by Possible Faulty<br>Reagents) | Q2M and BIK only. Note: Samples impacted by possible faulty reagents are those collected from Australia, Japan, USA and Canada between 21Dec 212020 and 30Mar2021, and those collected from all other European countries between 02Jan2021 to 28Feb2021. | M12 |
| 3.78. | Safety | Shell SAF_T7 | Summary of Maximum Maintenance Phase<br>Emergent Chemistry Toxicities – Creatinine<br>and GFR (Excluding Samples Impacted by<br>Possible Faulty Reagents) | Q2M and BIK only. Note: Samples impacted by possible faulty reagents are those collected from Australia, Japan, USA and Canada between 21Dec2020 and 30Mar2021, and those collected from all other European countries between 02Jan2021 to 28Feb2021. | M12 |
| 3.81. | Safety | Shell SAF_T6 | Summary of Change from Baseline in Weight and BMI by Visit | | M12, EOS |

## 16.15.8. Safety Figures

| Safety: Fi | gures | | | | |
|---|---|---|---|---|---|
| No. | Popul ation | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Adverse I | Events | | | | |
| 3.1. | Safety | AE10 | Plot of Common Maintenance Phase Adverse Events and Relative Risk(Excluding ISRs) – Q2M vs. BIK | 207966/primary_15/F3.1 | M6, M12 |
| 3.2. | Safety | mid201584/primary_07/T3.<br>14 | Plot of Incidence of Maintenance Phase Drug-Related Injection Site Reaction Adverse Events by Visit (Overall and Common) | Q2M only. 3 Sections: CAB and or RPV CAB RPV | M6, M12 |
| 3.3. | Safety | 201584/primary_07/F3.17 | Plot of Incidence of Grade 3-5 Maintenance Phase Drug-<br>Related Injection Site Reaction Adverse Events by Visit<br>(Overall and Common) | Q2M only. 3 Sections: CAB and or RPV CAB RPV | M6, M12 |
| Laborator | ry | | | | |
| 3.4. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT and BILT – Maintenance Phase | GSK Statistical Display Standard Q2M and BIK | M6, M12 |
| 3.5. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin–Maintenance Phase | GSK Statistical Display Standard Q2M and BIK. Remove the reference lines where ULN = 1X (only keep the 2X for BILT and 3X for ALT). | M6, M12 |

| Safety: Fig | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Popul<br>ation | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.6. | Safety | mid207966/primary_15/F3.<br>18 | Bar Chart of Fasting Lipid NCEP Categories | Baseline, M5/6 and M11/12. Include all 4 parameters: Triglycerides, Total Cholesterol, LDL, HDL | M6, M12 |
| 3.7. | Safety | mid215307/iss_01/F3.5 | Bar Chart of Total Cholesterol/HDL Ratio Categories | Q2M and BIK . Baseline, M5/6 and M11/12. Keep big N as denominator | M6, M12 |
| 3.8. | Safety | mid215307/iss_01/F3.6 | Bar Chart of Fasting Blood Glucose | Q2M and BIK . Baseline, M5/6 and M11/12 Keep big N as denominator | M6, M12 |
| 3.9. | Safety | 207966/primary_15/F3.21 | Plot of Incidence of Maintenance Phase Drug-Related Injection Site Reaction Adverse Events by Strata and Visit (Overall and Common) - CAB and/or RPV | Q2M only. Color-code Severity grade within each bar | M6, M12 |
| 3.10. | Safety | SAF_F1 | Line Plot of Mean Change from Baseline by Visit for Bone, Renal, Inflammation and Insulin Resistance Markers | | M12 |
| 3.11. | Safety | SAF_F2 | Patient Profile Plot of Clinical Diagnosis Factors for Patients with Metabolic Syndrome at Any Time Point (Treatment Q2M (OLI)) | Five parameters for each patient, see Section 16.6.4 waist circumference, triglycerides, HDL, BP, fasting glucose. Note for M12 analysis, due to space limit, only those with metabolic syndrome at M11/12 will be plotted. Full plot including all subjects will be produced post hoc. | M6, M12 |

| Safety: Fi | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Popul<br>ation | GSK Standard / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 3.12. | Safety | SAF_F2 | Patient Profile Plot of Clinical Diagnosis Factors for Patients with Metabolic Syndrome at Any Time Point (Treatment Q2M (D2I)) | Same as 3.11 | M6, M12 |
| 3.13. | Safety | SAF_F2 | Patient Profile Plot of Clinical Diagnosis Factors for Patients with Metabolic Syndrome at Any Time Point (Treatment BIK) | Same as 3.11 | M6, M12 |

### 16.15.9. Health Outcome Tables

Note analysis population below has been updated to reflect the M12 analysis plan. In the Month 6 analysis, ITT-E as used instead of mITT-E prior to this amendment.

| Healt | h Outcome: T | ables | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Perce | eption of INjec | tion Questionnaire (PIN) | | | |
| 6.1. | mITT-E | 201584/primary_07/T6.1 | Proportion of Subjects with each individual Questionnaire item score in PIN by Visit (Maintenance Phase) | No BIK | M12 |
| 6.2. | mITT-E | 201584/primary_07/T6.3 | Summary and Statistical Analysis of PIN in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | No BIK Wilcoxon Signed -rank test for analysis (acceptance score only) | M12 |
| 6.3. | mITT-E | 201584/primary_07/T6.4 | Summary of PIN Change from Month 2(OLI)/Month 1(D2I) in Domain Scores (Bother of ISRs, Leg movement, Sleep, and Acceptance) and Individual Items Scores (Anxiety before, Pain, Satisfaction, Anxiety After, Willingness) by Visit (Maintenance Phase) | No BIK | M12 |
| Treat | ment Satisfac | tion (HIVTSQs) | | | |
| 6.4. | mITT-E | 201584/primary_07/T6.18 | Proportion of Subjects with HIVTSQs – Treatment Satisfaction Individual Item Scores (Maintenance Phase) | | M6, M12 |
| 6.5. | mITT-E | 201584/primary_07/T6.18 | Proportion of Subjects with HIVTSQs – Change from baseline in Treatment Satisfaction Individual Item Scores (Maintenance Phase) | Include all possible categories for CFB | M6, M12 |

| Hoalt | h Outcome: T | abito | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 6.6. | mITT-E | 201584/primary_07/T6.21 | Summary of HIVTSQs - Absolute and Change from baseline in Treatment Satisfaction Score by Visit (Maintenance Phase) - Total and Individual | Observed, use section headers<br>"Absolute Value", "Change from<br>Baseline" | M6, M12 |
| 6.7. | mITT-E | HO_T1 | Statistical Analysis of HIVTSQs - Change from Maintenance<br>Baseline (Day 1) in Total Treatment Satisfaction Score and<br>individual items 5 (convenient), 6 (flexible) and 10 (continue)<br>(Maintenance Phase) | ANCOVA for M6, MMRM for M12<br>201584/primary_07/T6.24<br>201584/primary_16/T6.08 | M6, M12 |
| 6.8. | mITT-E | HO_T4 | Statistical Analysis of HIVTSQs - Change from Maintenance<br>Baseline (Day 1) in Total Treatment Satisfaction Score and<br>individual items 5 (convenient), 6 (flexible) and 10 (continue)<br>by Baseline Score Group (Maintenance Phase) | MMRM. See mock shell for details.<br>201584/primary_16/T6.09 | M12 |
| Treat | ment Satisfac | tion (HIVTSQc) | | | |
| 6.9. | mITT-E | 201584/primary_01/T6.25 | Proportion of Subjects with HIV-Treatment Satisfaction<br>Questionnaire Individual Item Score change (HIVTSQc) at<br>Month 12(OLI and BIK)/Month 11(D2I) (Maintenance Phase) | | M12 |
| 6.10. | mITT-E | 201584/primary_01/T6.26 | Summary of HIV-Treatment Satisfaction Questionnaire in<br>Treatment Satisfaction Score Change (HIVTSQc) at Month<br>12(OLI and BIK)/Month 11(D2I) (Maintenance Phase) - Total<br>and Individual | | M12 |
| 6.11. | mITT-E | 201584/primary_01/T6.27 | Statistical Analysis of HIV-Treatment Satisfaction Questionnaire in Treatment Satisfaction Score Change (HIVTSQc) at Month 12 (OLI and BIK)/Month 11(D2I) (Maintenance Phase) | | M12 |

#### CONFIDENTIAL

| Healt | Health Outcome: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| CCI | | | | | |

| No. | Population | GSK Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Treatr | nent Preferen | ice for Q2M vs. BIK | | | |
| 6.14. | mITT-E | HO_T2 | Summary of Treatment Preference and Reason for<br>Preference | | M12 |
| CI | | | | | |

### 16.15.10. Virology Tables

Q2M vs. BIK only for virology tables in this section. Note no summary tables will be produced if less than 5 CVFs in total are observed (excluding subjects from site PPD ). All planned listings will be produced regardless.

Note analysis population below has been updated to reflect the M12 analysis plan. No tables were produced at the M6 analysis (total number of CVFs <5).

| Virolo | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard<br>/ Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Geno | typic | | | | |
| 7.1. | mCVF | 207966/primary_15/T7.1 | Summary of the Prevalence of Known INI Resistance Mutations at time of CVF (Maintenance Phase) – Plasma Sample | | M6, M12 |
| 7.2. | mCVF | 207966/primary_15/T7.2 | Summary of the Prevalence of Major<br>Resistance Mutations of NRTI, NNRTI<br>and PI Class at time of CVF<br>(Maintenance Phase) - Plasma Sample | | M6, M12 |
| 7.3. | mCVF | 207966/primary_15/T7.3 | Summary of Genotypic Susceptibility at time of CVF (Maintenance Phase) - Plasma Sample | | M6, M12 |
| Pheno | otypic | | | | |
| 7.4. | mCVF | 207966/primary_15/T7.4 | Summary of Phenotype Susceptibility at<br>Time of CVF (Maintenance Phase) -<br>Plasma Sample | | M6, M12 |

| Virolo | Virology: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 7.5. | mCVF | 207966/primary_15/T7.5 | Summary of Phenotype: Number of<br>Drugs to Which Subject is Phenotypic<br>Resistant, Partially Sensitive or<br>Sensitive at Time of CVF (Maintenance<br>Phase) - Plasma Sample | | M6, M12 |
| 7.6. | mCVF | 207966/primary_15/T7.6 | Summary of Fold Change to CAB, RPV and BIC at Time of CVF (Maintenance Phase) - Plasma Sample | | M6, M12 |
| Other | , | | | | |
| 7.7. | mCVF | 207966/primary_15/T7.7 | Summary of Net Assessment at Time of CVF (Maintenance Phase) - Plasma Sample | | M6, M12 |

## 16.15.11. ICH Listings

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Stud | y Population | | | | |
| 1. | Randomized | mid207966/primary_15/Listing 1 | Listing of Subjects Randomized but Not Treated | ICH E3 | M6, M12 |
| 2. | ITT-E | Shell POP_L1 | Listing of Reasons for Study Withdrawal | ICH E3 Start from mid201584/primary_40 listing 40. Also see mock up. | HL, M6,<br>M12, EOS |
| 3. | ITT-E | ES2 | Listing of Reasons for Study Drug Discontinuation | ICH E3 | M6, M12,<br>EOS |
| 4. | ITT-E | DV2 | Listing of Important Protocol Deviations | ICH E3 mid201584/primary_07 listing 6. Note: add if related to COVID-19 Column | M6, M12,<br>EOS |
| 5. | ITT-E | DV2 | Listing of Protocol Deviations Leading to Exclusion from the Per-Protocol Population | | HL, M6,<br>M12 |
| 6. | ITT-E | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | ICH E3 | M6, M12,<br>EOS |
| 7. | ITT-E | DM2 | Listing of Demographic Characteristics including Race | ICH E3<br>mid201584/primary_07 listing 9<br>and 10 | M6, M12,<br>EOS |

| ICH: | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Effic | асу | | | | |
| 8. | ITT-E | 207966/primary_15/Listing 11 | Listing of Study Outcome (50 c/mL Threshold) at Month 12(OLI and BIK)/Month 11(D2I) – Snapshot Analysis | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" | HL, M6,<br>M12 |
| 9. | ITT-E | 207966/primary_15/Listing 11 | Listing of Study Outcome (50 c/mL Threshold) at Month 12(OLI and BIK)/Month 11(D2I) – Snapshot Analysis (All Data as Observed) | For Month 6/5 deliverable, replace "Month 12 (OLI and BIK) and Month 11 (D2I)" with "Month 6 (OLI and BIK) and Month 5 (D2I)" | M6, M12 |
| 10. | Randomized | Shell EFF_L1 | Listing of All Plasma HIV-1 RNA Data | | M6, M12,<br>EOS |
| Safe | ty: Exposure | | | | |
| 11. | Safety | 207966 primary_02, L14 / EX3 | Listing of Investigational Product Exposure Data | ICH E3 | M6, M12 |
| Safe | ty: Adverse Ev | ents | | | |
| 12. | Randomized | AE8 | Listing of All Adverse Events | ICH E3 | M6,M12,<br>EOS |
| 13. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse<br>Events | ICH E3 | M6,M12 |
| Safe | ty: Serious and | d Other Significant Adverse Event | ts | | |
| 14. | Safety | AE8 | Listing of Fatal Serious Adverse Events | ICH E3 | M6,M12 |

| ICH: | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard / Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 15. | Safety | AE8 | Listing of Non-Fatal Serious Adverse Events | ICH E3 | M6,M12 |
| 16. | Safety | AE14 | Listing of Reasons for Considering as a Serious<br>Adverse Event | ICH E3 | M6,M12,<br>EOS |
| 17. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study/Permanent Discontinuation of Study Treatment | ICH E3 | HL,<br>M6,M12,<br>EOS |
| 18. | Safety | PSRAE1 | Listing of Possible Suicidality-Related Adverse Event Data: Event and Description (Section 1-Section 2) | | M6, M12 |
| 19. | Safety | PSRAE3 | Listing of Possible Suicidality-Related Adverse Event Data: Possible Cause(s) (Section 3) | | M6, M12 |
| 20. | Safety | PSRAE4 | Listing of Possible Suicidality-Related Adverse Event Data (Section 4) | | M6, M12 |
| 21. | Safety | PSRAE5 | Listing of Possible Suicidality-Related Adverse Event Data (Section 5-Section 8) | | M6, M12 |

## 16.15.12. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study | Population | | | | |
| 22. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | M6, M12,<br>EOS |
| 23. | Randomized | TA1 | Listing of Randomized and Actual Strata and Treatment Assignment | GSK Statistical Display Standard Add "Choice of OLI/D2I" | M6, M12,<br>EOS |
| 24. | ITT-E | CA3 | Listing of Prior ART Medications | | M6, M12 |
| 25. | ITT-E | mid207966/primary_15/listing37 | Listing of Concomitant ART Medications during the Maintenance Phase | | M6, M12,<br>EOS |
| 26. | ITT-E | CA3 | Listing of ART Medications Received during LTFU Phase | | M6, M12 |
| 27. | ITT-E | mid207966/primary_15/listing39 | Listing of Investigational Product Accountability - Oral Regimens | | M6, M12 |
| 28. | ITT-E | mid207966/primary_15/listing40 | Listing of Medical History of Seizure | | M6, M12 |
| 29. | ITT-E | PAN 7 | Listing of All Subjects with Visits and Assessments Impacted by COVID-19 Pandemic | | M6, M12 |
| Effica | су | | | | |
| 30. | ITT-E | 201584/primary_07/L54 | Listing of Stage-3 HIV-1 Associated Conditions | | M6, M12 |
| 31. | CVF | Shell EFF_L1 | Listing of All Plasma HIV-1 RNA Data for Subjects with Confirmed Virologic Failure | | HL, M6, M12 |
| 32. | ITT-E | Shell EFF_L1 | Listing of HIV-1 RNA Data for Subjects Who Became Pregnant During the Study | Add: date of confirmed pregnancy. Only required if any subject becomes pregnant on Q2M. | M6, M12 |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | : Exposure | | | | |
| 33. | Safety | 201584/primary_07/L72 | Listing of Investigational Product Exposure Data during Oral Bridging | | M6, M12 |
| 34. | Safety | 201584/primary_07/L73 | Listing of Dosing Errors and IP Device Malfunctions | | M6, M12 |
| Safety | : Adverse Ever | nts | | | |
| 35. | [Insert] | AE2 | Listing of Relationship Between Adverse Event<br>System Organ Classes, Preferred Terms, and<br>Verbatim Text | GSK Statistical Display Standard | M6, M12 |
| 36. | Safety | AE8 | Listing of Changes in Intensity/Grades of Injection Site Adverse Events | 2011584/primary_07/Listing 22 | M6, M12 |
| 37. | Safety | PAN12 | Listing of COVID-19 Assessments and Symptom<br>Assessments for Subjects with COVID-19 Adverse<br>Events | | M6, M12 |
| 38. | Safety | AE8 | Listing of Grade 3 to 5 Adverse Events | | M6, M12 |
| Safety | : All Laborator | у | | | |
| 39. | Safety | 207966/primary_15/L59 | Listing of Clinical Chemistry Data for Subjects with Any Grade 3 to 5 Lab Toxicity | Remove PCI flag. Treatment as section header. Only include the parameters with G3-5. | M6, M12,<br>EOS |
| 40. | Safety | 207966/primary_15/L59 | Listing of Selected Laboratory Data for Subjects Who<br>Became Pregnant During the Study | Remove PCI flag. Treatment as section header. Selected parameters only. Do not produce if no subject became pregnant on Q2M. | M6, M12 |

| Non-I | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | : Hepatobiliary | (Liver) | | | |
| 41. | Safety | MH2 | Listing of Medical Conditions for Subjects with Liver Stopping Events | GSK Statistical Display Standard | M6, M12 |
| 42. | Safety | SU2 | Listing of Substance Use for Subjects with Liver Stopping Events | GSK Statistical Display Standard | M6, M12 |
| 43. | Safety | 201584/primary_07/L63 | Listing of All Subjects Meeting Liver Stopping Criteria | | M6, M12 |
| 44. | Safety | 207966/primary_15/L52 | Listing of Liver Monitoring/Stopping Event Reporting | | M6, M12 |
| 45. | Safety | 207966/primary_15/L53 | Listing of Liver Event Information for RUCAM Score | | M6, M12 |
| 46. | Safety | 207966/primary_15/L54 | Listing of Liver Biopsy Details | | M6, M12 |
| 47. | Safety | 207966/primary_15/L55 | Listing of Liver Imaging Details | | M6, M12 |
| 48. | Safety | 207966/primary_15/L56 | Listing of Subjects Meeting Hepatobiliary Lab Criteria | | M6, M12 |
| 49. | Safety | 207966/primary_15/L59 | Listing of ALT, AST, Bilirubin (including Total and Direct Bilirubin), INR, and ALP for Subjects Meeting Hepatobiliary Lab Abnormality Criteria | | HL, M6, M12 |
| Safety | : ECG | | | | |
| 50. | Safety | EG3 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | GSK Statistical Display Standard<br>Check all 3: QTcB, QTcF, and<br>Unspecified for PCI criteria | M6, M12 |
| 51. | Safety | EG5 | Listing of Abnormal ECG Findings | GSK Statistical Display Standard | M6, M12 |
| 52. | Safety | 207966/primary_15/L57 | Listing of Potential QTc Interval Prolonging Events of Interest | | M6, M12 |
| 53. | Safety | 207966/primary_15/L58 | Listing of ECG values for Subjects with Potential QTc Interval Prolonging Events of Interest | | M6, M12 |

| Non-IC | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Safety | : Vital Signs | | | | |
| 54. | Safety | VS4 | Listing of All Vital Signs and Anthropometric Parameters | GSK Statistical Display Standard Include weight, height and BMI, waist and hip circumference, and Tanita scale measurements (body Fat, bone mass, musl mass, TBW) | M6, M12 |
| 55. | Safety | PREG1A | Listing of Subjects Who Became Pregnant During the Study | GSK Statistical Display<br>Standard<br>Required by GCSP<br>Include Date of confirmed<br>pregnancy | M6, M12 |
| Safety | : Metabolic Sy | ndrome | , | 1 | |
| 56. | Safety | SAF_L2 | Listing of Clinical Diagnosis Factor Data by Visit for Subjects Diagnosed with Metabolic Syndrome (Maintenance Phase) | | M6, M12 |
| Safety | : Abacavir Hyp | persensitivity | | | |
| 57. | Safety | ABC_HSR<br>_EXPO2 | Listing of Abacavir Hypersensitivity Reaction Record - Exposure to Abacavir | Produce empty listing if no data to report | M6, M12 |
| 58. | Safety | ABC_HSR<br>_DRUG2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject History of Drug Allergies | Do not produce if no data to report | M6, M12 |
| 59. | Safety | ABC_HSR<br>COND2 | Listing of Abacavir Hypersensitivity Reaction Record - Subject and Family Conditions | Do not produce if no data to report | M6, M12 |
| 60. | Safety | ABC_HSR<br>_RASH2 | Listing of Abacavir Hypersensitivity Reaction Record - Skin Rash Details | Do not produce if no data to report | M6, M12 |

| Non-IC | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 61. | Safety | ABC_HSR<br>_SYMP4 | Listing of Abacavir Hypersensitivity Reaction Record - Symptoms | Do not produce if no data to report | M6, M12 |
| 62. | Safety | VS4 | Listing of Abacavir Hypersensitivity Reaction Record - Vital Signs | Do not produce if no data to report | M6, M12 |
| 63. | Safety | ABC_HSR<br>_SYMP6 | Listing of Abacavir Hypersensitivity Reaction Record - Individual Symptoms and Diagnostic Category Assignments | Do not produce if no data to report | M6, M12 |
| Virolo | gy | | | | |
| 64. | CVF | 207966/primary_15/T7.8 | Listing of Viral load, Genotypic, Phenotypic data for Subjects Who Met Confirmed Virologic Failure Criteria | | HL, M6,<br>M12, EOS |
| 65. | Safety | 207966/primary_15/T7.10 | Listing of Viral load, Genotypic, Phenotypic data for Non-CVF Subjects with Genotypic and/or Phenotypic Data | | M6, M12,<br>EOS |
| 66. | CVF | 207966/primary_15/Listing 62 | Listing of Replication Capacity in IN and PR/RT Region | | M6, M12,<br>EOS |
| 67. | Safety | 207966/primary_15/Listing 63 | Listing of Resistance Associated Mutations (Prespecified INSTI and IAS-USA NNRTI) | | M6, M12,<br>EOS |
| 68. | CVF | | Listing of Net Assessment data for Subjects Who Met Confirmed Virologic Failure Criteria | | M6, M12,<br>EOS |
| 69. | Safety | | Listing of Net Assessment data for Non-CVF Subjects with Genotypic and/or Phenotypic Data | | M6, M12,<br>EOS |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | GSK Standard GSK<br>Statistical Display Standard /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK | PK | | | | |
| 70. | PK | 207966/primary_15/L63 | Listing of Plasma PK Concentrations for Subjects Who Became Pregnant During the Study | CAB and RPV With Section<br>Headers. Do not produce if no<br>subject became pregnant on Q2M<br>and continued study | M12 |
| 71. | ITT-E | 207966/primary_15/L63 | Listing of Plasma PK Concentrations at Withdrawal | | M12 |
| 72. | CVF | 207966/primary_15/L63 | Listing of All Plasma PK Concentrations for CVF Subjects | | M12 |

# 16.16. Appendix 16: Example Mock Shells for Data Displays

Available upon request